### Janssen Research & Development \*

### Statistical Analysis Plan Amendment 1

A Phase 3 Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Pimodivir in Combination With the Standard-of-care Treatment in Adolescent, Adult, and Elderly Hospitalized Patients With Influenza A Infection

Protocol 63623872FLZ3001; Phase 3

JNJ-63623872-ZCD (Pimodivir)

Status: Approved

Date: 1 July 2020

**Prepared by:** Janssen Research & Development, a division of Janssen Pharmaceutica NV

**Document No.:** EDMS-ERI-149599549, 2.0

**Compliance:** The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

# **Confidentiality Statement**

The information provided herein contains Company trade secrets, commercial or financial information that the Company customarily holds close and treats as confidential. The information is being provided under the assurance that the recipient will maintain the confidentiality of the information under applicable statutes, regulations, rules, protective orders or otherwise.

# **TABLE OF CONTENTS**

| TABLE | OF CONTENTS | <mark>2</mark> |
|---|---|---|
| AMEN | DMENT HISTORY | 5 |
| ABBRI | EVIATIONS | 9 |
| 1. II | NTRODUCTION | 44 |
| 1.1. | Trial Objectives | |
| 1.2. | Trial Design | |
| 1.3. | Statistical Hypotheses for Trial Objectives | |
| 1.4. | Sample Size Justification | |
| 1.5. | Randomization and Blinding | |
| 2. G | ENERAL ANALYSIS DEFINITIONS | 15 |
| 2.1. | Visit Windows, Phase Definitions and Baseline | |
| 2.1. | Phase Definitions | |
| 2.1.1. | Analysis Visits | |
| 2.1.3. | Analysis Timepoints | |
| 2.1.4. | Use of Records per Analysis Visit and Timepoint | |
| 2.1.5. | Unscheduled Assessments | |
| 2.2. | Analysis Sets | |
| 2.2.1. | All Randomized Analysis Sets | |
| 2.2.1.1 | | |
| 2.2.1.2 | | |
| 2.2.2. | Efficacy Analysis Sets | |
| 2.2.2.1 | | |
| 2.2.2.2 | | |
| 2.2.2.3 | \ / | |
| 2.2.3. | Safety Analysis Set | |
| 2.2.3.1 | | 21 |
| 2.2.4. | Pharmacokinetics (PK) Analysis Set | |
| 2.2.5. | Pharmacodynamics (PD) Analysis Set | |
| 2.3. | Definition of Subgroups | |
| 2.4. | Study Day and Relative Day | 24 |
| 2.5. | Baseline and Endpoint | 24 |
| 2.6. | Other Definitions | 25 |
| 3. II | NTERIM ANALYSIS AND DATA MONITORING COMMITTEE REVIEW | 25 |
| 3.1. | Interim Analyses | 25 |
| 3.2. | Independent Data Monitoring Committee | 26 |
| 4. S | UBJECT INFORMATION | 27 |
| 4.1. | Demographics and Baseline Characteristics | |
| 4.2. | Disposition Information | |
| 4.3. | Treatment Compliance | |
| 4.4. | Extent of Exposure | |
| 4.5. | Protocol Deviations | |
| 4.6. | Prior and Concomitant Medications | 30 |
| 4.7. | Medical history | 31 |
| 5. E | FFICACY | 33 |
| 5.1. | Analysis Specifications | 33 |
| 5.1.1. | Level of Significance | |
| 5.1.2. | Statistical Methodology for Evaluation at the Final Analysis | 35 |

| <b>-</b> 4 0 | Data Hara Wara Data | 0.0 |
|---|---|---|
| 5.1.3. | <b>J</b> | |
| 5.1.4. | | |
| 5.2. | Primary Efficacy Endpoint(s) | |
| 5.2.1. | | |
| 5.2.2. | | |
| 5.2.3. | <b>,</b> | |
| 5.3. | Major Secondary Endpoints | |
| 5.3.1. | | |
| 5.3.1. | | |
| 5.3.1. | | |
| 5.3.1. | · | |
| 5.3.2. | , and the state of | |
| 5.3.2. | | |
| 5.3.2. | | |
| 5.3.2. | 3. Patient Reported Outcomes | 61 |
| _ | | |
| | TASTE AND SWALLOWABILITY | |
| 6.1. | Definition | |
| 6.2. | Analysis Methods | 62 |
| _ | | |
| | SAFETY | |
| 7.1. | Adverse Events | |
| 7.1.1. | | |
| 7.1.2. | <b>,</b> | |
| 7.2. | Clinical Laboratory Tests | |
| 7.2.1. | | |
| 7.2.2. | , and the state of | |
| 7.3. | Vital signs | |
| 7.3.1. | | |
| 7.3.2. | Analysis Methods | <mark>7</mark> 0 |
| 7.4. | Physical examinations | 70 |
| 7.5. | Electrocardiogram | 71 |
| 7.5.1. | Definitions | 71 |
| 7.5.2. | Analysis Methods | 71 |
| 7.6. | National Early Warning Score | 72 |
| 7.6.1. | Definitions | <mark>72</mark> |
| 7.6.2. | Analysis Methods | 74 |
| | RESISTANCE | |
| 8.1. | Viral Phenotype | 75 |
| 8.2. | Viral Genotype | 75 |
| _ | | |
| | PHARMACOKINETICS/PHARMACODYNAMICS | |
| 9.1. | Pharmacokinetics | |
| 9.2. | Pharmacokinetic/Pharmacodynamic Relationships | 76 |
| 40 | HEALTH FOONOMICS | |
| | HEALTH ECONOMICS | |
| 10.1. | Definitions | |
| 10.2. | Analysis Methods | 78 |
| DEEE | PENOEO | 70 |
| KEFE | RENCES | /9 |
| ATT 4 | ACHMENTS | 90 |
| ALIA | NOTINILIA I O | 60 |
| ΔΤΤΛ | ACHMENT 1. : ANTICIPATED EVENTS AND ANTICIPATED EVENT GROUPS | 20 |
| ~: IA | ACTIVIDITATION AT LE EVENTO AND ANTIONATED EVENT GROUPS | |
| ΑΤΤΔ | ACHMENT 2. : WHO TOXICITY GRADING SCALE FOR DETERMINING THE SEVER | ITY |
| | OF ADVERSE EVENTS (FEB 2003) | |

| ATTACHMENT 3. | : WHO GRADING SCALE VITAL SIGNS | 90 |
|---------------|---------------------------------|-------|
| ATTACHMENT 4. | : ECG ABNORMALITIES | 91 |
| ATTACHMENT 5. | : EQ-5D VALUATION INDEX | 92 |
| ATTACHMENT 6. | : HRS DERIVATION | . 110 |

#### **AMENDMENT HISTORY**

### Amendment 1 (1 July 2020)

The overall reason for the amendment: The overall reason for the amendment is to make general updates to the text including minor grammatical, formatting, or spelling changes throughout the SAP for clarification purposes and to align with protocol amendment 2. A new section is added: to include analysis of pharmacokinetic parameters and pharmacodynamic analyses. Three new subgroups were added namely influenza season, study period (before interim, after interim) and COVID-19 impacted (Yes/No). To assess the impact of COVID-19, several tables and listings are added presenting the COVID-19 impacted subjects separately. Two new secondary endpoints based on a clinically relevant change from baseline in EQ-5D VAS are included. A new endpoint related to the HRS is added: the fundamental hospital recovery scale, reflecting the actual location/situation, which will be analysed each day from Day 2 to 14. Additionally, the following four new secondary endpoints were also added: time to NEWS2 ≤ 2, time to clinical improvement, time to clinical failure and incidence of mortality per day.

#### The table below gives an overview of the changes in all applicable sections

**Summary of changes:** An additional analysis set was defined for the analysis of the primary endpoint and the six most important secondary endpoints. Additional analysis sets were defined for the pharmacodynamic analyses and the analysis of pharmacokinetics parameters. The criterion: "Subjects did not switch to another influenza antiviral as a part of the SOC during the treatment period" was added and the criterion: "subjects that did not use a concomitant medication that may have affected the efficacy of the study drug" was removed from the definition of the per protocol analysis set. The in- and exclusion criteria needed to define the per protocol analysis set are updated and added.

- 2.2.2 Efficacy Analysis Sets
- 2.2.2.2 Per Protocol Set (PP)
- 2.2.2.3 Intent-To-Treat non-infected (ITT-ni) Set
- 2.2.4 Pharmacokinetics Analysis Set
- 2.2.5 Pharmacodynamics Analysis Set

**Summary of changes:** Baseline resistance categories were defined based on influenza polymerase basic protein 2 genotype and phenotype. General re-formatting to assist readability of the section. The subgroups influenza season, study period (pre- and post-interim) and COVID-19 impacted (yes/no) are added.

2.3 Definition of Subgroups

**Summary of changes:** Detailing the definition of baseline ECG measurement was added. The baseline HRS is clarified. The last study visits for vital signs, NEWS2, ECG and central laboratory parameters are also defined.

2.5 Baseline and Endpoint

**Summary of changes:** A new section (2.6) was added to describe details of the analysis to support marketing authorization approval by FDA and EMA where a subset of patients is used with oseltamivir use as part of their SOC treatment and to include text to allow for potential analyses for other regions or countries

### 2.6 Other Definitions

**Summary of changes:** The number of subjects impacted by COVID-19 are added in the disposition table per analysis set. The table showing the number of subjects that discontinued is extended to show the number of subjects that discontinued due to COVID-19. Missed visits or changed visits due to COVID will also be presented. A listing showing the exposure to study drug for subjects impacted by COVID-19 is added. Major and minor protocol deviations related to COVID-19 are included. Concomitant therapy that was taken for COVID-19 infection are presented in an additional table.

### **4 SUBJECT INFORMATION**

- 4.1 Demographics and Baseline Characteristics
- 4.2 Disposition Information
- 4.4 Extent of Exposure
- 4.5 Protocol Deviations
- 4.6 Prior and Concomitant Medications

**Summary of changes:** A new section (5.1.3) was added to describe how the actual values of the stratification factors are derived.

#### 5.1.3 Stratification Factors

**Summary of changes:** The text describing the estimand is updated to align with the ICH E9 addendum guidance and to include MI methods for missing HRS values due to COVID-19 and not due to COVID-19

#### 5.2.2 Estimand

**Summary of changes:** the multiple imputation methods are applied on the missing HRS values at day 6 due to COVID-19 and to missing HRS values on day 6 not due to COVID-19 in case the prevalence is more then > 5%. A table is added to show the number (%) missing HRS values on day 6 by reason of missing.

# 5.2.3 Analysis Methods

Summary of changes: The fundamental hospital recovery scale, reflecting the actual location/situation of the subject evaluated daily from Day 2 to Day 14 is added. Time to NEWS2  $\leq 2$ , time to clinical improvement, time to clinical failure and incidence of mortality per day are

added secondary endpoints. Re-hospitalizations are defined at the description of time to hospital discharge.

### 5.3.1.1 Clinical Outcome

**Summary of changes:** Adverse events leading to study discontinuation, AEs, serious AEs and non-serious AEs related to COVID-19 were added to the list for the adverse events summary table. The definition of a treatment emergent AE was detailed. A table of influenza related complications as assessed by the investigator was added. Tables that show AEs related to COVID-19 infection, SAEs related to COVID-19 infection, AEs related to COVID-19 infection leading to death and a listing showing the AEs related to COVID-19 infection are added.

#### 7.1.1 Definitions

### 7.1.2 Analysis Methods

**Summary of changes:** The change from baseline in EQ-5D VAS is categorized in two ways providing two additional endpoints.

# 5.3.1.3 Other Patient Reported Outcome

**Summary of changes:** A bootstrapping method for calculating the median time to event with 95% confidence interval from the accelerated failure time model was added.

### 5.3.2 Analysis Methods

**Summary of changes:** Additional details regarding number of loose stools per day and stool consistency will be collected for subjects who report diarrhea adverse events. A confirmed diarrhea event is defined and the analysis of these events is described.

#### 7.1.1 Definitions

#### 7.1.2 Analysis Methods

**Summary of changes:** The use and definition of NEWS2 is explained and added.

NEWS2 will be used in the analyses.

#### 7.6 NEW Score

**Summary of changes:** A new section was added to describe the analysis of the pharmacokinetic parameters and to explore their relationships with efficacy and safety.

## 9 Pharmacokinetics/Pharmacodynamics

#### 9.1 Pharmacokinetics

# 9.2 Pharmacokinetic/Pharmacodynamic Relationships

**Summary of changes:** the anticipated events table has been corrected for a typo and to include an additional MedDRA preferred term for diabetic complications

Attachment 1

#### **ABBREVIATIONS**

ACVPU Alert, new confusion, voice, pain, unresponsive

AE adverse event

AFT accelerated failure time

ATC Anatomical Therapeutic Chemical

AUC area under the curve

AUC<sub>12h</sub> area under the plasma concentration-time curve from time 0 to 12 hours

bid bis in die; twice daily
BMI body mass index
CI confidence interval

C<sub>max</sub> maximum plasma concentration COPD Chronic Obstructive Pulmonary Disease

CTP clinical trial protocol

C<sub>trough</sub> Plasma concentration just prior to the beginning or at the end of a dosing interval

 $\begin{array}{lll} CV & coefficient of variation \\ DBP & diastolic blood pressure \\ DMC & Data Monitoring Committee \\ DPS & Data Presentation Specifications \\ EC_{50} & 50\% \ effective \ concentration \\ \end{array}$ 

ECG electrocardiogram

eCRF electronic case report form EMA European Medicines Agency

ePRO Electronic Patient-reported outcome (Device used for recording of patient-reported outcomes)

EQ-5D European Quality of Life 5 Dimensions

FDA Food and Drug Administration

GMR geometric mean ratio
HRS Hospital recovery scale
IC<sub>50</sub> 50% inhibitory concentration
ICF informed consent form

ICH International Conference on Harmonization

ICU Intensive Care Unit

IDMC Independent Data Monitoring Committee

ITT Intent-To-Treat

ITT-i Intent-To-Treat infected
ITT-ni Intent-To-Treat non-infected
IWRS Interactive web response system

LOD limit of detection LOQ Limit of quantification

MedDRA Medical Dictionary for Regulatory Activities

MT Mid-turbinate

NAI neuraminidase inhibitor NEWS National early warning score NEWS2 National early warning score 2

OST oseltamivir

PA Polymerase acidic protein
PB2 (1) polymerase basic protein 2 (1)
PD pharmacodynamic(s)

PGIC Patient Global Impression of Change PGIS Patient Global Impression of Severity

PK pharmacokinetic(s)
PP Per Protocol
PT preferred term

qRT-PCR quantitative real time polymerase chain reaction

SDTM Subject Data Tabulation Model

SAE serious adverse event SAP statistical analysis plan

| SBP | systolic blood pressure |
|-----|-------------------------|
| SI | international system |
| SOC | standard of care |

SSG Statistical support group

TEAE Treatment Emergent Adverse Events

 $\begin{array}{ll} T_{max} & Time \ to \ reach \ C_{max} \\ VAS & Visual \ analogue \ scale \end{array}$ 

#### 1. INTRODUCTION

This statistical analysis plan (SAP) contains definitions of analysis sets, derived variables and statistical methods for the analysis of efficacy and safety of the investigational compound pimodivir (JNJ-63623872). Separate documents for mock shells and table of contents for TFLs (DPS) are also produced. The SAP is to be interpreted in conjunction with the protocol.

Pimodivir (formerly known as VX-787 and JNJ-63623872) is a non-nucleotide inhibitor of the polymerase basic protein 2 (PB2) subunit of the influenza A virus polymerase complex and is currently in Phase 3 development as treatment for influenza A infection.

# 1.1. Trial Objectives

## **Primary Objective**

The primary objective is to evaluate superiority of pimodivir in combination with standard-of-care (SOC) treatment compared to placebo in combination with SOC treatment on Day 6, with respect to the clinical outcome on the hospital recovery scale.

### **Secondary Objectives**

The secondary objectives are:

- To investigate the safety and tolerability of pimodivir in combination with SOC treatment compared to placebo in combination with SOC treatment.
- To evaluate superiority with respect to the time from start of study drug to hospital discharge
  in subjects treated with pimodivir in combination with SOC treatment compared to placebo
  in combination with SOC treatment.
- To evaluate superiority with respect to the time from intensive care unit (ICU) admission to ICU discharge in subjects treated with pimodivir in combination with SOC treatment compared to placebo in combination with SOC treatment.
- To evaluate superiority with respect to the time from start to end of mechanical ventilation in subjects treated with pimodivir in combination with SOC treatment compared to placebo in combination with SOC treatment.
- To evaluate superiority of pimodivir in combination with SOC treatment compared to placebo in combination with SOC treatment each separated day from Days 2 to 14 (excluding the primary time point), with respect to the clinical outcome on the hospital recovery scale.
- To evaluate superiority with respect to the time to return to daily activities in subjects treated with pimodivir in combination with SOC treatment compared to placebo in combination with SOC treatment.
- To evaluate superiority with respect to the incidence of complications associated with influenza after the start of study treatment in subjects treated with pimodivir in combination with SOC treatment compared to placebo in combination with SOC treatment.
- To investigate all-cause mortality in the pimodivir in combination with SOC treatment arm, compared to the placebo in combination with SOC treatment arm.

- To investigate the incidence and duration of antibiotic treatment in the pimodivir in combination with SOC treatment arm, compared to the placebo in combination with SOC treatment arm.
- To investigate the number (proportion) of subjects needing extended treatment in the pimodivir in combination with SOC treatment arm, compared to the placebo in combination with SOC treatment arm.
- To investigate the number (proportion) of subjects requiring re-hospitalization in the pimodivir in combination with SOC treatment arm, compared to the placebo in combination with SOC treatment arm.
- To investigate the number (proportion) of subjects not hospitalized at Day 6 in the pimodivir in combination with SOC treatment arm, compared to the placebo in combination with SOC treatment arm.
- To investigate the time to clinical response in the pimodivir in combination with SOC treatment arm, compared to the placebo in combination with SOC treatment arm.
- To investigate the time to improvement of respiratory status in the pimodivir in combination with SOC treatment arm, compared to the placebo in combination with SOC treatment arm.
- To assess the pharmacokinetics (PK) of pimodivir and to explore the PK/pharmacodynamics (PD) relationships of pimodivir for efficacy and safety.
- To investigate the acceptability (taste and swallowability) of the pimodivir formulation in adolescents.
- To evaluate superiority with respect to the following influenza A viral parameters in the pimodivir treatment arm compared to the control arm by qRT-PCR and viral culture:
  - Time to viral negativity.
  - Viral load over time.
- To investigate the emergence of viral resistance against pimodivir detected by genotyping and/or phenotyping.

# 1.2. Trial Design

This is a Phase 3 randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy and safety of pimodivir in combination with SOC treatment vs placebo in combination with SOC treatment in adolescent (13 to 17 years), adult (18 to 65 years), and elderly (>65 to ≤85 years) hospitalized subjects with influenza A infection. A target of 600 hospitalized influenza A-infected subjects will be randomly enrolled in this study with 300 subjects planned per treatment arm. The aim is to enroll a minimum of 60 adolescent subjects in this study in selected countries and study sites consistent with local regulations. The randomization will be stratified for screening NEWS2 (4-5 or >5) (NEWS is changed to NEWS2 per CTP amendment 2), type of baseline SOC (including or not including influenza antiviral treatment), and time since onset of influenza symptoms (first administration of study drug within 72 hours or between 72 and 96 hours since onset of influenza symptoms). The study population should consist of at least 75% of subjects

(75% of the total planned sample size of 600 subjects) with first administration of study drug  $\leq$ 72 hours since onset of influenza symptoms.

Subjects who meet all eligibility criteria will be randomized in a 1:1 ratio to receive 1 of the following treatments.

- Treatment Arm 1: pimodivir 600 mg bid for 5 days + SOC treatment\*
- Treatment Arm 2: pimodivir placebo bid for 5 days + SOC treatment\*

\*SOC treatment is determined by the investigator based on local practice, and may include influenza antivirals and/or supportive care only. For further details see protocol Section 3.1.

# 1.3. Statistical Hypotheses for Trial Objectives

The primary endpoint is the hospital recovery scale as assessed on Day 6. The alternative hypothesis is that the outcome on the hospital recovery scale with pimodivir in combination with SOC treatment is statistically superior to treatment with placebo in combination with SOC treatment on Day 6 in hospitalized subjects with influenza A infection.

# 1.4. Sample Size Justification

The study will enroll 600 subjects between the ages of 13 and 85 years, inclusive. Subjects will be randomized 1:1 to one of the treatment arms.

The sample size is based on the primary endpoint of the hospital recovery scale at Day 6. Based on the proportional odds model and assuming a benefit of approximately 38% reduction of the common odds ratio, a total sample size of 600 subjects (randomized 1:1) is required to obtain a power of 90% [11]. Inclusion of stratification factors would provide some improvement on the derived power.

In the sample size calculation it is assumed that the distribution of subjects treated with placebo in combination with SOC treatment will be as follows on Day 6:

- Not hospitalized: 30%
- Non-ICU hospitalization, not requiring supplemental oxygen: 30%
- Non-ICU hospitalization, requiring supplemental oxygen: 25%
- Admitted to the ICU, not requiring invasive mechanical ventilation: 5%
- Requiring invasive mechanical ventilation: 5%
- Death: 5%

This sample size is robust to mild to moderate changes in this distribution.

# 1.5. Randomization and Blinding

#### Randomization

Central randomization will be implemented in this study. Subjects will be randomly assigned to 1 of 2 treatment arms in a 1:1 ratio based on a computer-generated randomization schedule prepared before the study by or under the supervision of the sponsor. The randomization will be balanced by using randomly permuted blocks and will be stratified for NEWS2 (4-5 or >5) (NEWS

is changed to NEWS2 per CTP amendment 2) at screening, type of baseline SOC (including or not including influenza antiviral treatment), and time since onset of influenza symptoms (first administration of study drug ≤72 hours or between 72 and 96 hours since onset of influenza symptoms). The interactive web response system (IWRS) will assign a unique treatment code, which will dictate the treatment assignment and matching study drug kit for the subject. The requestor must use his or her own user identification and personal identification number when contacting the IWRS and will then give the relevant subject details to uniquely identify the subject.

#### **Blinding**

The investigator will not be provided with randomization codes. The codes will be maintained within the IWRS, which has the functionality to allow the investigator to break the blind for an individual subject.

Data that may potentially unblind the treatment assignment (ie, study drug plasma concentrations) will be handled with special care to ensure that the integrity of the blind is maintained and the potential for bias is minimized. This can include making special provisions, such as segregating the data in question from view by the investigators, clinical team, or others as appropriate until the time of database lock and unblinding.

Under normal circumstances, the blind should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the blind should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the investigator may in an emergency determine the identity of the treatment by contacting the IWRS. It is recommended that the investigator contact the sponsor or its designee if possible to discuss the particular situation, before breaking the blind. Telephone contact with the sponsor or its designee will be available 24 hours per day, 7 days per week. In the event the blind is broken, the sponsor must be informed as soon as possible. The date, time, and reason for the unblinding must be documented by the IWRS, in the appropriate section of the electronic case report form (eCRF) and in the source documents. The documentation received from the IWRS indicating the code break must be retained with the subject's source documents in a secure manner.

#### 2. GENERAL ANALYSIS DEFINITIONS

All analysis dataset preparations and statistical analyses will be performed using SAS® version 9.2 or higher.

## 2.1. Visit Windows, Phase Definitions and Baseline

The study is set up as shown in Figure 1. The phases will be constructed as shown in Table 1.

Figure 1: Study time line.

| Day | 0 | 1 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 14 | 19 | 28 | 33 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm<br>1 | Scr. | | odivir<br>- SOC | | _ | SOC | | | mg b<br>treatr | | Fo | ollow-up | | |
| Arm<br>2 | Scr. | | ebo bi<br>ment | d + \$ | SOC | | | bid<br>exter | | | Fo | ollow-up | | |

<sup>&</sup>lt;sup>1</sup> A subject with extended treatment will be treated an extra 5 days compared to the subjects without extended treatment.

Note: Depending on the time of screening/enrollment, subjects will receive 1 dose (evening) or 2 doses (morning and evening) of study drug on Day 1. For subjects who receive only 1 dose of pimodivir or placebo on Day 1 (evening), dosing should continue until the morning of Day 6 so that all subjects receive 10 doses in total, or for subjects with extended treatment until the morning of Day 11, so all subjects with extended treatment receive 20 doses in total.

#### 2.1.1. Phase Definitions

**Table 1: Construction of phases** 

| Trial phase | Trial subperiod*1 | Start date | End date |
|---|---|---|---|
| Screening (phase 1) | | The date of signing the informed consent with 00:00 as a timepart | 1 minute before the first study drug intake |
| Treatment (phase 2) | | Datetime of first study drug intake *4 | Datetime of last study drug intake*4 + 24 hours |
| | Planned Treatment (subperiod 1)*2 | Datetime of first study drug intake *4 | If extended treatment then Datetime of first study drug intake in extended treatment subperiod – 1 minute Else Datetime of last study drug intake*4 + 24 hours |
| | Extended Treatment (subperiod 2)*3 | Datetime of first study drug intake in extended treatment subperiod*4 | Datetime of last study drug intake*4 + 24 hours |
| Follow-up (phase 3) | | End of the treatment phase +1 minute | Trial termination date (or date of last contact if later) |

<sup>\*1:</sup> A treatment period will be constructed in the derived datasets with the same start and end date as the treatment phase.

<sup>\*2:</sup> The planned treatment subperiod will be present for all treated subjects.

<sup>\*3:</sup> The extended treatment subperiod will only be present for all subjects with extended treatment.

<sup>\*4:</sup> In case the time part of the study drug intake is missing the imputed time part will be used as described below.

Additionally, the treatment phase and follow-up phase will be combined in the analysis.

In case the time part of first study drug intake is missing the randomization time will be used. In case the time part of the randomization time is also missing we impute the time part with 8:00 if taken in the morning or with 20:00 if study drug was taken in the evening. In case the time of the last study drug intake is missing, the time part will be imputed with 8:00 if the last study drug was taken in the morning or with 20:00 if the last study drug was taken in the evening.

In case the time part of first intake of the treatment extension is missing, the time part will be imputed with 8:00 if the last study drug of the planned 5 days of treatment was taken in the morning or with 20:00 if the last study drug was taken in the evening.

The last phase, whichever it is for a subject, always ends on 23:59 of the day of trial termination (or date of last contact if later).

Assessments will be assigned to phases and subperiods based on their start datetime, but seconds will not be taken into account. If only one assessment is expected per day and the day part of the start date of the assessment is present but the time part is missing, the assessment will be treated as if it happened at 00:00 of the day of the assessment (except for Adverse Events see details in Section 7.1). No imputations on missing times/time parts will be made in the analysis datasets.

In case more than one assessment per day is expected and time part is missing:

- 1. Allocate according to the timepoint: Morning=00:00, Middle of the day=12:00, Evening=20:00
- 2. If 1 timepoint is missing on day x: Check the non-missing timepoints of the other records on this day x. Allocate this record to the timepoint of day x that is not already covered. Then apply 1.
- 3. If 2 timepoints are missing on day x: Check the non-missing timepoint of the other record on this day x. Allocate these records to the timepoints of day x that are not already covered, assigning the smallest XXSPID value to the earlier timepoint and the larger XXSPID value to the later timepoint. Then apply 1.
- 4. If 3 timepoints are missing on day x: allocate using the values of XXSPID, i.e. lowest number is morning, next is middle of the day, highest number is evening. Then apply 1.

### 2.1.2. Analysis Visits

In general, AVISIT will be derived as the day of a scheduled visit, assessment or self-assessment as recorded in the respective SDTM, including the safety follow-up visit and day 28 final study visit (e.g. 'Day 4'). AVISITN will be the numeric counterpart (e.g. for 'Day 4' AVISITN will be 4). The AVISIT for scheduled measurements before first intake will be set to 'Screening' with AVISITN = -1. For specifications on the baseline record and endpoint record see Section 2.5.

For post-baseline assessments of the Daily Activities Resumption (Return to daily activity), Patient Global Impression of Severity (PGIS), Patient Global Impression of Change (PGIC) and

the European Quality of Life 5 Dimensions (EQ-5D) questionnaires, AVISIT and AVISITN will be derived from the number of days in the study relative to the start of study treatment (reldy, see Section 2.4). Post-baseline assessments taken from 00:00 until 02:00 will be assigned to the day before (e.g. a recording on Day 4 at 01:00 will be assigned AVISIT= Day 3).

# 2.1.3. Analysis Timepoints

For parameters that were assessed more than once daily, the analysis timepoint (ATPT) will be the timepoint as reported in the database. In case there are multiple records per planned timepoint take the last in time.

For hospitalized subjects we expect 3 assessments per day. If the timepoint is missing but the date time is known, then we impute as follows:

If date time is within [00:00, 11:00] then allocate the morning timepoint If date time is within [11:01, 16:00] then allocate the midday timepoint if date time is within [16:01, 23:59] then allocate the evening timepoint For subjects that are discharged we expect only 1 vital sign assessment. Therefore

For subjects that are discharged we expect only 1 vital sign assessment. Therefore in case the timepoint is filled in, we set it to empty.

For NEWS2, select for each of the parameters one record per timepoint as described above. The date and time of the NEWS2 will be derived from the last date time of each of the parameters and this will be used to allocate the NEWS2 to a phase. A subject received oxygen at the planned timepoint if the date time of the oxygen saturation measurement falls within the period that the subject received supplemental oxygen.

# 2.1.4. Use of Records per Analysis Visit and Timepoint

To ensure only one record is used per analysis visit for the Return to daily activity and PGIS questionnaires only one questionnaire should be selected for analysis. Following rules should be followed to select the questionnaire.

- 1. The questionnaire latest in time is used.
- 2. If more than one questionnaire is still selected, the questionnaire with the highest sequence number is used.

To ensure only one record is used per analysis visit for the PGIC and EQ-5D questionnaires the following rules should be followed to select the questionnaire.

Listed below (Table 2) are the visit windows and the target days for each visit where PGIC and EQ-5D are recorded. The reference day is Study Day 1, the date of first intake of study drug.

- 1. If a subject has 2 or more actual visits in one visit window, the visit closest to the target day will be used as the protocol visit for that visit window.
- 2. If 2 actual visits are equidistant from the target day within a visit window, the later visit in time is used.

Table 2: Visit Windows for PGIC and EQ-5D

| Scheduled Visit<br>Number | Time Interval (label on output) | Time Interval (Day)* | Target Time Point (Day) |
|---|---|---|---|
| 6 | Day 6 | [2 to 10] | 6 |
| 14 | Day 14 | [11 to 20] | 14 |
| 28 | Day 28 | [21 to 38] | 28 |
| For subjects on extende | For subjects on extended treatment: | | |
| 14 | Day 14 | [11 to 16] | 14 |
| 19 | Day 19 | [17 to 22] | 19 |
| 33 | Day 33 | [23 to 38] | 33 |

<sup>\*</sup>Relative to Study Day 1

#### 2.1.5. Unscheduled Assessments

In general, all scheduled assessments after first administration of study drug will be used. Unscheduled assessments will not be used in descriptive statistics or any per-time point analysis, but will be shown in listings as applicable. Pre-dose unscheduled assessments will be taken into account for baseline determination and post first dose unscheduled assessments will be taken into account for worst-case determination.

For PRO assessments, both scheduled and unscheduled assessments will be taken into account to determine which assessment will be used per analysis visit / timepoint as described in Section 2.1.4.

For time to response endpoints, recordings taken at unscheduled visits will be taken into account unless indicated differently.

# 2.2. Analysis Sets

## 2.2.1. All Randomized Analysis Sets

### 2.2.1.1. All Randomized Analysis Set (RAND)

All randomized subjects with a randomization date time at or before the date time of first intake of study drug, or with a randomization date time and no study drug intake.

## 2.2.1.2. Randomized and/or Treated Analysis Set (RT)

All randomized subjects and/or all subjects who received at least 1 dose of study drug. The Randomized and/or Treated Analysis Set (RT) will be used in all listings unless specified otherwise for a specific display.

### 2.2.2. Efficacy Analysis Sets

Efficacy will be analyzed on the intent-to-treat infected (ITT-i) set and by randomized treatment. The primary efficacy endpoint will also be analyzed on the Per Protocol set. The primary efficacy endpoint and the six most important secondary endpoints (all endpoints included in the hierarchical

18

testing procedure at the final analysis) will also be analyzed on the intent-to-treat non-infected (ITT-ni) set and by randomized treatment.

## 2.2.2.1. Intent-To-Treat infected (ITT-i) set

All subjects from the RAND analysis set who receive at least 1 dose of study drug and who have a confirmed infection with influenza A. Confirmation of Influenza A infection will be obtained from virology data. If there are no virology data available at the final analysis, then a subject will be excluded from the ITT-i set. Analysis on the ITT-i set will be analyzed as randomized.

A subject is considered to have a confirmed infection with influenza A if he/she has:

at least one positive PCR result from central lab testing at baseline or pre-baseline;

else

at least two positive PCR results from central lab testing post-baseline;

else

• at least one positive result from local lab testing for influenza A at baseline or pre-baseline, provided that no central lab testing is available at baseline or pre-baseline.

Note: viral load (PCR) results from central lab testing recorded as 'TARGET NOT DETECTED' will be considered as negative, all other non-missing results as positive (i.e. between LOD and LOQ, or quantifiable (above LOQ)).

Note: If no viral load measurement is available prior to first study drug intake then the first viral load result from the central lab testing obtained up to and including 30 minutes after first dose of study drug will be considered as the baseline assessment. If no baseline central lab measurement is available, the first viral load result from the local lab test obtained up to and including 30 minutes after first dose of study drug will be considered as the baseline local test assessment in case no local lab test is available at baseline or pre-baseline.

Note: viral load results from the central lab testing obtained from leftover samples from the local virology test will be considered in determining confirmed infection with influenza A.

### 2.2.2.2. Per Protocol Set (PP)

All subjects in the ITT-i set without major protocol deviations that may have an impact on the efficacy analysis.

Decisions regarding which subjects are included in the per protocol set will be made before database lock on following criteria. Subjects will be included in the PP set in case:

- Subjects missed at most 3 doses in total or at most 2 consecutive doses. On the day of randomization or the next day at least one dose needs to be taken.
- The actual treatment must be the same as the planned treatment
- No unblinding may have taken place

- Subjects may not violate inclusion criteria 2,3,4 and 6 and exclusion criteria 1, 6, 9, 12 and 13.
- Influenza antiviral as part of the SOC was started no later than the day of first study drug intake,
- Subjects did not switch to another influenza antiviral as a part of the SOC

| Inclusion/ | Criterion | Description |
|---|---|---|
| Exclusion | number | |
| Inclusion | 2 | Tested positive for influenza A infection after the onset of symptoms, using a rapid influenza diagnostic test (RIDT) or, if available, a PCR-based or other rapid molecular diagnostic assay. |
| Inclusion | 3 | Requires hospitalization to treat influenza infection and/or to treat complications of influenza infection (eg, radiological signs of lower respiratory tract disease, septic shock, central nervous system [CNS] involvement, myositis, rhabdomyolysis, acute exacerbation of chronic kidney disease, severe dehydration, myocarditis, pericarditis, ischemic heart disease, exacerbation of underlying chronic pulmonary disease, including asthma, chronic obstructive pulmonary disease [COPD], decompensation of previously controlled diabetes mellitus), including subjects admitted to the ICU. Note: for the purpose of the protocol, subjects admitted under "observation" status with an anticipated length of stay beyond 24 hours are eligible for enrollment. |
| Inclusion | 4 | Enrollment and initiation of study drug treatment ≤96hours after onset of influenza symptoms. |
| Inclusion | 6 | Having a screening/baseline NEWS2 of ≥4. |
| Exclusion | 1 | Received more than 3 doses of influenza antiviral medication (eg, OST or zanamivir), or any dose of RBV within 2 weeks, prior to first study drug intake. Received IV peramivir more than 1 day prior to screening. |
| Exclusion | 6 | Severely immunocompromised in the opinion of the investigator (eg, known cluster of differentiation 4 <sup>+</sup> [CD4 <sup>+</sup> ] count <200 cells/mm <sup>3</sup> , absolute neutrophil count <750/mm <sup>3</sup> , first course of chemotherapy completed within 2 weeks prior to screening, history of stem cell transplant within 1 year prior to screening, history of a lung transplant). |
| Exclusion | 9 | Taken any disallowed therapies as noted in the Protocol, pre-study and concomitant therapy before the planned first dose of study drug. |
| Exclusion | 12 | Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments (eg, subject is unable to swallow medication tablets outside the hospital setting), with the exception of ePRO completion (see the protocol) ie, if a subject is not able to complete ePRO, the subject is still allowed to be enrolled in the study. |
| Exclusion | 13 | Subject has presence of any pre-existing illness, clinically significant laboratory abnormalities, ECG findings, or physical examination findings that, in the opinion of the investigator, would place the subject at an unreasonably increased risk through participation in this study. The investigator should consider the laboratory parameter criteria for study drug discontinuation when screening a subject for enrollment. |

# 2.2.2.3. Intent-To-Treat non-infected (ITT-ni) Set

All subjects from the RAND analysis set who receive at least 1 dose of study drug and who do not have a confirmed infection with influenza A.

### 2.2.3. Safety Analysis Set

# 2.2.3.1. Safety Set or All Subjects Treated (AST)

All safety endpoints will be evaluated on the Safety population, consisting of all subjects who received at least one dose of study drug and will be analyzed by treatment arm as treated.

## 2.2.4. Pharmacokinetics (PK) Analysis Set

The PK analysis set is defined as subjects who have received at least 1 dose of pimodivir and have at least 1 valid blood sample drawn for PK analysis.

# 2.2.5. Pharmacodynamics (PD) Analysis Set

The PD analysis set is defined as all subjects in the PK analysis set for whom at least one PK parameter could be derived.

# 2.3. Definition of Subgroups

See Table 3 for the definitions of all the subgroups. The third column in the table indicates for which endpoints the subgroup is applied.

Descriptive statistics will be produced for the different subgroups.

In demographics and baseline disease characteristics, the following subgroups will be used:

- Region
- Influenza A subtype category
- Treatment extension
- Age group
- Time since onset of influenza symptoms (actual: ≤72 hours, >72 hours)
- Time since onset of influenza symptoms (actual: ≤48 hours, >48 72 hours, >72 hours)
- Type of SOC at baseline (actual)
- NEWS2 at screening (actual)
- Baseline resistance
- Any baseline polymorphism
- Influenza season
- Study Period
- COVID-19 impacted

Stratification factors (actual) will be used as subgroups for concomitant medication.

For the primary and the six most important secondary endpoints (i.e.: All endpoints included in the hierarchy testing) the subgroup with subgroup\*treatment interaction term will be added in the statistical analysis models, except for the study period subgroup, where the analysis will be performed separately for each individual category of the subgroup. For further details see Section 5.2.3. and Section 5.3.2. For other endpoints, the statistical analysis will be performed separately for each individual category of the subgroup.

Table 3: Subgroups with their definition

| Subgroup | Definition | Endpoints |
|---|---|---|
| Region | Based on country according to UN classification of | |
| | Geographic regions <sup>[9]</sup> : | secondary endpoints, excluding |
| | • Europe/Africa | viral kinetics endpoints) |
| | Northern-America | , |
| | Latin America and the Caribbean | |
| | Asia and Oceania | |
| Age group (years) | • 13-17 years | - Efficacy (primary and |
| rige group (years) | • 18-65 years | secondary endpoints, excluding |
| | • 66-85 years | viral kinetics endpoints) |
| | • 00-65 years | - All Safety |
| NEWS2 at screening (actual) | • 4-5 | - All Efficacy |
| 1 12 W 52 at sereening (actuar) | • ≥6 | - Viral Phenotype |
| | ● ≥0 | - Viral Genotype |
| Type of SOC at baseline | - COC: 1 1' ' C | 4.11 E.CC |
| (actual) | SOC including influenza antiviral treatment | - Viral Phenotype |
| (actual) | <ul> <li>SOC not including influenza antiviral</li> </ul> | - Viral Genotype |
| | treatment | - Safety(AE summary, AEs |
| | | and SAEs by MedDRA |
| | | system organ class and |
| | | preferred term, , influenza- |
| | | related complications, |
| | | laboratory toxicity) |
| Time (hours) from onset of | • ≤72 hours | - All Efficacy |
| influenza symptoms to first | _ | - Viral Phenotype |
| study drug intake (actual) | • >72 - 96 hours | - Viral Genotype |
| Study drug ilitake (actual) | | - Safety(AE summary, AEs |
| | | and SAEs by MedDRA |
| | | system organ class and |
| | | preferred term, , influenza- |
| | | related complications, |
| | | laboratory toxicity) |
| Time (hours) from onset of | • <48 hours | - All Efficacy |
| influenza symptoms to first | • >48 - 72 hours | - Viral Phenotype |
| study drug intake (actual) – 3 | | - Viral Genotype |
| categories | • >72 - 96 hours | - Vital Genotype |
| Influenza A subtype category | • A/H1N1 | - Primary endpoint |
| limitediza it sastype eategory | • A/H3N2 | - The six most important |
| | • Other | secondary endpoints |
| | Other | - All viral kinetics |
| | | - Viral phenotype |
| | | - Viral genotype |
| Hospitalization status | Hospitalized | - Only CM TLFs |
| 220 primite month buttus | • Outpatient | |
| Treatment extension | Extended treatment | - All Efficacy |
| Treatment extension | | - Viral Phenotype |
| | No extended treatment | - Viral Genotype |
| | | - viiai Genotype |

| Subgroup | Definition | Endpoints |
|---|---|---|
| Baseline | Polymorphism on one or any of these amino-acid | - Primary endpoint |
| polymorphism | positions of interest: | - Viral Phenotype |
| (based on | • Q306 | - Viral Genotype |
| influenza PB2 | • F323 | - Viral kinetics |
| genotype) | • S324 | |
| | • F325 | |
| | • S337 | |
| | • H357 | |
| | • F363 | |
| | • K376 | |
| | • T378 | |
| | • F404 | |
| | • Q406 | |
| | • M431 | |
| | • 2N510 | |
| Baseline Resistance (Based o | on Based on fold change (FC) in EC <sub>50</sub> for pimodivir: | - Primary endpoint |
| influenza PB2 phenotype) | • FC≤4 | - Viral Phenotype |
| 1 31 / | • FC>4 | - Viral Genotype |
| | 1074 | - Viral kinetics |
| Influenza Season | Northern Hemisphere 2017/2018 | - Efficacy (primary and the six |
| | Southern Hemisphere 2018 | most important secondary |
| | Northern Hemisphere 2018/2019 | endpoints only) |
| | Southern Hemisphere 2019 | - All viral kinetics |
| | Northern Hemisphere 2019/2020 | - Viral phenotype |
| | • Southern Hemisphere 2020 | Viral genotype |
| | and so on to capture all enrolled subjects | |
| Study period | • pre interim (subjects enrolled for the interin | -Efficacy (primary and the six |
| | analysis, i.e.: randomized before or on | most important secondary |
| | February 28, 2020) | endpoints only) |
| | <ul> <li>post interim (subjects enrolled after the</li> </ul> | -safety (Safety(AE summary, |
| | interim analysis, i.e.: randomized after | AEs and SAEs by MedDRA |
| | February 28, 2020) | system organ class and |
| | | preferred term, , influenza- |
| | | related complications, |
| COVID-19 impacted | • Voc | laboratory toxicity)) -Efficacy (primary and the six |
| CO v ID-13 IIIIpacicu | • Yes<br>• No | most important secondary |
| | • NO | endpoints only) |
| | COVID-19 impacted is based on any COVID-19 | - Safety (AE summary, AEs |
| | related AEs, COVID-19 related PD, any COVID- | and SAEs by MedDRA system |
| | 19 related treatment or study withdrawal | organ class and preferred term, |
| | j | influenza-related |
| | | complications, laboratory |
| | | toxicity) |

Subjects enrolled from 1<sup>st</sup> October 2017 to 31<sup>th</sup> March 2018 are considered to be in the Northern Hemisphere 2017/2018 category and subjects enrolled from 1<sup>st</sup> April 2018 to 30<sup>st</sup> September 2018 are considered to be in the Southern Hemisphere 2018 category. Subjects enrolled from 1<sup>st</sup> October 2018 to 31<sup>th</sup> March 2019 are considered to be in the Northern Hemisphere 2018/2019 category and subjects enrolled from 1<sup>st</sup> April 2019 to 30<sup>st</sup> September 2019 are considered to be in the Southern Hemisphere 2019 category, and so on.

Note: The six most important secondary endpoints are: incidence in post-baseline complications, time to hospital discharge, time from ICU admission to ICU discharge, time to return to daily activities, time from start of mechanical ventilation to end of mechanical ventilation, rate of rehospitalization.

Additional subgroup analysis may be specified in a separate analysis plan and reported separately from the clinical study report.

### 2.4. Study Day and Relative Day

Reference date refers to the start date of the first study drug administration. All efficacy and safety assessments at all visits will be assigned a day relative to this date.

The relative day (reldy) will be defined as:

 $reldy = visit \ date - reference \ date + 1$  for visits on or after the reference date,

*reldy* = *visit date* – *reference date* for visits before the reference date.

Consequently there is no 'day 0' defined.

## 2.5. Baseline and Endpoint

The baseline analysis visit is defined as the last assessment before the first intake of the study drug, with the possible exception for height, weight, viral load results from the central lab testing and the hospital recovery scale (HRS). Height and weight are only recorded once, at screening/baseline visit, and the values recorded at this visit will be allocated to the baseline analysis visits irrespective of start of study drug For viral load, if no measurement is available prior to first dose of study drug, then the first result from the central lab testing obtained up to and including 30 minutes after first dose of study drug will be considered as the baseline assessment and will be flagged in the analysis dataset. The baseline HRS is defined irrespective of the time of the start of study drug, and is covering the screening/baseline/day 1 visit which may be performed over two days as defined per protocol. Baseline HRS will be assigned to Day 1.

As specified in the protocol, an ECG recording within 1 calendar day before signing of the ICF/assent form can be used as baseline ECG requirement, if no ECG measurement was performed between signing ICF and first study drug intake.

For programming purposes the baseline record will be doubled in the ADAM datasets, the doubled record will be renamed with AVISIT = 'Baseline', AVISITN = 0 and will be assigned to the treatment phase.

For vital signs, NEWS2, ECG and central laboratory data the last study visit (Endpoint) is defined as the last scheduled study visit/timepoint and will be either the final study visit (day 28) or the safety follow-up visit.

For viral phenotyping, the last visit (Endpoint) is defined as the last study visit/timepoint for which an EC<sub>50</sub> and/or IC<sub>50</sub> result is available (including unscheduled visit results).

#### 2.6. Other Definitions

For FDA marketing authorization approval in the US all subjects will be included in the analysis.

The oseltamivir subset (OST subset) contains only those subjects with oseltamivir (OST) use as part of their SOC treatment. The first dose of OST may be given before the subject was randomized but should be started no later than the day of first study drug intake.

The complete analysis will be repeated restricted to the OST subset to support marketing authorization approval in EMA.

Analyses to support authorization approval in other regions or countries, will include all subjects (depending on the enrichment of the interim analysis) unless the Health Authority of the regions or country requests otherwise and may be specified in a separate analysis plan and may also be reported separately

#### 3. INTERIM ANALYSIS AND DATA MONITORING COMMITTEE REVIEW

# 3.1. Interim Analyses

An interim analyses will be performed by an independent Statistical Support Group (SSG) and will be reviewed by the Independent Data Monitoring Committee (IDMC). Only the IDMC and the SSG will be unblinded to the data. The IDMC will provide recommendations to a Sponsor Committee.

An interim analysis will be implemented to assess lack of efficacy in the subgroup with time since onset of influenza symptoms between 72 and 96 hours.

- In case lack of efficacy is concluded for the subgroup with time since onset of influenza symptoms between 72 and 96 hours:
  - Enrollment in this subgroup will be stopped
  - Sample size re-estimation will be performed based on the subgroup with time since onset of influenza symptoms ≤72 hours and consequently, the sample size of this subgroup may be increased. The maximum number of subjects that may be enrolled in this subgroup will be approximately 900.
  - Futility will be assessed in the subgroup with time since onset of influenza symptoms
     ≤72 hours based on re-estimated sample size.
  - At the final analysis, hypotheses will be evaluated in the subgroup with time since onset of influenza symptoms <72 hours.</li>
- In case no lack of efficacy is concluded for the subgroup with time since onset of influenza symptoms between 72 and 96 hours:
  - The subgroup with time since onset of influenza symptoms between 72 and 96 hours will be continued in the study.
  - Sample size re-estimation will be performed based on all subjects. The sample size may
    be increased. The maximum total number of subjects that may be enrolled in the study

will be approximately 900. The study population should consist of at least 75% of subjects with first administration of study drug  $\leq$ 72 hours since onset of influenza symptoms.

- Futility will be assessed in all subjects based on re-estimated sample size.
- At the final analysis, hypotheses will be evaluated in all subjects.

Details on the statistical decision rules will be provided in the IDMC SAP. The interim analysis will be conducted at the end of the first influenza season when between 300 and 450 subjects have been enrolled or during the season when 450 subjects have been enrolled. Further details will be specified in the IDMC charter.

### 3.2. Independent Data Monitoring Committee

An IDMC will be established to monitor data on a regular basis. The committee will meet periodically to review interim data. After the review, the IDMC will make recommendations regarding the continuation of the study. The details will be provided in a separate IDMC charter.

The IDMC will consist of at least 3 members, including one medical expert in the relevant therapeutic area and at least one statistician knowledgeable about statistical methods for clinical studies and sequential analysis of study data. One of these individuals will chair the Committee. The IDMC responsibilities, authorities, and procedures will be documented in its charter.

#### 4. SUBJECT INFORMATION

All general analyses will be done on the ITT-i Set and the Safety Set unless specified otherwise for a specific display.

# 4.1. Demographics and Baseline Characteristics

Demographics and baseline disease characteristics will also be done on the PP and ITT-ni sets.

Descriptive statistics or frequency tabulation will be provided for the following parameters.

- Demographic parameters:
  - Sex (Male, Female)
  - Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Multiple). The specification of the category 'Multiple' will only be listed. The 'Not reported category' will not be added for the denominator.
  - Ethnicity (Hispanic or Latino, Not Hispanic or Latino)
  - Country
  - Geographic region (Based on country according to UN classification of Geographic regions<sup>[9]</sup>: Europe/Africa, Northern-America, Latin America and the Caribbean, Asia and Oceania)
  - Age (years and categories: 13-17 years [ $\geq$ 13 <18], 18-65 years [ $\geq$ 18  $\leq$ 65], 66-85 years [>65  $\leq$ 85])
  - Age (years and categories: Adolescents (12-17 years) [≥12 ≤17], Adults (18-64 years) [≥18 ≤64], From 65 to 84 years [≥65 ≤84], 85 years and over [≥85])
  - Weight at baseline (kg)
  - Height at baseline (cm)
  - BMI at baseline = Weight at baseline (kg) / (Height at baseline (m))<sup>2</sup> (rounded to 1 decimal. Although available in the raw data, BMI will be recalculated from last weight and height measurement before start of treatment)
  - Current Tobacco use: tobacco, cigarettes, cigars, patches/gum, pipes, E-cigarettes or equivalent, smokeless tobacco (Yes, No, Missing). Note that 'No' also includes exsmokers.
  - Childbearing potential (only listed)
- Baseline disease characteristics:
  - Influenza A subtype category (A/H1N1, A/H3N2, No subtype)
  - Baseline influenza A viral load (log<sub>10</sub> vp/mL), assessed by qRT-PCR
  - Baseline influenza A viral titer (log<sub>10</sub> TCID<sub>50</sub>/mL) assessed by viral culture

- qRT-PCR negativity at baseline
- Viral culture negativity at baseline
- Broad respiratory panel (show the reported pathogen)
- Return to daily activities at baseline
- Patient Global Impression of Severity of Influenza symptoms at baseline
- EQ-5D VAS at baseline
- EQ-5D Valuation index at baseline
- NEW2 Score at screening (4-5, >=6), as randomized
- NEW2 Score at screening (4-5, >=6), actual
- Hospital recovery scale category at baseline
- Fundamental hospital recovery scale category at baseline
- Respiration rate at baseline (breaths/min)
- Arterial oxygen saturation at baseline on room air (%)
- Arterial oxygen saturation at baseline overall (%)
- Supplemental oxygen at baseline (yes, no) (following supplemental oxygen types are considered: nasal cannula, venturi mask, simple face mask and nonrebreathing face mask with reservoir and one way valve)
- Mechanical ventilation use at baseline (yes, no)
- Temperature (°C) at baseline
- Systolic blood pressure at baseline (mmHg)
- Heart rate at baseline (beats/min)
- Level of consciousness at baseline
- Time since onset of influenza symptoms as randomized ( $\leq$ 72,  $\geq$ 72 hours),
- Time since onset of influenza symptoms, actual time (hours) [the actual time will be calculated from start date and time of acute respiratory symptoms until datetime of first study drug intake, if the time is missing, the midpoint of the time interval as recorded per CRF will be used.]
- Time since onset of influenza symptoms, actual ( $\leq 72$ ,  $\geq 72$  hours)
- Time since onset of influenza symptoms, actual − 3 categories (≤48, >48 − 72h, >72 hours)
- Type of SOC at baseline, as randomized (including or not including influenza antiviral treatment)
- Type of SOC at baseline, actual (including or not including influenza antiviral treatment), for the SOC including antiviral treatment the influenza antiviral will also be shown

- SOC including oseltamivir (yes, no)
- Chronic oxygen use(yes, no)
- Primary reason for hospitalization at baseline (prioritize influenza in case >=2 reasons are selected, then adverse event and then medical history)
- Type of influenza A diagnostic assay (Rapid antigen-based diagnostic test, Rapid molecular diagnostic test)
- In ICU at baseline (yes, no)
- Baseline resistance
- Any baseline polymorphism

### 4.2. Disposition Information

Summaries will be provided for the following disposition information:

- Number of subjects screened, screening failures, randomized, randomized and not treated, randomized and/or treated, randomized and treated, randomized and no confirmed Influenza A, ITT-i set, ITT-ni set, per protocol set, and safety set. The planned treatment arm will be shown, except for the randomized and/or treated and safety sets where the actual treatment will be shown. The number (%) of subjects impacted by the COVID-19 pandemic will be presented for the ITT-i, ITT-ni, per protocol and safety analysis sets.
- Number of subjects who completed/discontinued treatment and/or the trial, with the reasons of discontinuation. The number of subjects that discontinued due to an AE that is related to COVID-19 and that discontinued due to another reason related to COVID -19 will be added.
- Kaplan-Meier curves of the time to completion or discontinuation (in days) of the treatment/trial per treatment group, overall and separately for subjects with/ without treatment extension. Note at the final analysis all subjects will have the event of completion or discontinuation and no subjects will be censored.
- Number of subjects with a visit at each scheduled analysis timepoint by phase and the missing visits and visits different from planned due to COVID-19 per phase.
- Number of subjects enrolled per month, quarter, season and year.

### 4.3. Treatment Compliance

Treatment compliance for pimodivir/placebo is calculated as the actual number of doses taken, as a percentage of the planned number of doses. The actual number of doses taken will be derived from the drug accountability information (DA domain) as the amount of drug dispensed minus the returned amount (in case both amounts are known, otherwise treatment compliance will be missing)

To differentiate between the compliance during the planned treatment subperiod and the planned treatment extension subperiod, the date of dispensing the tablets will be compared with the treatment extension start date (DS Domain). If the drug is dispensed before the treatment extension

start date it will be used for the compliance of the treatment subperiod. If the drug is dispensed on or after the treatment extension start date the amount will be used for the compliance of the treatment extension subperiod.

For placebo or pimodivir the actual number of doses needs to be divided by 2 as the study uses 300 mg tablets. For subjects without treatment extension the planned number of study drug is 20 tablets of placebo or pimodivir hence the planned number of doses per study drug equals 10 doses. For subjects with treatment extension the planned dose is doubled. Note that the planned number of doses is irrespective of whether the subject discontinued during the treatment phase.

Dosing compliance will be summarized descriptively in the treatment phase and per subperiod and by discontinuing the trial during the treatment period (Yes, No).

### 4.4. Extent of Exposure

The extent of exposure (hours) is defined as datetime of last study drug intake – datetime of first study drug intake + 12 hours. Note: treatment interruptions will not be taken into account.

Extent of exposure will be summarized descriptively in the treatment phase, overall and by treatment subperiod.

A listing will be made to present the exposure to study drug for subjects impacted by COVID-19 (based on reason 'Other' containing 'COVID').

#### 4.5. Protocol Deviations

The number and percentage of subjects with major protocol deviations will be tabulated overall and per coded major protocol deviation.

A listing will be made of all major protocol deviations for the subjects in the safety set.

Additionally, a listing of major and separately a listing for minor protocol deviations related to COVID-19 will be made.

Additionally, for subjects in the ITT-i set, the number and percentage of subjects with a reason for exclusion from the per protocol set will be tabulated overall and for each reason for exclusion.(see Section 2.2.2.2).

A listing will also be made of all reasons for exclusion from the per protocol set for subjects in the ITT-i set.

#### 4.6. Prior and Concomitant Medications

Medications reported from 7 days before first dose of study drug and up to last contact date will be summarized by preferred term using the World Health Organization-Drug Dictionary for the ITT-i Set and the Safety Set as frequency tables in 2 parts:

- 1. Prior medication: medication that started before the first dose of study drug, regardless of when dosing of the medication ended
- 2. Concomitant medication: medication received at or after the first dose of study drug, medication that was received before initial dosing and continued after initial dosing of study drug, or medication with missing stop date.

(Medication that started before the first dose of study drug and continued after the first dose of study drug will be summarized as prior medication and separately as concomitant medication.)

A frequency tabulation of concomitant medication will be shown by ATC class level up to level 3. Frequency tabulations will be made for concomitant antibiotics, type of SOC, corticosteroids, and medication administered to treat COVID-19 infection by ATC class and by hospitalization status. Additionally, tabulations will be made of concomitant corticosteroids and antibiotics administered because of adverse events reported as influenza complications.

The ATC level 2 code J01 will be used to identify concomitant antibiotics.

The ATC level 2 code H02 and the ATC level 4 codes M01BA, R03BA, and R03AK will be used for identifying corticosteroids. Separate frequency tabulations will be made for antipyretic medication and oxygen supplementation. The ATC level 4 codes N02BA and N02BE and the generic medication names paracetamol, ibuprofen, and acetylsalicylic acid will be used to identify antipyretic medications. The table showing oxygen supplementation will be tabulated per analysis visit, phase and treatment subperiod. If a prior/concomitant therapy record misses components of its start and/or stop dates (time and/or day and/or month and/or year), the following actions will be taken:

- 1. In case of partial start or stop datetimes, the concomitant therapy records will be allocated to prior and/or concomitant using the available partial information, without imputations.
- 2. In case of a completely missing start date, the prior and/or concomitant therapy will be considered as having started before the trial.
- 3. In case of a completely missing end date, the prior and/or concomitant therapy will be considered as ongoing at the end of the trial.

# 4.7. Medical history

The influenza vaccination status will be tabulated by:

- Vaccinated in previous season, not in current season
- Vaccinated in current season, not in previous season
- Vaccinated in previous and current season.
- Not vaccinated in previous and current season

The use of antiviral influenza medication prior to study drug initiation will be tabulated separately.

Influenza history will be listed, including information on first acute respiratory symptoms, influenza vaccination status, chronic oxygen use and previous antiviral influenza therapy. Pretreatment influenza complications will also be listed.

Other medical history will be tabulated by subcategory and/or will be listed.

#### 5. EFFICACY

Descriptive statistics will be used for all efficacy endpoints and will be tabulated by treatment arm and stratification factors (NEWS2 at screening, baseline SOC and time since onset of symptoms). For the analyses restricted to subjects who received OST as part of their SOC, type of baseline SOC will not be included as a stratification factor or model parameter.

## 5.1. Analysis Specifications

### 5.1.1. Level of Significance

The population used for the evaluation at the final analysis will depend on the outcome scenario of the interim analysis: i.e.; scenario 1: continue with the full study population or scenario 2: continue only with the subjects with an onset of symptoms less than 72 hours before first study drug intake. Tables/graphs/listings will account for the selected scenario.

As a confirmatory strategy, to account for multiplicity in the statistical evaluation of the most important efficacy endpoints, in either scenario, a combination of hierarchical testing and the Bonferroni-Holm testing procedure will be applied to control for the overall Type I error rate at the 5% level. The following endpoints are included in the confirmatory strategy:

- 1. Hospital recovery scale at Day 6, ie, primary endpoint
- 2. Incidence in post-baseline complications
- 3. Time to hospital discharge
- 4. Time from ICU admission to ICU discharge
- 5. Time to return to daily activities
- 6. Time from start of mechanical ventilation to end of mechanical ventilation
- 7. Rate of re-hospitalization

First, the primary endpoint will be tested for superiority of pimodivir in combination with SOC over placebo in combination with SOC at the 2-sided 5% significance level.

The confirmatory test procedure follows the Serial Gate Keeping strategy as outlined in Section 7 of the FDA's draft guidance on Multiple Endpoints to control the overall type I error at the 5% 2-sided level. The primary and six most important secondary endpoints (listed above) will be tested in the hierarchical order per the 5 steps outlined below. All alphas and p-values specified are 2-sided.

Step 1: Test the primary hypothesis ("Hospital recovery scale at Day 6")

- If the p-value is  $\leq 5\%$ , continue to Step 2.
- If the p-value is >5%, stop testing, and no claim will be made.

Step 2: Test first set of 2 secondary endpoints ("Incidence in post-baseline complications" and "Time from start of study drug to hospital discharge"). The Bonferroni-Holm procedure will be applied to control the type I error within Step 2.

- If the smallest of the 2 p-values is ≤2.5% and the largest of the 2 p-values is ≤5%, continue to Step 3.
- If the p-value for "Incidence in post-baseline complications" is ≤2.5% but the p-value for "Time from start of study drug to hospital discharge" is >5%, stop further testing of the secondary endpoints, and make a claim on "Hospital recovery scale at Day 6" and "Incidence in post-baseline complications".
- If the p-value for "Time from start of study drug to hospital discharge" is ≤2.5% but the p-value for "Incidence in post-baseline complications" is >5%, stop further testing of the secondary endpoints, and make a claim on "Hospital recovery scale at Day 6" and "Time from start of study drug to hospital discharge".
- If the smallest of the 2 p-values is >2.5%, stop further testing of the secondary endpoints, and make a claim on "Hospital recovery scale at Day 6" only.

<u>Step 3</u>: Test second set of 2 secondary endpoints ("Time from ICU admission to ICU discharge" and "Time to return to daily activities"). The Bonferroni-Holm procedure will be applied within Step 3.

- If the smallest of the 2 p-values is ≤2.5% and the largest of the 2 p-values is ≤5%, continue to Step 4.
- If the p-value for "Time from ICU admission to ICU discharge" is ≤2.5% but the pvalue for "Time to return to daily activities" is >5%, stop further testing of the secondary endpoints, and make a claim on "Hospital recovery scale at Day 6", "Incidence in post-baseline complications", "Time from start of study drug to hospital discharge" and "Time from ICU admission to ICU discharge".
- If the p-value for "Time to return to daily activities" is ≤2.5% but the p-value for "Time from ICU admission to ICU discharge" is >5%, stop further testing of the secondary endpoints, and make a claim on "Hospital recovery scale at Day 6", "Incidence in postbaseline complications", "Time from start of study drug to hospital discharge" and "Time to return to daily activities".
- If the smallest of the 2 p-values is >2.5%, stop further testing of the secondary endpoints, and make a claim on "Hospital recovery scale at Day 6", "Incidence in postbaseline complications" and "Time from start of study drug to hospital discharge".

<u>Step 4</u>: Test the fifth secondary endpoint ("Time from start to end of mechanical ventilation")

- If the p-value is  $\leq 5\%$ , continue to Step 6.
- If the p-value is >5%, stop further testing of the secondary endpoints, and make a claim on "Hospital recovery scale at Day 6", "Incidence in post-baseline complications", "Time from start of study drug to hospital discharge", "Time from ICU admission to ICU discharge", and "Time to return to daily activities".

Step 5: Test the sixth secondary endpoint ("Rate of re-hospitalization")

• If the p-value is ≤5%, make a claim on "Hospital recovery scale at Day 6", "Incidence in post-baseline complications", "Time from start of study drug to hospital discharge", "Time

- from ICU admission to ICU discharge", "Time to return to daily activities", "Time from start to end of mechanical ventilation", and "Rate of re-hospitalization".
- If the p-value is >5%, make a claim on "Hospital recovery scale at Day 6", "Incidence in post-baseline complications", "Time from start of study drug to hospital discharge", "Time from ICU admission to ICU discharge", "Time to return to daily activities", and "Time from start to end of mechanical ventilation".

For the primary endpoint, the results from the proportional odds model will be used in the hypothesis testing. If the proportional odds assumption would not hold on the treatment effect, the p-value from the van Elteren test will be used. For the secondary endpoints time from start of study drug to hospital discharge, time from ICU admission to ICU discharge, time to return to daily activities, and time from start to end of mechanical ventilation, the results of the Gehan-Wilcoxon test will be used in the hypothesis testing. For incidence in post-baseline complications and rate of re-hospitalization the results of the logistic regression will be used. For all these evaluations p-value combination tests will be used, as described below.

The final analysis on the ITT-i set (to support FDA marketing approval) and the final analysis on the OST subset (to support marketing authorization approval in EMA) will be performed independently, using a 5% two-sided significance level for each.

# 5.1.2. Statistical Methodology for Evaluation at the Final Analysis

All p-values below are one-sided p-values, to evaluate rejection of the null hypothesis that pimodivir is not better than placebo.

<u>Scenario 1</u>: The final analysis will be performed in the subgroup with time between onset of symptoms and start of treatment between 0 and 72 hours only. P-values for the final analysis will be based on 2 inverse-normal combination tests of p-values as outlined below.

Let:

p = p-value (one-sided) from full study population of the pre-interim' category of the study period subgroup

p-value (one-sided) from subgroup with time between onset of symptoms and start treatment between 0 and 72 hours of the pre-interim' category of the study period subgroup

 $p_2 = 2*\min(p,p_1)$ 

q<sub>1</sub> = p-value (one-sided), from subgroup with time between onset of symptoms and start treatment between 0 and 72 hours on the patients enrolled of the 'post-interim' category of the study period subgroup

N<sub>1</sub> = actual sample size at interim i.e.:all randomized subjects analysis set (RAND) included in the IA

N = 600, the initially planned study sample size

 $w_1 = sqrt(N_1/N)$ 

 $w_2 = \operatorname{sqrt}(1-(N_1/N))$ 

 $\varphi^{-1}(x)$  = the inverse of the standard normal cumulative distribution function in x

Note:  $p_1$  and  $q_1$  are based on a subset of subjects with onset of symptoms and start treatment between 0 and 72 hours, and therefore this stratification factor is not included in the respective models.

The p-values resulting from the following 2 combination tests both should be below the prespecified alpha (2.5% one-sided) to claim superiority in subgroup with time between onset of symptoms and start of treatment between 0 and 72 hours:

1-
$$\varphi$$
(C(p<sub>1</sub>,q<sub>1</sub>)) where C(p<sub>1</sub>,q<sub>1</sub>) = w<sub>1</sub> \*  $\varphi$ <sup>-1</sup>(1-p<sub>1</sub>) + w<sub>2</sub> \*  $\varphi$ <sup>-1</sup>(1-q<sub>1</sub>)  
1- $\varphi$ (C(p<sub>2</sub>,q<sub>1</sub>)) where C(p<sub>2</sub>,q<sub>1</sub>) = w<sub>1</sub> \*  $\varphi$ <sup>-1</sup>(1-p<sub>2</sub>) + w<sub>2</sub> \*  $\varphi$ <sup>-1</sup>(1-q<sub>1</sub>)

<u>Scenario 2</u>: The final analysis will be performed in the full study population. P-values for the final analysis will be based on 2 inverse-normal combination tests of p-values.

Let additionally:

q = p-value from full study population on the patients enrolled of the 'post-interim' category of the study period subgroup

The p-values resulting from the following 2 combination tests both should be below the prespecified alpha to claim superiority in the full study population:

$$\begin{split} &1\text{-}\phi(C(p,q)) \text{ where } C(p,q) &= w_1 * \phi^{\text{-}1}(1\text{-}p) + w_2 * \phi^{\text{-}1}(1\text{-}q) \\ &1\text{-}\phi(C(p_2,q)) \text{ where } C(p_2,q) = w_1 * \phi^{\text{-}1}(1\text{-}p_2) + w_2 * \phi^{\text{-}1}(1\text{-}q) \end{split}$$

# 5.1.3. Data Handling Rules

For analysis purposes the  $log_{10}$  qRT-PCR viral load will be imputed with 2.12 when the result is 'TARGET DETECTED' (i.e. below the limit of quantification: <2.18) and with 2.05 if result is
'TARGET NOT DETECTED' (i.e. below limit of detection: <2.05). The log<sub>10</sub> TCID<sub>50</sub> viral titer will be imputed with 0.74 when the result is '<0.75' (below limit of quantification).

#### 5.1.4. Stratification Factors

The actual values of the stratification factors will be used for all analyses.

The concomitant medications indicated as standard-of-care treatment on the concomitant medication form will be used for determining the actual strata for type of baseline SOC. If no influenza antiviral is recorded it will be assumed that the subject received SOC not including influenza antiviral. The following ATC level 4 code and generic medication names indicate an influenza antiviral:

- J05AH (including neuraminidase inhibitors)
- Laninamivir
- Umifenovir
- Amantadine
- Rimantadine
- Ribavirin
- Baloxavir Marboxil

The datetime when first acute respiratory symptoms appeared and the datetime of first dose of study drug will be used for determining the actual strata for time since symptom onset relative to treatment initiation.

The actual NEWS2 will be calculated as explained in Section 7.6. Note that a subject is considered to receive supplemental oxygen if the subject received oxygen according to the CM dataset at least at one point between 15 min before randomization date time to the randomization date time.

When an incorrect stratification occurred for the NEWS(2) such that the actual NEWS2 is lower than 4 or for the time to onset of symptoms to first study drug intake (i.e.: >96 hours) then use the randomized stratification category instead. Similarly, in case of missing data to calculate the actual NEWS2 stratification the randomized stratification factor will be used, except if the NEWS2 is greater or equal to 6 based on the available non-missing parameters, then the actual stratification will be '6 or more'.

There will be no missing stratification factors values for randomized subjects receiving study drug.

# 5.2. Primary Efficacy Endpoint(s)

#### 5.2.1. Definition

The primary efficacy analysis will be based on the ITT-i analysis set and consists of the analysis of the hospital recovery scale outcome on Day 6.

The hospital recovery scale provides 6 mutually exclusive conditions ordered from best to worst, and the score reflects the subject's worst situation on the day of assessment:

- 1. Not hospitalized
- 2. Non-ICU hospitalization, not requiring supplemental oxygen
- 3. Non-ICU hospitalization, requiring supplemental oxygen
- 4. Admitted to the ICU, not requiring invasive mechanical ventilation
- 5. Requiring invasive mechanical ventilation
- 6. Death

The hospital recovery scale categories are defined below. For ease of categorization, the categories are defined from worst to best. A subject will be evaluated in the same ordering of the categories as below. Once a subject fulfils the criteria for a category, the category is assigned to the subject and the evaluation stops.

#### 6. Death

- Subject died at any time on the day of assessment or earlier (all-cause mortality).
- 5. Requiring invasive mechanical ventilation
  - Any oxygen support requiring intubation or extracorporeal oxygenation
  - Invasive mechanical ventilation is used at any time on the day of assessment.
- 4. Admitted to the ICU, not requiring invasive mechanical ventilation

Subject met either of the 2 following criteria:

- In the ICU (and ICU level of care is required during the day of assessment)
- On the hospital ward, with or without supplemental oxygen, but deemed to require ICU level of care at any time during the day of assessment (e.g., not transferred to ICU due to bed availability)

Requiring ICU level of care is defined by:

- Some specific conditions:
- o Treatment of acute unstable arrhythmias
- o Treatment of complicated acid-base or electrolyte imbalances
- o Large volume resuscitation
- Utilization of intravenous vasoactive medications
- o S/P cardiac arrest
- Cardiogenic Shock
- Acute myocardial infarct with complications
- Cardiac tamponade
- Acute congestive heart failure
- o Acute or imminent respiratory failure
- Hemodynamic instability

- O Diabetic ketoacidosis complicated by hemodynamic instability, altered mental status, respiratory insufficiency, or severe acidosis
- Other conditions requiring specialized equipment and/or staff competencies only available in the ICU
- 3. Non-ICU hospitalization, requiring supplemental oxygen

Subject met either of the 2 following criteria:

- Non-ICU hospitalized on the day of assessment (including readmittance), not ready for discharge during the whole day of assessment, as judged by the investigator and supplemental oxygen is required by the subject
- In the ICU but there is no medical reason to be in the ICU during the day of assessment, and supplemental oxygen is required by the subject

Requiring supplemental oxygen is defined by:

- Receiving supplemental oxygen through a face mask or nasal cannula and not being able to sustain a blood oxygen saturation of ≥94% when breathing room air for 15 minutes at any time on the day of assessment.
- If supplemental oxygen was provided chronically pre-influenza infection (based on medical history), that amount of supplemental oxygen is exceeded to prevent hypoxia, tachypnea or dyspnea at some point on the day of assessment.
- Not receiving supplemental oxygen and either:
  - O Having a blood oxygen saturation of <94% when breathing room air for 15 minutes at any measurement on the day of assessment, or
  - O In case of known pre-influenza SpO<sub>2</sub> <94% (e.g., due to COPD), the current blood oxygen saturation on room air is lower than pre-influenza infection levels by at least 3%.
- 2. Non-ICU hospitalization, not requiring supplemental oxygen

Subject met either of the 2 following criteria:

- Non-ICU hospitalized on the day of assessment (including readmittance) and not ready for discharge during the whole day of assessment, as judged by the investigator
- In the ICU but there is no medical reason to be in the ICU during the day of assessment
- 1. Not hospitalized

Any of the following:

- Discharged from the hospital before the day of assessment
- Hospitalized at the day of assessment but ready for discharge on both the day of assessment and the day prior, as judged by the investigator (e.g., in case of lack of bed availability in a skilled nursing facility, lack of social support at home).

Notes: If a subject was discharged from the hospital "Against Medical Advice" on the day prior to the day of assessment, the subject will be considered as hospitalized (evaluating the other aspects of the HRS to define the correct category based on available data, e.g.: requiring supplemental oxygen, on the day of assessment). The hospital recovery scale category will be considered missing on subsequent days.

The HRS will be missing after a subject withdrew (except for withdrawal due to death) from the study.

See Attachment 6 for details of the derivation of the HRS categories.

#### 5.2.2. Estimand

The population of interest is hospitalized subjects between 13 to 85 years old with a confirmed influenza A infection.

The primary variable is the hospital recovery scale as assessed on Day 6 and will be compared between pimodivir and placebo on top of SOC. The hospital recovery scale is an ordinal mutually exclusive scale of six categories (death, requiring mechanical ventilation, requiring ICU, non-ICU hospitalized requiring supplemental oxygen, non-ICU hospitalized not requiring supplemental oxygen and non-hospitalized).

The intercurrent event of the use of influenza antivirals as part of SOC is handled in a treatment policy strategy as the primary endpoint is derived in the same way irrespective of the components of SOC. Treatment discontinuation is an intercurrent event that is also handled in a treatment policy strategy. Death as intercurrent event is handled in a composite strategy as it is one of the categories of the HRS. Other factors as for example bed availability that can influence the status of the subject are intercurrent events that are also handled with the composite strategy as the HRS accounts for the status of where the subject 'should be' instead of where the subject physically is.

The common odds ratio estimated by a proportional odds model is used as the population-level summary. If the assumption (by testing the parallel slopes for the treatment effect only) of the proportional odds would not hold for the treatment effect, the Van Elteren test will be used in a sensitivity analysis and the resulting p-value would be used in the formal testing. A second sensitivity analysis is conducted to handle missing data by an MAR/MNAR multiple imputations method. This is done for all missing HRS values on day 6 and separately for HRS values on day 6 that are missing due to COVID-19 and for HRS values that are missing not due to COVID-19.

#### 5.2.3. Analysis Methods

A proportional odds model will be used as primary model to analyze the hospital recovery scale on Day 6, modeling the common odds ratio of improvement on the ordinal scale of active treatment versus placebo. The model will include treatment, hospital recovery scale category at baseline and the stratification factors (NEWS2 category at screening, type of baseline SOC, and time since onset of influenza symptoms). In a first step equal slopes (i.e. proportional odds) for the treatment effect only and unequal slopes for the other covariates, will be modeled. If this model does not fit a full

proportional odds model will be applied, i.e. implying proportional odds for all covariates in the model. The common odds ratio from the final model will be considered as the estimate of the treatment effect. The actual values of the stratification factors will be used for all models, not as randomized. The proportional odds model will be defined in such a way that a common odds ratio smaller than 1 indicates larger improvement in the pimodivir treatment group.

Graphical displays and tabulations will be provided showing the proportion of subjects per hospital recovery scale category and day. Also, shift tabulations will be provided of the baseline hospital recovery scale category versus the post-baseline hospital recovery scale category, per day.

The proportional odds assumption will be assessed by testing for parallel slopes for the treatment effect only.

In addition, each of 5 dichotomizations of the hospital recovery scale, ie,

- Not hospitalized, vs worse (ie, hospitalized)
- Non-ICU hospitalized without supplemental oxygen (or better), vs worse
- Non-ICU hospitalized with supplemental oxygen (or better), vs worse
- In the ICU without invasive mechanical ventilation (or better), vs worse
- Invasive mechanical ventilation (or better), vs worse (ie, died)

will be analyzed using a logistic regression model, including treatment, hospital recovery scale category at baseline and stratification factors.

The hospital recovery scale will also be analyzed using the Van Elteren test with strata defined by the stratification factors<sup>[3, 6]</sup>.

A table will be created showing the number (%) missing HRS values at day 6 overall and by reason: study discontinuation: due to COVID-19 and not due to COVID-19, discharged against medical advice prior to day 5 and subjects that have no confirmed influenza A.

In case of more than 10% missing data on Day 6: multiple imputation will be employed as sensitivity analyses for the proportional odds model of the HRS (excluding the subgroup analyses), under the missing-at-random (MAR) assumption and missing-not-at-random (NMAR) assumption.

- If more than 5% of the patients have a missing HRS value due to COVID-19 (i.e.: discontinued due to COVID-19), the multiple imputation method will also be done separately on these subjects.
- If more than 5% of the patients have a missing HRS values unrelated to COVID-19, then also multiple imputation will be done separately in this group.

The Markov Chain Monte Carlo (MCMC) method will be used to create a number of multiple imputation datasets with monotone missingness in the clinical outcomes (baseline until Day 14). The number of imputation datasets will be the same as the percentage of missing data<sup>[10]</sup>. For MAR assumptions, a monotone ordinal logistic regression imputation model will be used to complete the remaining missing clinical outcomes.

For the NMAR assumption, the imputed datasets obtained from the MAR assumption described above will be used, but with a structural shift in hospital recovery scale category on Day 6 of the imputed values, to introduce non-ignorable missing patterns:

- To reflect missingness patterns as a result of study discontinuation due to a dissatisfying treatment effect or safety issues in the placebo treatment group, the following shifts will be applied in the placebo treatment group only:
  - o 1 category down, eg, from '1. Not hospitalized' to '2. Non-ICU hospitalization, not requiring supplemental oxygen'
  - o 2 categories down, eg, from '1. Not hospitalized' to '3. Non-ICU hospitalization, requiring supplemental oxygen'
- To reflect missingness patterns as a result of study discontinuation due to a dissatisfying treatment effect or safety issues in the pimodivir treatment group, the following shifts will be applied in the pimodivir treatment group only:
  - o 1 category down, eg, from '1. Not hospitalized' to '2. Non-ICU hospitalization, not requiring supplemental oxygen'
  - o 2 categories down, eg, from '1. Not hospitalized' to '3. Non-ICU hospitalization, requiring supplemental oxygen'

In all cases, '6. Death' will be the worst hospital recovery scale category after imputation and structural shift and '1 Not hospitalized' will be the best hospital recovery category after imputation and structural shift.

The models fitted using the multiple imputation datasets will be the same as the final model on the actual data. The results from the models on the multiple imputation datasets will be combined taking into account the between and within variation of the results.

The analyses on the primary endpoint will be repeated by subgroups for efficacy as defined in Section 2.3. The final model above will be repeated adding these subgroups (defined in Section 2.3) as an additional covariate and interaction with treatment. Per subgroup the common odds ratio and the odds ratios calculated for the dichotomizations will be derived from these models. In addition, for each category in a subgroup, the Van Elteren test with strata defined by the stratification factors will be repeated.

# 5.3. Major Secondary Endpoints

#### 5.3.1. Definition

Formulae to be used for derived variables, including data conversions, are provided in the tables below.

Note that for time-to event variables the actual date or times that the endpoint is met will be used. For the time-to-event variables, in case of death prior to the event, the subject will be censored using a time-to equal to the maximum time across all subjects.

# 5.3.1.1. Clinical Outcome

| Measurement | Formula |
|---|---|
| Time to hospital discharge (hours) [Time-to event] | The time from first study drug intake to first hospital discharge (=event) in hours. Note this excludes time in hospital because of rehospitalization (a new hospitalization is considered as a rehospitalization if there is at least 1 day in between the start date of the new hospitalization and the end date of the previous hospitalization) and hospitalizations that ended before first intake. |
| | Subjects who complete or withdraw from the study while still hospitalized will be censored at the date of completion or withdrawal. If the time is not available they will be censored at 23:59. |
| | If time of end of hospitalization is not known but we have a date of discharge then time will be imputed at 23:59. |
| | (Date and time of event or censoring— date and time of first dose of study drug)/3600, rounded to one decimal. |
| Time to readiness for | The time from first study drug intake until the time to readiness for |
| hospital discharge<br>(days) [Time-to event] | hospital discharge (= event) in days, with readiness for hospital discharge defined by the investigator. In case at the date of discharge the subject is not ready to be discharged as per investigator assessment, the discharge readiness day will be set to the next day. |
| | Censoring of the time will be done analogous to "Time to hospital discharge", only using the date information, as time is not available for the event. |
| Total length of hospital stay (hours) [Duration] | The total number of hours a subject stayed in the hospital during the period from first study drug intake until study termination, calculated as sum of [(end date and time of hospitalization— start date and time of first intake)/3600], rounded to one decimal for all separate hospital stays per subject. If the time is not available it will be put at 23:59 |
| | If hospitalization started before first study drug intake, then datetime of first study drug will be used. |
| | If hospitalization is still ongoing at study end, the end date and time will be imputed by the end date and time of the last phase as defined in table 1. |

| ICU admission started post-baseline | Incidence of post-baseline ICU admission - Admitted to ICU post-baseline - Not admitted to ICU post-baseline Note: In case a patient is in the ICU at baseline and (after discharge from the ICU) the patient is re-admitted post-baseline, this subject will be counted as "Admitted to ICU post-baseline". |
|---|---|
| First admission to intensive care unit | When was the subject first admitted to the ICU during the study? |
| (ICU) | Categories: - In ICU at baseline - Admitted in ICU Post-baseline - Never admitted to ICU |
| Time from ICU admission to ICU discharge (hours) [Time-to event] | The time from max(first admission to ICU, first study drug intake) until the time of first discharge from the ICU. Censoring and calculation of the time will be done analogous to "Time to hospital discharge". Only subjects admitted to the ICU (at any point during the trial) are included in the analysis and analysis is restricted to the first ICU |
| Time from ICU admission requiredness to ICU discharge readiness (days) [Time-to event] | admission. The date from max(requiring ICU level of care, first study drug intake) until the date of not requiring ICU anymore(= event), requiring ICU level of care to be defined by the investigator. Censoring and calculation of the time (days) will be done analogous to "Time to hospital discharge" Subjects that do not require ICU level of care will be excluded from this analysis and this analysis is restricted to the first required ICU level of care. |

| Total time in intensive care unit (ICU) stay (hours) [Duration] The total number of hours a subject stayed in ICU during the period from first intake until study termination, calculated as sum of [(end date and time of discharge—start date and time of admission)/3600], rounded to one decimal for all separate events per subject In case ICU admission took place before first intake or in case the start date time of ICU is missing, then the date and time of first intake will be used. In case the ICU stay ended after the end of the trial or in case the end date time of ICU stay is missing, then the end datetime of last contact date will be used. If time of the start of ICU admission is missing then use 00:00. If time of the end of ICU admission is missing then use 02:359. The derivation of total time in ICU is analogous to "total length of hospital stay". Type of supplemental oxygen administration Tabulation will be done as collected per CRF page "Oxygen Supplementation". In addition, the following categorization will be done: - Invasive Mechanical Ventilation - Non-Invasive Mechanical Ventilation - Non-Invasive Mechanical Ventilation - Non-Invasive Mechanical Ventilation (invasive or non-invasive) Categories: - Mechanical ventilation of mechanical ventilation post-baseline - First administration of mechanical ventilation (invasive or non-invasive) Started post-baseline - Not started post-baseline mechanical ventilation is initiated post-baseline, this subject will be counted as started post-baseline. | | |
|---|---|---|
| datetime of ICU is missing, then the date and time of first intake will be used. In case the ICU stay ended after the end of the trial or in case the end datetime of ICU stay is missing, then the end datetime of last contact date will be used. If time of the start of ICU admission is missing then use 00:00. If time of the end of ICU admission is missing then use 23:59. The derivation of total time in ICU is analogous to "total length of hospital stay". Type of supplemental oxygen administration Tabulation will be done as collected per CRF page "Oxygen Supplementation". In addition, the following categorization will be done: - Invasive Mechanical Ventilation - Non-Invasive Mechanical Ventilation - None Mechanical ventilation - None Mechanical ventilation (invasive or non-invasive) Categories: - Mechanical ventilation of mechanical ventilation post-baseline - No administration of mechanical ventilation Incidence of post-baseline - Not started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | care unit (ICU) stay | from first intake until study termination, calculated as sum of [(end date and time of discharge— start date and time of admission)/3600], |
| datetime of ICU stay is missing, then the end datetime of last contact date will be used. If time of the start of ICU admission is missing then use 00:00. If time of the end of ICU admission is missing then use 23:59. The derivation of total time in ICU is analogous to "total length of hospital stay". Type of supplemental oxygen administration Tabulation will be done as collected per CRF page "Oxygen Supplementation". In addition, the following categorization will be done: - Invasive Mechanical Ventilation - Non-Invasive Mechanical Ventilation - Non-Invasive, Non-mechanical Ventilation - None Mechanical ventilation during study Incidence of mechanical ventilation (invasive or non-invasive) Categories: - Mechanical ventilation at baseline - First administration of mechanical ventilation post-baseline - No administration of mechanical ventilation (invasive or non-invasive) Mechanical ventilation - Not started post-baseline - Not started post-baseline - Not started post-baseline - Not started post-baseline - Not started post-baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | | datetime of ICU is missing, then the date and time of first intake will |
| of the end of ICU admission is missing then use 23:59. The derivation of total time in ICU is analogous to "total length of hospital stay". Type of supplemental oxygen administration Tabulation will be done as collected per CRF page "Oxygen Supplementation". In addition, the following categorization will be done: - Invasive Mechanical Ventilation - Non-Invasive Mechanical Ventilation - Non-Invasive, Non-mechanical Ventilation - None Mechanical ventilation during study Incidence of mechanical ventilation (invasive or non-invasive) Categories: - Mechanical ventilation at baseline - First administration of mechanical ventilation post-baseline - No administration of mechanical ventilation Incidence of post-baseline mechanical ventilation (invasive or non-invasive) - Started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | | datetime of ICU stay is missing, then the end datetime of last contact |
| oxygen administration Supplementation". In addition, the following categorization will be done: - Invasive Mechanical Ventilation - Non-Invasive Mechanical Ventilation - Non-Invasive, Non-mechanical Ventilation - None Mechanical ventilation during study Incidence of mechanical ventilation (invasive or non-invasive) Categories: - Mechanical ventilation at baseline - First administration of mechanical ventilation post-baseline - No administration of mechanical ventilation Mechanical ventilation started post-baseline - Not started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | | of the end of ICU admission is missing then use 23:59. The derivation |
| oxygen administration Supplementation". In addition, the following categorization will be done: - Invasive Mechanical Ventilation - Non-Invasive Mechanical Ventilation - Non-Invasive, Non-mechanical Ventilation - None Mechanical ventilation during study Incidence of mechanical ventilation (invasive or non-invasive) Categories: - Mechanical ventilation at baseline - First administration of mechanical ventilation post-baseline - No administration of mechanical ventilation Mechanical ventilation started post-baseline - Not started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | Type of supplemental | Tabulation will be done as collected per CRF page "Oxygen |
| - Non-Invasive Mechanical Ventilation - Non-Invasive, Non-mechanical Ventilation - None Mechanical ventilation during study Incidence of mechanical ventilation (invasive or non-invasive) Categories: - Mechanical ventilation at baseline - First administration of mechanical ventilation post-baseline - No administration of mechanical ventilation Mechanical ventilation Incidence of post-baseline mechanical ventilation (invasive or non-invasive) - Started post-baseline - Not started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | | Supplementation". In addition, the following categorization will be |
| - Non-Invasive Mechanical Ventilation - Non-Invasive, Non-mechanical Ventilation - None Mechanical ventilation during study Incidence of mechanical ventilation (invasive or non-invasive) Categories: - Mechanical ventilation at baseline - First administration of mechanical ventilation post-baseline - No administration of mechanical ventilation Mechanical ventilation Incidence of post-baseline mechanical ventilation (invasive or non-invasive) - Started post-baseline - Not started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | | - Invasive Mechanical Ventilation |
| - Non-Invasive, Non-mechanical Ventilation - None Mechanical ventilation during study Incidence of mechanical ventilation (invasive or non-invasive) Categories: - Mechanical ventilation at baseline - First administration of mechanical ventilation post-baseline - No administration of mechanical ventilation Mechanical ventilation Incidence of post-baseline mechanical ventilation (invasive or non-invasive) - Started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | | |
| Mechanical ventilation during study Categories: - Mechanical ventilation at baseline - First administration of mechanical ventilation post-baseline - No administration of mechanical ventilation Mechanical ventilation Incidence of post-baseline mechanical ventilation (invasive or non-invasive) - Started post-baseline - Not started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | | |
| Mechanical ventilation during study Categories: - Mechanical ventilation at baseline - First administration of mechanical ventilation post-baseline - No administration of mechanical ventilation Mechanical ventilation Incidence of post-baseline mechanical ventilation (invasive or non-invasive) - Started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | | |
| during study Categories: - Mechanical ventilation at baseline - First administration of mechanical ventilation post-baseline - No administration of mechanical ventilation Mechanical ventilation started post-baseline Incidence of post-baseline mechanical ventilation (invasive or non-invasive) - Started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | Mechanical ventilation | |
| - Mechanical ventilation at baseline - First administration of mechanical ventilation post-baseline - No administration of mechanical ventilation Mechanical ventilation Incidence of post-baseline mechanical ventilation (invasive or non-invasive) - Started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | during study | ` |
| - No administration of mechanical ventilation Mechanical ventilation started post-baseline Incidence of post-baseline mechanical ventilation (invasive or non- invasive) - Started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | | |
| - No administration of mechanical ventilation Mechanical ventilation started post-baseline Incidence of post-baseline mechanical ventilation (invasive or non- invasive) - Started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | | - First administration of mechanical ventilation post-baseline |
| started post-baseline - Started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | | _ |
| started post-baseline - Started post-baseline - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | Mechanical ventilation | Incidence of post-baseline mechanical ventilation (invasive or pon- |
| <ul> <li>Started post-baseline</li> <li>Not started post-baseline</li> <li>Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject</li> </ul> | | |
| - Not started post-baseline Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | Post ouseille | , · |
| Note: In case mechanical ventilation is present at baseline and a second episode of mechanical ventilation is initiated post-baseline, this subject | | <u> </u> |
| episode of mechanical ventilation is initiated post-baseline, this subject | | <u> </u> |
| will be counted as started post-baseline. | | will be counted as started post-baseline. |

| Time from start of mechanical ventilation to end of mechanical ventilation (hours) [Time-to event] | The time from max(start date and time of first mechanical ventilation, study drug intake) until the end date and time of mechanical ventilation. Note: Invasive and non-invasive mechanical ventilation are considered and are defined on the Oxygen Supplementation form: Type of supplemental oxygen administration. Only the first mechanical ventilation period is considered. Censoring and calculation of the end time will be done analogous to "Time to hospital discharge" if time part of the start of mechanical ventilation is missing then it will be imputed with 00:00. Subjects that are not on mechanical ventilation (at any point during the trial) are excluded from this analysis and this analysis is restricted to |
|---|---|
| Total time on mechanical ventilation (hours) [Duration] | the first time mechanical ventilation is used. The total number of hours of mechanical ventilation during the period from first intake until study termination, calculated as sum of [(end date and time of mechanical ventilation— start date and time of mechanical ventilation)/3600], rounded to one decimal for all separate events per subject |
| | In case mechanical ventilation was started before first intake or in case the start datetime of mechanical ventilation is missing, then the date and time of first intake will be used. In case mechanical ventilation ended after the end of the trial or in case |
| | the end datetime of mechanical ventilation is missing, then the end datetime of last contact date will be used. If time of the start of mechanical ventilation is missing, then use 00:00. If time of the end of mechanical ventilation is missing, then use 23:59. The derivation of the total time is analogous to "Total length of hospital stay". |
| Time to clinical response (hours) [Time-to event] | The time to clinical response is defined as the time (in hours) from first study drug intake until the first assessment (actual date and time) of a successive series of 4 recordings (over 5 scheduled successive analysis timepoints, 1 missing timepoint is allowed) where at least 4 of 5 symptoms (temperature, blood oxygen saturation, heart rate, SBP, respiration rate) are normalized, with at least normalization of temperature and blood oxygen saturation. Normalization of clinical response is defined in Table 4. |

2020

Only vital signs assessments performed during hospitalization (excluding measurements during re-hospitalization) and up to Day 14 (during hospitalization) or Day 19 (for subjects with extended treatment during hospitalization) will be taken into account to determine time to clinical response. Assessments taken after hospital discharge or after Day 14 or Day 19 (for subjects with extended treatment), whichever comes first, will not be taken into account. In case there was more than one hospitalization period, only assessments of the first hospitalization period will be used.

In case clinical response is not met, data will be censored. Censoring will be done as follows

1) Last non-missing record in the applicable period indicate normalization (but insufficient recordings to meet the time to clinical response criteria)

Censoring will be done at the first record of normalization

2) Last non-missing record in applicable period does not indicate normalization

Censoring will be done after the last observation of vital signs recordings, which is 13:00 on the same day if the last observation was a morning assessment (from 3:01 until 11:00), 21:00 if the last observation was an afternoon assessment (from 11:01 until 19:00), 5:00 the next day if the last assessment was an evening assessment (from 19:01 until 03:00).

When not all parameters are available on a certain timepoint then following rules apply:

- If temperature or oxygen saturation are available but not normalized then there is no resolution for this timepoint
- If more than 2 parameters are not normalized then there is no resolution for this timepoint
- If 4 parameters including temperature and oxygen saturation are normalized (allowing 1 missing parameter) then there is resolution for this timepoint.

Else the resolution on this timepoint is missing

Subjects without postbaseline data are excluded.

Within 1 timepoint the assessments of the different parameters are taken together for evaluating the clinical response and the time of the last record within that time point is used. Unscheduled assessments are not taken into account. When multiple assessments for 1 parameter occur within one timepoint then only the last is used for that parameter.

**Table 4: Resolution Criteria for Vital Signs** 

| Assessment | Resolution Criterion |
|---|---|
| Temperature | Oral temperature $\leq$ 37.0 °C (without the use of antipyretics within 8 hours)*1 |
| Oxygen saturation | a) $\geq$ 94% on room air without supplemental oxygen* <sup>2</sup> |
| | b) In case pre-influenza infection oxygen saturation |
| | <94%*3: Return to pre-influenza oxygen saturation*4 |
| Respiration rate | ≤ 24/min or |
| | return to pre-influenza infection oxygen requirement in |
| | patients with chronic oxygen use*4,5 |
| Heart rate | ≤ 100/min |
| Systolic blood | $\geq$ 90 mmHg (without inotropic support given within 2 |
| pressure | hours of assessment) *6 |

<sup>\*</sup>¹Based on the Vital Signs form, question""Were there any antipyretic medications given within 8 hours before temperature measurement""

# Time to respiratory response (hours) [Time-to event]

Time respiratory response is defined as the time (in hours) from first study drug intake until the first assessment (actual date and time) of a successive series of 4 recordings (over 5 scheduled successive analysis timepoints, 1 missing timepoint is allowed) where the resolution criteria of both blood oxygen saturation and respiration rate as specified in Table 4 are met.

Censoring and calculation of the time will be done analogous to "Time to clinical response".

In case 1 of the parameters is missing and the available parameter is not normalized then there is no resolution on this timepoint.

In the other cases where 1 or 2 parameters are missing, the resolution will be also missing.

<sup>\*2</sup>Based on the oxygen saturation level measured on room air and "YES" on the question 'Is the patient able to sustain a blood oxygen saturation >= 94% when breathing room air for 15 min at any time on the day of assessment?' on the vital signs form.

<sup>\*&</sup>lt;sup>3</sup>If pre-influenza oxygen saturation level is below 94% and measured on room air \*<sup>4</sup>Return to pre-influenza infection oxygen requirement is based on the oxygen supplementation form: "Has supplemental oxygen administration returned to that level provided prior to the current respiratory infection?"

<sup>\*5</sup>Chronic oxygen use is based on the question "Does the subject require chronic oxygen"

<sup>\*6</sup> Inotropic support given within 2 hours of assessment as recorded in the vital signs form.

| Incidence of treatment-<br>emergent adjudicated<br>influenza complications | The incidence of treatment-emergent adjudicated influenza complications from first study drug intake until the end of the study will be categorized in a hierarchical fashion. The incidence will be presented for the overall category, for the subcategories and for each adjudicated complication within a subcategory. |
|---|---|
| | The overall category will consist of any adjudicated complication. |
| | The following subcategories are defined: |
| | Pulmonary complications: |
| | <ul> <li>respiratory failure,</li> <li>primary viral pneumonia,</li> <li>secondary bacterial pneumonia,</li> <li>exacerbations of chronic underlying pulmonary diseases,</li> <li>bronchitis</li> </ul> |
| | o other complications |
| | Extrapulmonary complications: |
| | <ul> <li>Cardiovascular and cerebrovascular disease (eg, myocardial infarction, congestive heart failure, arrhythmia, stroke),</li> <li>Muscular disorders (eg, myositis, rhabdomyolysis),</li> <li>Central nervous system (CNS) involvement,</li> <li>Acute exacerbation of chronic kidney disease,</li> <li>Decompensation of previously controlled diabetes mellitus,</li> <li>Other infections (eg, sinusitis, otitis)</li> </ul> |
| | <ul> <li>Other complications</li> </ul> |
| | <ul> <li>Pulmonary complications including sinusitis and otitis</li> <li>Major / minor complications</li> <li>Infectious / non-infectious complications</li> <li>The complications sinusitis and otitis are determined based on their MedDRA preferred terms as listed in Attachment 1, table 6, for the protocol terms 'Sinus infection' and 'ear infection' respectively. Only if those terms are judged to be complications by the adjudication committee they will be included for the endpoint 'Pulmonary complications including sinusitis and otitis.</li> </ul> |
| Incidence of not being | On Day 6 (relative day) subject is in the hospital at least a part of the |
| hospitalized on Day 6. | day ('Yes') or the subject is not in the hospital during the whole day ('No'). |
| Incidence of hospital readmission | Does the subject require hospital readmission after first discharge (The start date of the hospital readmission must be at least 1 day in between the end of the previous hospitalization)? Categories will be Yes (1) or No (0). |

| Incidence of all-cause | Did the subject die after first dose of study drug? |
|---|---|
| mortality | Categories will be Yes (1) or No (0). |
| Hospital recovery scale outcome assessed on Day 2 to 14 excluding Day 6 | The hospital recovery scale outcome defined per day for Day 2 to 14 excluding Day 6 is defined analogous to the primary endpoint. |
| Fundamental Hospital recovery scale outcome assessed on Day 2 to 14 | The fundamental hospital recovery scale reflects the status of the subject objectively independent of the opinion of the investigator (irrespective of being ready for discharge or requiring ICU level of care). The Fundamental hospital recovery scale outcome assessed on Day 2 to Day 14 is defined as follows: 6. Death |
| | <ul> <li>Subject died at any time on the day of assessment or earlier<br/>(all-cause mortality).</li> </ul> |
| | 5. On invasive mechanical ventilation |
| | <ul> <li>Invasive mechanical ventilation is used at any time on the day<br/>of assessment.</li> </ul> |
| | 4. In ICU |
| | 3. Non-ICU hospitalization, on supplemental oxygen |
| | <ul> <li>Non-ICU hospitalized on the day of assessment (including<br/>readmittance) and the subject is on supplemental oxygen. On<br/>supplemental oxygen is defined by:</li> </ul> |
| | <ul> <li>Receiving supplemental oxygen through a face mask or nasal cannula.</li> </ul> |
| | 2. Non-ICU hospitalization, without supplemental oxygen |
| | <ul> <li>Non-ICU hospitalized on the day of assessment (including readmittance)</li> </ul> |
| | 1. Not hospitalized |
| | <ul> <li>Discharged from the hospital before the day of assessment.</li> </ul> |
| Incidence of antibiotic treatment | Did the subject use antibiotic treatment after first dose of study drug? |
| treatment | Categories will be Yes (1) or No (0). The derivation of the categories will be based on the ATC level 2 categorization of concomitant medications. Concomitant medications coded as "J01" will be indicated as antibiotic treatment. |

| Duration of antibiotic treatment (hours) [Duration] | The total number of hours a subject used antibiotic treatment (= event) during the period from first intake until study termination, calculated as sum of [(end date and time of event – start date and time of event)/3600], rounded to one decimal for all separate events per subject. |
|---|---|
| | In case the start datetime is entirely or partially unknown and the medication was used before start of first intake the date and time of first intake will be used. |
| | In case the end datetime is entirely or partially unknown and the medication was used after the trial ended, the last contact date will be used to calculate the duration. |
| | If time of the start antibiotic treatment is missing, then use 00:00. If time of the end of antibiotic treatment is missing, then use 23:59The derivation of the duration is analogous to "Total length of hospital stay". |
| Time to NEWS2 <= 2 (hours) [Time- to event] | The time (hours) from first study drug to first time NEWS2<=2 maintained for 24 hours i.e. the time of the first of at least 2 consecutive NEWS2 assessments with 24 hours in between. |
| [Time to event] | If time is missing for the NEWS2, but timepoint is available then time will be imputed: if morning then time will be 08:00, if midday then time will be 12:00, if evening then time will be 20:00. |
| | Subjects that did not maintain a NEWS2<= 2 for 24 hours until completion of the trial or withdrawal, will be censored at the time of completion of withdrawal of the study. If time is not available then it will be imputed with 23:59. |
| | If the subject died before having a NEWS2 <=2 for 24 hours, the subject will be censored at the maximum time of all subjects. |
| Time to clinical improvement (hours) | The time (hours) from first study drug to clinical improvement. Clinical improvement is defined as the minimum of the time to hospital discharge or time to NEWS2 <=2 maintained for 24 hours. |
| [time- to event] | Censoring will be done similarly as 'time to hospital discharge' and 'time to NEWS2<=2'. |

| Time to clinical failure (days) | The time (in days) from first study drug intake to first clinical failure(=event). |
|---|---|
| [Time-to event] | Clinical failure is defined as having one of the following events |
| | • HRS >3 |
| | The first event will be considered. In case mechanical ventilation is started multiple times, only the first start of mechanical ventilation after first study drug intake is used. |
| | Subjects without a clinical failure at the time of completion or at the time of withdrawal from the study will be censored at the date of completion or withdrawal. |
| | (Date of event or censoring— date of first dose of study drug) + 1 |
| Incidence of Mortality per day | Number and percentage of subjects that died and cumulative number and percentage of subjects that died per day after first study drug. |

#### 5.3.1.2. Viral kinetics

The viral culture (TCID<sub>50</sub>) measurements are analyzed using two methods (depending on influenza subtype); i.e. NP ELISA and Hemagglutination Inhibition Assay. For analysis purposes the results from the NP ELISA method will be used when available, otherwise the results from the Hemagglutination Inhibition Assay will be used. This will be determined per analysis visit. As a consequence, the series of results of a subject can be a combination of both methods (for example at baseline the NP ELISA result is used and at Day 3 the Hemagglutination Inhibition Assay result is used).

Endpoints listed below will be based on results from nasal mid-turbinate (MT) swabs taken from central testing, excluding data from leftover samples from local virology tests.

| Measurement | Formula |
|---|---|
| Log <sub>10</sub> viral load actual values | Log <sub>10</sub> of the actual values as measured with qRT PCR |
| Viral load negativity (Log <sub>10</sub> vp/mL) | Viral load will be categorized as Negative or Positive: • Negative ("TARGET NOT DETECTED") • Positive ('TARGET DETECTED' or an actual value). |

| Viral load categorization (Log10 | Viral load will be categorized as Target not detected, Target detected, and Quantifiable: |
|---|---|
| vp/mL) | Target not detected |
| | Target detected |
| | Quantifiable |
| Log <sub>10</sub> viral load change from baseline | Log <sub>10</sub> viral load post-baseline value – log <sub>10</sub> viral load baseline value |
| Log <sub>10</sub> viral titer actual values | Log <sub>10</sub> of the actual values as measured with viral culture |
| Viral titer negativity | Viral titer will be categorized as Negative or Positive: |
| $(\text{Log}_{10} \text{ TCID}_{50}/\text{mL})$ | Negative (lower than LOQ) |
| | Positive (quantifiable results) |
| Log <sub>10</sub> viral titer change from baseline | Log <sub>10</sub> viral titer post-baseline value – log <sub>10</sub> viral titer baseline value |
| Viral load AUC <sub>0-10d</sub> | ■ Viral load AUC calculated from baseline to Day 10: |
| trapezoidal method | AUC is calculated by the trapezoidal summation rule, based on planned days of sampling, including the timepoints with (imputed) values available: |
| | Sum over $i$ of $(t_{i+1}-t_i)*(Viral\ load_{ti+1}+Viral\ load_{ti})/2$ |
| | The following rules will be applied in the order described below to deal with missing values before calculating the Viral load AUC: |
| | • If the baseline value is missing, then the mean baseline value over all subjects in the ITT-i set will be used. |
| | • If a single or sequential intermediate value (not the baseline value) is missing, then the missing value will be replaced by linear interpolation of the two adjacent values. Note: this is done automatically when applying the trapezoidal summation rule. If Day 10 value is missing, but there is an assessment after Day 10, then this value will be used to interpolate the value of Day 10. |
| | • If the Day 10 value is missing, and there are no values available after Day 10, then it will be imputed with the last observed post-baseline value (LOCF). |
| | Note: In case no post baseline value is available the AUC will be missing. |

| Viral titer AUC <sub>0-10d</sub> | Viral titer AUC calculated from baseline to Day 10: |
|---|---|
| trapezoidal method | AUC is calculated by the trapezoidal summation rule, based on planned days of, including the timepoints with (imputed) values available: |
| | Sum over i of $(t_{i+1}-t_i)*(Viral\ titer_{ti+1}+Viral\ titer_{ti})/2$ |
| | The following rules will be applied in the order described below to deal with missing values before calculating the Viral titer AUC: |
| | • If the baseline value is missing, then the mean baseline value over all subjects in the ITT-i set will be used. |
| | • If a single or sequential intermediate value (not the baseline value) is missing, then the missing value will be replaced by linear interpolation of the two adjacent values. Note: this is done automatically when applying the trapezoidal summation rule. If Day 10 value is missing, but there is an assessment after Day 10, then this value will be used to interpolate the value of Day 10. |
| | • If the Day 10 value is missing, and there are no values available after Day 10, then it will be imputed with the last observed post-baseline value (LOCF). |
| | Note: In case no post baseline value is available the AUC will be missing. |
| Time to viral negativity<br>by qRT-PCR (days)<br>[Time-to event] | The time to viral negativity is defined as the time (in days) from first study drug intake until a subject is considered influenza A viral negative. This is the first timepoint of two consecutive timepoints with a negative nasal MT swab, i.e. the first and next assessment equal to 'negative' (ignoring missing values). In case the first 'negative' is the last available assessment the subject is considered to have reached viral negativity at this last assessment. If this doesn't occur, a subject will be censored at the time of the last observed non-negative swab + 1 day. Note that for deriving the time to viral negativity by qRT-PCR every subject is considered positive at baseline. For subjects without postbaseline records, they are censored at Day 1. |
| Time to viral negativity<br>by viral culture (days)<br>[Time-to event] | The algorithm for Time to viral negativity by viral titer is similar as 'Time to viral negativity by viral load' but viral titer assessments are used instead. |

# **5.3.1.3.** Patient Reported Outcomes

| Measurement | Formula |
|---|---|
| Daily activities resumption | The daily activities resumption will be assessed once daily by means of the question 'Over the past 24 hours, how much has influenza interfered with your ability to carry out your daily activities?' The responses will be dichotomized: 'Not at all' and 'A little bit' will be considered as category "returned to daily activities" and responses 'Somewhat', 'Quite a Bit' and 'Very much' will be considered in category "not returned to daily activities". |
| Time to return to daily activities (days) [Time-to event] | The time to return to daily activities is defined as the time in days from initiation of study treatment (baseline assessment excluded) to the first of a successive series of 2 recordings in which the response is considered as returned to daily activities. The 2 successive recordings may have been done over 3 scheduled successive analysis timepoints, in case of 1 missing in between timepoint. |
| | In case the return to daily activities is not achieved, data will be censored. |
| | Censoring will be done as follows: |
| | Last non-missing record in indicate return to daily activities (but insufficient recordings) |
| | Censoring will be done at the first record of return to daily activities |
| | 2) Last non-missing record does not indicate return to daily activities |
| | Censoring will be done one day (24 hours) after the last observation. |
| | The time to return to daily activities is calculated as: Date and time of event (actual) or censoring - date and time of first dose of study drug)/(3600*24), rounded to one decimal. |
| | Subjects without postbaseline records are excluded from the analysis. |
| Patient Global<br>Impression of Severity<br>of Influenza symptoms | The PGIS captures daily influenza symptom severity from the subjects' perspective per timepoint. Responses will be categorized as :"No Flu symptoms today", and "Mild", "Moderate", "Severe" or "Very Severe". |

Patient global Impression of Change in Influenza symptoms The PGIC<sup>[4]</sup> is aimed to capture the subject's perceptions of improvement or deterioration in the severity of influenza symptoms compared to when the subject arrived to the hospital for influenza treatment and this is done per timepoint.<sup>[5]</sup>

Categories are: "Much better", "Somewhat better", "A little better" "About the same", "A little worse", "Somewhat worse" and "Much worse".

EQ-5D dimension parameters: Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression The EQ-5D (Attachment 5)<sup>[2]</sup> descriptive system consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with 5 possible levels (no problems (level code = 1), slight problems (level code = 2), moderate problems (level code = 3), severe problems (level code = 4), extreme problems (level code = 5)) (see Table 5). Each dimension will be captured in one parameter

**Table 5: EQ-5D Dimensions** 

| Di | mension | Le | vel | Interpretation |
|---|---|---|---|---|
| 1 | Mobility | 1 | No problems | I have no problems in walking about |
| | - | 2 | Slight problems | I have slight problems in walking about |
| | | 3 | Moderate | I have moderate problems in walking about |
| | | | problems | |
| | | 4 | Severe | I have severe problems in walking about |
| | | | problems | |
| | | 5 | Extreme | I am unable to walk about |
| | | | problems | |
| 2 | Self-care | 1 | No problems | I have no problems washing or dressing mysel |
| | | 2 | Slight problems | I have slight problems washing or dressin |
| | | | | myself |
| | | 3 | Moderate | I have moderate problems washing or dressin |
| | | | problems | myself |
| | | 4 | Severe | I have severe problems washing or dressin |
| | | | problems | myself |
| | | 5 | Extreme | I am unable to wash or dress myself |
| | | | problems | |
| 3 | Usual activities | 1 | No problems | I have no problems doing my usual activities |
| | | 2 | Slight problems | I have slight problems doing my usual activities |
| | | 3 | Moderate | I have moderate problems doing my usua |
| | | | problems | activities |
| | | 4 | Severe | I have severe problems doing my usual activitie |
| | | | problems | |
| | | 5 | Extreme | I am unable to do my usual activities |
| | | | problems | |
| | | L . | | |
| 4 | Pain/discomfort | 1 | No problems | I have no pain or discomfort |
| | | 2 | Slight problems | I have slight pain or discomfort |
| | | 3 | Moderate | I have moderate pain or discomfort |
| | | _ | problems | 111 |
| | | 4 | Severe | I have severe pain or discomfort |
| | | Ļ | problems | 71 |
| | | 5 | Extreme | I have extreme pain or discomfort |
| | | | problems | |
| - | A /1 . | - | NT 11 | Y |
| 5 | Anxiety/depression | 1 | No problems | I am not anxious or depressed |
| | | 2 | Slight problems | I am slightly anxious or depressed |

| | 3 Moderate I am moderately anxious or depressed problems |
|---|---|
| | 4 Severe I am severely anxious or depressed problems |
| | 5 Extreme I am extremely anxious or depressed problems |
| EQ-5D visual analogue scale (VAS) | EQ-5D VAS is a continuous score ranging from 0 (worst health you can imagine) to 100 (best health you can imagine). |
| EQ-5D VAS change from baseline | EQ-5D VAS post-baseline value – EQ-5D VAS baseline value |
| EQ-5D VAS clinically relevant change from baseline | The change from baseline in EQ-5D VAS will be categorized in two ways: 1. $\leq$ -7, -6 to 6, $\geq$ 7 2. $\leq$ -10, -9 to 9, $\geq$ 10 |
| EQ-5D Valuation index | |
| EQ-5D Valuation index change from baseline | EQ-5D valuation index post-baseline value – EQ-5D valuation index baseline value |

# 5.3.2. Analysis Methods

# **Descriptive statistics**

The descriptive statistics that will be shown may include the number of subjects, mean, standard deviation, standard error, 95% CI, median, range, interquartile range and geometric mean with corresponding 95% CI.

# Kaplan-Meier analysis, Gehan-Wilcoxon test and Log-rank test

All Time-to event variables will be analyzed using a stratified Gehan-Wilcoxon test, a stratified log-rank test and Kaplan-Meier estimates. For endpoints where the start time is not the start of the treatment A summary table including number of subjects included in the analysis, number of subjects censored, 25th and 75th percentiles and median time-to event, with 95% confidence intervals based on log-log transformation method, and the p-values calculated based on the stratified Gehan-Wilcoxon test and stratified log-rank test will be presented.

The data will be presented graphically using the Kaplan-Meier estimate of the survival function by treatment.

For all subgroup analyses, Kaplan-Meier plots will be produced per subgroup and Gehan-Wilcoxon test will be produced for each category of a subgroup.

# Accelerated failure time (AFT) model

When indicated, time-to event variables will be compared between pimodivir and placebo using an accelerated failure time (AFT) model. The distribution to be used will be determined based on the goodness of fit of the model using Akaike's information criterion and will be selected from the following parametric families: lognormal, log-logistic, or Weibull. The AFT model will include the fixed, categorical effects for treatment (with placebo as the reference), the time from admission to start of treatment (for the time to hospital discharge and time to hospital discharge readiness) and stratification factors (type of baseline SOC, time of onset of symptoms and screening NEWS2). The scale parameter will be the same across groups

A summary of the final AFT model will include parameter estimates and associated standard errors, estimated accelerated failure time ratios versus placebo and associated 95% confidence intervals, and p-values. The survival curves per treatment group of the accelerated failure time model will also be shown with the Kaplan-Meier plots included in the same output.

For subgroup analyses the survival curves will be shown for each subgroup category separately.

Bootstrapping with replacement, considering also the actual proportion of subjects in each stratum, will be used to obtain a 100% sample size 10001 times. The median (95% CI) time-to event will be derived from the 10001 bootstrapped samples.

#### Cox Proportional Hazard model

A stratified Cox proportional hazards model will be used adjusted for the stratification factors and for the time from admission to start of treatment (for the time to hospital discharge and time to hospital discharge readiness),. The hazard ratio for the comparison of pimodivir versus placebo will be reported together with the 95% confidence interval. A Log-log plot of survival will be added to check the proportional hazard assumption of the Cox proportional hazards model.

For the subgroup analyses the Log-Log plot of survival will be shown for each subgroup category separately.

#### **Logistic regression model**

A logistic regression model (Firth's penalized likelihood approach), with treatment group and stratification factors as fixed effects, will be used to analyze binary outcomes and to obtain the odds ratios (95% CI) for the comparison of pimodivir versus placebo.

#### 5.3.2.1. Clinical outcome

#### Time-to event parameters for clinical outcome

The time-to event parameters for clinical outcome will be analyzed as described above using a stratified Gehan-Wilcoxon test, a stratified log-rank test, a Kaplan-Meier analysis, an accelerated failure time model and a Cox proportional hazards model The Gehan-Wilcoxon test is the primary analysis for time-to-event parameters. The Kaplan-Meier analysis will provide the primary estimation of time-to-event.

#### **Duration parameters**

Descriptive statistics of the duration parameters will be shown for all subjects that had the specific event. e.g. only subjects admitted to ICU will be included in the total time in ICU analysis

Total length of hospitalization, total time in ICU, total duration of antibiotics, and total time on mechanical ventilation will be analyzed by using the Hodges-Lehman approach. Corresponding 95% CIs will be presented as well.

#### **Incidence parameters**

For each parameter the number and percentage of subjects in each category and subcategory will be tabulated and listed. All Subjects in the applicable analysis set will be counted for the denominator of the proportion.

The occurrence (yes/no) as described for the incidence parameters will be analyzed using logistic regression as described above (Section 5.3.2).

The occurrence (yes/no) of influenza complications will be analyzed using logistic regression as described above for the following categories:

- the overall influenza complications
- the pulmonary complications,
- the extrapulmonary complications
- the infectious complications
- the non-infectious complications
- the major complications
- the minor complications
- the pulmonary complications including sinusitis and otitis

# Hospital recovery scale outcome and fundamental hospital recovery scale outcome on Day 2 to 14

This parameter will be analyzed analogous to the primary endpoint: hospital recovery scale outcome on Day 6, but then for Day 2 to 14 with Day 6 excluded for the HRS and including Day 6 for the fundamental HRS. The proportional odds model will be applied, and the proportional odds assumption will be tested for the treatment effect. The same 5 dichotomization of the HRS will be analyzed using a logistic regression model. Also, similarly as the primary endpoint the Van Elteren test will be provided in case the proportional odds assumption is not valid. The MI analysis will not be applied.

A tabulation will be made of the (fundamental) hospital recovery scale outcomes at each day (including Day 6), taking only non-missing values into account (i.e.: the percentages of the six categories per day should sum up to 100%). A second tabulation will be made of the hospital recovery scale outcomes at each day including a category for missing values. The first day with 30% of subjects not hospitalized will be identified. All Subjects in the applicable analysis set will be counted for the denominator of the calculation.

# 5.3.2.2. Viral Kinetics

# Viral load and viral titer over time

The actual values and change from baseline of the viral load and viral titer over time will be shown descriptively and by mean (SE) plots per analysis timepoint.

Individual AUCs from baseline to Day 10 for both viral load and viral titer will be calculated using the trapezoid method and summarized using descriptive statistics.

Viral load negativity, viral load categorization and viral titer negativity will be summarized using frequency tabulations (n and %) at each analysis visit. All subjects with lab data on the specific visits/timepoints will be used as denominator.

■ Difference in mean viral load AUC calculated from baseline to Day 10:

Post-baseline mean viral load values up to and including Day 10 over time will be analyzed using a restricted maximum likelihood based repeated measures approach. Analyses will include the fixed, categorical effects of treatment, strata, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline viral load and baseline viral load -by-visit interaction. The following list of covariance structures will be applied in the model fit, in the specified order, and the first correlation structure to yield convergence will be applied in the analysis:

- Unstructured [UN]
- Ante-dependence [ANTE(1)]
- Heterogenous Toeplitz [TOEPH]
- Heterogeneous CS [CSH]
- Heterogeneous AR(1) [ARH(1)]
- Toeplitz [TOEP]

The Kenward-Roger approximation will be used to estimate denominator degrees of freedom.

The model above will be used to estimate the difference in the viral AUCs for active versus placebo.

Post-baseline mean viral titer values up to and including Day 10 will be analyzed similarly.

A least squares means  $\pm 95\%$  CI plot will also be provided for the estimated viral load and estimated viral titer over time.

# Time to viral negativity by viral load and by viral titer

Analysis will be done analogous to the time-to event parameters for clinical outcome. The baseline viral load or viral titer will be added as covariate to the AFT and Cox Proportional Hazard model.

# 5.3.2.3. Patient Reported Outcomes

# Time to return to daily activities

Time to return to daily activities will be analyzed analogous to the time-to event parameters for clinical outcomes.

#### Patient Global Impression parameters and daily activities resumption

The subject's perception of severity and changes of influenza symptoms (PGIS, PGIC) and daily activities resumption will be tabulated per parameter and per category by analysis timepoint using frequency tabulations.

#### **EQ-5D** dimension parameters

Tabulations of the number (and percentage) of subjects per parameter, response and time point will be shown per treatment group.

#### **EQ-5D VAS, EQ-5D Valuation index**

The actual values and changes from baseline will be shown descriptively and by mean (SE) plots per analysis visit.

The proportion of subjects with a clinically relevant change from baseline of 7 or more (decrease or increase) and of 10 or more (decrease or increase) will be tabulated.

#### Missing data

- 1) If for a questionnaire one (or more) dimensions of the descriptive system are missing then
  - The EQ-5D VAS will be included in the analysis
  - The valuation index will not be included in the analysis
  - The non-missing dimensions of EQ-5D descriptive system will be

included in the analysis of the separate dimensions

2) If – for a questionnaire – the EQ-5D VAS is missing then the EQ-5D descriptive system and valuation index will be included in the analysis if complete (otherwise see 1)

#### 6. TASTE AND SWALLOWABILITY

#### 6.1. Definition

Taste and swallowability will only be assessed for adolescents in this study.

The acceptability of the taste will be derived from the responses to the overall question on taste, dichotomizing the responses 'None' and 'Weak' as acceptable and responses 'Moderate' or 'Strong' as unacceptable.

For swallowability, a dichotomization of the responses will be made of 'slightly difficult' or worse vs 'neither difficult nor easy' or better.

# 6.2. Analysis Methods

Taste and swallowability questionnaire results (collected for adolescents only who take pimodivir or placebo tablets; not applicable when tablets are administered via nasogastric tube) will be summarized per tablet intake (first and last intake of the study drug) by means of frequency tabulations of the actual responses. Additionally the number of subjects (%) will be presented by response category (including dichotomization) for swallowability and taste separately. Analyses will be done on the safety set.

#### 7. SAFETY

All safety analyses will be done on the Safety Set.

#### 7.1. Adverse Events

#### 7.1.1. Definitions

# **Coding of AE**

The verbatim terms used in the eCRF by investigators to identify AEs will be coded using the Medical Dictionary for Regulatory Activities. Events are looked at on the level of their preferred term.

# **Treatment-emergent AE**

Pre-treatment AEs are defined as AEs that were reported or worsened after signing the ICF up to the start of study drug dosing. Treatment-emergent AEs (TEAE) are defined as AEs that were reported or worsened on or after the start of study drug dosing and up to and including the end of the follow-up phase.

An AE, at the preferred term level, is considered treatment-emergent if:

- an AE starts after or at first dose of study drug and
  - o The AE was not present prior to first dose of study drug
- an AE was present prior to first dose of study drug:
  - the same AE (based on preferred term) starts at the end date or the day after the end date of the AE present prior to first dose and new AE has worsened, ie an increase in toxicity grade or changed to an SAE
  - the same AE (based on preferred term) started 2 or more days after the end date of the AE present prior to first dose
- The start date of the AE is missing
- The start time of the AE is missing, and the AE was not present the day before first dose of study drug, and the start date of the AE is the same as the start date of first dose of study drug
- The day is missing of the AE start date but month and year are the same as month and year of first study drug intake.
- The month is missing of the AE start date but the year is the same as the year of the first study drug intake.

#### Phase allocation of AE

Adverse events present in the SDTM database are allocated to phases based on their start date and time. If the start date and time of an event falls between (or on) the start and stop date and time of a phase, the AE is attributed to that phase (treatment-emergent principle).

Rule: phase start datetime  $\leq$  AE start datetime  $\leq$  phase stop datetime.

Incomplete AE dates and or times (i.e. time and/or day and/or month and/or year missing):

• In case of partial AE start dates and or times, the events are allocated to the phases using the available partial information on start and end datetime; no imputation will be done. If, for instance, for the AE start date only month and year are available, these data are compared to

the month and year information of the phases. This rule may lead to multiplication of the event as a consequence of its assignment to multiple phases or subperiods.

- In case of a completely missing AE start date, the event is allocated to the first active treatment phase and subperiod, except if the end date of the AE falls before the start of this active treatment phase and subperiod.
- In case of a completely missing AE end date, the following rules apply:
  - in case the date is identified as unknown the date will remain missing;
  - in case the date is not flagged as unknown the date is assumed to be the cut-off date of the analysis for subjects still ongoing in the study, and the end date of the last phase for subjects who discontinued or completed the study.

# Examples:

Screening phase: start date: 02JAN2017 - stop date: 28JAN2017 Treatment phase: start date: 29JAN2017 - stop date: 12AUG2017

- 1) Adverse event: start date: JAN2017- stop date: 15JUL2017
  As the AE start date only has information about month and year, only this information will be used from the phases and therefore the AE will be assigned to the screening phase as well as to the treatment phase.
- 2) Adverse event: start date: JAN2017- stop date 27JAN2017 As the AE stops before or at the start of the treatment phase, it is only assigned to the Screening phase.

*Remarks:* In addition to the date information, time information is taken into account to allocate AEs to phases.

#### **Adverse events**

The variables attributed to adverse events are

- AE term (verbatim and MedDRA preferred term and system organ class)
- Onset datetime, End datetime and duration of AE
- Serious AE (Yes/No), if yes classification will be listed
- Toxicity grade (Mild, Moderate, Severe, Potentially life-threatening)
- Action taken with study treatment (Dose not changed, Dose interrupted, Drug withdrawn, Not applicable, Unknown)
- Relation to study treatment (Not related, Doubtful, Possible, Probable, Very likely)
- Outcome of AE
- AE leading to death (Yes/No)
- Concomitant treatment taken for AE (Yes/No)
- Influenza-related complication (Yes/No)
- Required hospitalization/prolonged hospitalization (Yes/No)

# **Anticipated Events**

An anticipated event is an AE (serious or non-serious) that commonly occurs as a consequence of the underlying disease or condition under investigation (disease related) or background regimen.

For the purposes of this study the following events will be considered anticipated events (see Attachment 1: for the classification of AEs into Anticipated Events and Anticipated Event Groups):

- Pneumonia
- Bronchitis
- Sinus infections
- Ear infections
- Worsening of asthma, asthma attack
- COPD exacerbation
- Complications of sickle cell disease, sickle cell crisis
- Complications of diabetes mellitus, diabetic ketoacidosis
- Acute respiratory distress syndrome (ARDS)

# **Influenza-related complications**

The categories of influenza-related complications are defined in 5.3.1.1

#### **Confirmed diarrhea events**

Additional details required to confirm a diarrhea event, including number of loose stools episodes per day and stool consistency, will be collected for subjects who report a diarrhea type event.

A confirmed diarrhea event is defined as three or more loose stools episodes per day with a consistency of 'loose' or 'watery'.

# 7.1.2. Analysis Methods

#### **Treatment-emergent adverse events**

There will be no formal statistical testing unless indicated otherwise.

A summary will be provided for the following TEAEs per phase (Treatment phase, Follow-up phase), subperiod and for the combination of Treatment and Follow-up phase:

- any adverse events,
- serious adverse events,
- deaths due to AE.
- adverse events by worst toxicity grade,
- AEs of worst grade 3 or 4
- AEs of worst grade 3
- AEs of worst grade 4
- AEs at least possibly related to study drug,
- AEs for which study drug was temporarily stopped,
- AEs for which study drug was permanently stopped,
- AEs leading to study discontinuation
- serious adverse events that were at least possibly related to study drug,
- Adjudicated influenza related complications
- COVID-19 AEs
- COVID-19 Serious AEs
- COVID-19 Non-serious AEs

The adverse events will be shown by MedDRA system organ class and preferred term, in order of descending overall frequency in the pimodivir group. For each AE, the percentage of subjects who experience at least 1 occurrence of the given event will be summarized by treatment group and per phase (Treatment phase, Follow-up phase), subperiod and for the combination of Treatment and Follow-up phase. The tabulations will be provided for the following categories:

- any adverse events
- serious adverse events
- AEs at least possibly related to study drug
- AEs for which study drug was temporarily stopped
- AEs for which study drug was permanently stopped
- AEs leading to study discontinuation
- serious adverse events that were at least possibly related to study drug
- AEs related to COVID-19 infection
- Serious AEs related COVID-19 infection
- AEs related to COVID-19 infection leading to death

and in addition for treatment emergent adverse events with incidence of at least 5% in any treatment group.

In order to fulfil requirements for the plain language summary document and presentations for EudraCT the following adverse event categories will be shown by MedDRA system organ class and preferred term per phase (Treatment phase, Follow-up phase) and subperiods (treatment subperiod and treatment extension subperiod) and for the combination of Treatment and Follow-up phases. No tabulations by subgroups will be provided for these categories:

- deaths due to AEs that were at least possibly related to study drug
- AEs for which study drug was permanently stopped that were at least possibly related to study drug
- non-serious AEs that were at least possibly related to study drug
- any non-serious AEs

AEs leading to death, SAEs, AEs leading to dose interruption or permanent stop of study drug, AEs related to COVID-19 infection will be listed separately. All AEs will be listed in an individual subject data listing, including pre-treatment AEs. All listings will be provided for the safety set.

The duration (in days) of an AE is calculated based on the AE start date and AE end date as:

AE duration = AE end date - AE start date +1

Note that the AE duration will be calculated in case the start date and end date is fully known, in case of partial or missing start and end dates the AE duration will be put on missing.

# **Anticipated Events**

Frequency tabulations of anticipated events and anticipated event grouped terms will be shown for treatment phase and subperiods, follow-up phase and for the combination of treatment + follow-up phases. The tabulation will show per treatment the number (%) of subjects with serious, non-serious and total anticipated events and anticipated event grouped terms and a one-sided p-value of Fisher exact test for anticipated events and anticipated event grouped terms.

A listing of the anticipated events will be added.

More details on the anticipated events analysis can be found in the Anticipated Events Safety Monitoring plan.

# Influenza-related complications

Adverse Events adjudicated as influenza-related complications will be will be tabulated for treatment phase and subperiods, follow-up phase and for the combination of treatment + follow-up phases.

Adverse events that were assessed by the investigator as influenza-related complications will also be tabulated by category, subcategory (see Section 5.3.1.1) and adverse event, for treatment phase and subperiods, follow-up phase and for the combination of treatment and follow-up phases. A listing showing the AEs reported as influenza-related complications and complication information will be made linking the information to the AE listing. Additional analyses on adjudicated influenza-related complications are described in Section 5.3.2.1.

#### Confirmed diarrhea events

The number and percentage of subjects who experience at least 1 occurrence of confirmed diarrhea events will be summarized by treatment group and per phase (Treatment phase, Follow-up phase) and subperiods (treatment subperiod and treatment extension subperiod) and for the combination of Treatment and Follow-up phases.

For all subjects that complete the additional diarrhea form, a cross-tabulation of number of loose stools episodes per day (categorized as 1, 2, 3 or more) versus stool consistency will be produced by treatment group and per phase (Treatment phase, Follow-up phase) and for the combination of Treatment and Follow-up phases. If a subject has more than 1 diarrhea event per phase, then the worst response from all events in that phase will be tabulated.

Descriptive statistics will be produced by treatment group for the number of days from first dose of study drug to onset of first diarrhea event and for total duration of diarrhea events. A frequency tabulation will be produced by treatment group for the number of days from last dose of study drug to resolution of last diarrhea event.

Frequency tabulations will be produced by treatment group and per phase (Treatment phase, Follow-up phase and subperiods) and for the combination of Treatment and Follow-up phases for the severity grade of the diarrhea event and for whether any concomitant medication was used to treat the diarrhea event.

No tabulations by subgroups will be provided.

All information recorded on the specific diarrhea form will be listed.

# 7.2. Clinical Laboratory Tests

#### 7.2.1. Definitions

Laboratory parameters of hematology, serum chemistry and urinalysis will be investigated: all analyses will be done on SI-converted values as available in the database.

#### Imputations of numerical values expressed as characters

In case a laboratory test result is censored (no numeric value is available, but only a verbatim term), the following rules are applied:

- '<x' or '>x': a numeric value will be imputed by the cut-off value decreased or increased with one unit respectively
- ' $\leq$ x' or ' $\geq$ x': imputation by x.

# **Toxicity grades and abnormalities for laboratory parameters:**

The laboratory abnormalities will be determined according to the criteria specified in the WHO grading table<sup>[12]</sup> (see Attachment 2). Available toxicity grades in the laboratory raw data will not be used. In case no toxicity grades are defined for a test, the abnormalities (above/below normal range) will be used.

In determining toxicity grades/abnormalities for each subject the following rules are applied:

- Worst grades/abnormalities are determined over the whole observational period, per phase (treatment, follow-up and combination treatment + follow-up) and per subperiod (treatment, treatment extension) separately, including all post-baseline scheduled and unscheduled measurements of that phase.
- The abnormalities "abnormally low" and "abnormally high" are considered equally important, i.e. if a subject has as well an abnormally low as an abnormally high value post-baseline, both abnormalities are shown in the tables. (This implies that the sum of the percentages can be more than 100%)
- If, for a specific test, the grading list provides distinct limits for abnormally low (=hypo) values as well as for abnormally high (=hyper) values, this test should be repeated for hyper and hypo limits separately in cross-tabulations.

# Treatment-emergent definition for toxicity grades and abnormalities

An abnormality (toxicity grade or abnormality based on normal ranges) will be considered treatment-emergent if it is worse than the baseline abnormality. If the baseline abnormality is missing, the abnormality is always considered as treatment-emergent. A shift from "abnormally low" at baseline to "abnormally high" post-baseline (or vice versa) is also treatment-emergent.

# 7.2.2. Analysis Methods

Actual values and changes from baseline will be summarized by treatment group at each scheduled timepoint.

A tabulation of the toxicities/abnormalities per timepoint will be presented. This table will also show the number and percentage of subjects per toxicity/abnormality, the number and percentage of subjects per treatment-emergent abnormality, and the cumulative number of subjects per treatment-emergent abnormality per post-baseline timepoint. Include in this table the safety follow-up visit, the Day 28 final study visit and the last study visit.

Additionally, a tabulation of the worst toxicity/abnormality will be presented. This table will show the number and percentage of subjects per worst toxicity/abnormality. A cross-tabulation of the worst toxicity/abnormality versus baseline will be presented per phase (treatment, follow-up and combination treatment + follow-up) and per subperiod (treatment, treatment extension). This table will also show the number and percentage of subjects per worst toxicity/abnormality, the number and percentage of subjects per treatment-emergent worst toxicity/abnormality, and the cumulative number of subjects per treatment-emergent toxicity/abnormality.

For tabulations of hyperglycemia, the results will also be presented for the subgroup of subjects that had been fasting for at least 10 hours.

Mean  $\pm$  SE graphs over time for the actual values and changes from baseline will be generated for all tests performed.

A listing of abnormal individual subject hematology and clinical chemistry values from scheduled and unscheduled timepoints will be provided. This listing will include all other timepoints for the corresponding subject/parameter.

Grade 3 or higher toxicity laboratory values will be listed separately

Frequency tables (n %) will be produced for the categorical urinalysis parameters by treatment group at each scheduled timepoint. Include in this table the safety follow-up visit, the Day 28 final study visit and the last study visit.

All urinalysis results will be listed.

# 7.3. Vital signs

#### 7.3.1. Definitions

Vital signs (including temperature, pulse rate, respiratory rate, and blood pressure), peripheral capillary oxygen saturation, and level of consciousness (AVPU) will be included in the analysis.

Vital Signs abnormalities will be determined according to the WHO grading scale boundaries defined in Attachment 3, Table 4: Resolution Criteria for Vital Signs.

Worst abnormalities are determined over the whole observational period and per phase (treatment, follow-up and combination treatment + follow-up) and per subperiod (treatment, treatment extension), including all post-baseline scheduled and unscheduled measurements.

An abnormality (based on normal ranges) will be considered treatment-emergent if it is worse than the baseline abnormality. If the baseline abnormality is missing, the abnormality is always considered as treatment-emergent. A shift from "abnormally low" at baseline to "abnormally high" post-baseline (or vice versa) is also treatment-emergent.

Assessments (except oxygen saturation) taken while the subject was not in a supine position will not be included in descriptive statistics but will be considered in determining worst case values.

# 7.3.2. Analysis Methods

Actual values and changes from baseline will be summarized by treatment group at each scheduled timepoint.

A tabulation of the abnormalities per timepoint will be presented. This table will also show the number and percentage of subjects per abnormality, the number and percentage of subjects per treatment-emergent abnormality, and the cumulative number of subjects per treatment-emergent abnormality per post-baseline timepoint. Include in this table the safety follow-up visit, the Day 28 final study visit and the last study visit.

Additionally, a tabulation of the worst abnormality will be presented. This table will show the number and percentage of subjects per worst abnormality.

A cross-tabulation of the worst abnormality versus baseline will be presented per phase (treatment, follow-up and combination treatment + follow-up) and per subperiod (treatment, treatment extension). This table will also show the number and percentage of subjects per worst abnormality, the number and percentage of subjects per treatment-emergent worst abnormality, and the cumulative number of subjects per treatment-emergent abnormality.

Mean  $\pm$  SE graphs over time for the actual values and changes from baseline will be generated for all tests performed.

Vital signs data for subjects having at least one treatment-emergent abnormality will be listed.

# 7.4. Physical examinations

Abnormal physical examination results will be listed.

# 7.5. Electrocardiogram

PR interval, QT interval, QRS interval, Heart Rate and QTc intervals using Bazett's correction formula and Fridericia's correction formula will be investigated<sup>[1]</sup>. QTc values will be used as reported, they will not be recalculated. If the ECG is performed in triplicates the mean of the non-missing ECG recordings will be used as the value for each specific parameter and timepoint.

#### 7.5.1. Definitions

ECG abnormalities will be determined according to the boundaries defined in Attachment 4.

An abnormality (based on normal ranges) will be considered treatment-emergent if it is worse than the baseline abnormality. If the baseline abnormality is missing, the abnormality is always considered as treatment-emergent. A shift from "abnormally low" at baseline to "abnormally high" post-baseline (or vice versa) is also treatment-emergent. The treatment-emergent definition is applicable in both, the treatment and follow-up phase.

Assessments taken while the subject was not in a supine position will not be included in descriptive statistics but will be considered in determining worst case values.

# 7.5.2. Analysis Methods

Actual values and changes from baseline will be summarized by treatment group at each scheduled timepoint.

A tabulation of the abnormalities per timepoint will be presented. This table will also show the number and percentage of subjects per abnormality, the number and percentage of subjects per treatment-emergent abnormality, and the cumulative number of subjects per treatment-emergent abnormality per post-baseline timepoint. Include in this table the safety follow-up visit, the Day 28 final study visit and the last study visit.

A cross-tabulation of the worst abnormalities versus baseline will be presented per phase (treatment and follow-up, treatment and follow-up phase and subperiods). This table will also show the number and percentage of subjects per worst abnormality, the number and percentage of subjects per treatment-emergent abnormality, and the cumulative number of subjects per treatment-emergent abnormality.

Mean  $\pm$  SE graphs over time for the actual values and changes from baseline will be generated for all tests performed.

A frequency tabulation of the QT/QTc change categories at Day 28 versus baseline will be presented.

ECG data for subjects having at least one treatment-emergent abnormality will be listed.

# 7.6. National Early Warning Score

#### 7.6.1. Definitions

#### **NEWS**

The NEW Score<sup>[7]</sup> is an aggregated score with a range from 0 to 20 calculated as the sum of the scores per parameter (see Table 6, all parameters are based on the VS dataset and CM). However, in case information for a parameter is missing the NEW score cannot be calculated.

Table 6: National Early Warning Score (NEWS)\*

| Physiological<br>Parameters | 3 | 2 | 1 | 0 | 1 | 2 | 3 |
|---|---|---|---|---|---|---|---|
| Respiration<br>Rate | ≤8 | | 9 - 11 | 12 - 20 | | 21 - 24 | ≥25 |
| Oxygen<br>Saturations | ≤91 | 92 - 93 | 94 - 95 | ≥96 | | | |
| Any<br>Supplemental<br>Oxygen | | Yes | | No | | | |
| Temperature | ≤35.0 | | 35.1 - 36.0 | 36.1 - 38.0 | 38.1 - 39.0 | ≥39.1 | |
| Systolic BP | ≤90 | 91 - 100 | 101 - 110 | 111 - 219 | | | ≥220 |
| Heart Rate | ≤40 | | 41 - 50 | 51 - 90 | 91 - 110 | 111 - 130 | ≥131 |
| Level Of<br>Consciousness | | | | A | | | V,P, or U |

<sup>\*</sup>The NEWS initiative flowed from the Royal College of Physicians' NEWS Development and Implementation Group (NEWSDIG) report, and was jointly developed and funded in collaboration with the Royal College of Physicians, Royal College of Nursing, National Outreach Forum and NHS Training for Innovation

Note: The following parameters for the NEWS for subjects that are on invasive mechanically ventilation while NEWS is assessed will be adjusted:

Oxygen saturation = 90%

Any Supplemental oxygen = YES

Level of Consciousness = Unresponsive

The observed data values for these parameters will be ignored and replaced by above values. Subsequently all parameters will be evaluated according to Table 6.

#### **NEWS2**

The original NEWS was designed for patients whose normal range for oxygen saturation is between 96 - 100%. For SpO2 values below this, the NEW score increases. The NEWS is updated by a new version, NEWS2<sup>[8]</sup>, to more accurately score the acute-illness severity of subjects with routinely low oxygen saturation. Subjects that have a prescribed oxygen saturation requirement of
88 - 92%, i.e. patients with hypercapnic respiratory failure, often referred to as 'type 2' respiratory failure (Although COPD is the most common cause of hypercapnic respiratory failure, there are other causes such as morbid obesity, chest-wall deformities or neuromuscular disorders) will be evaluated with the new SpO2 scoring scale 2.

In addition, a new consciousness level is added to capture a change in confusion: new Confusion (C). Note: The following parameters for the NEWS2 for subjects that are on invasive mechanical ventilation and that met the criteria for the SpO2 scale 2 will be adjusted:

Oxygen saturation = 82% Any Supplemental oxygen = YES Level of Consciousness = Unresponsive

The observed data values for these parameters will be ignored and replaced by above values. Subsequently all parameters will be evaluated according to Table 7

Table 7: The NEWS2 scoring system

| Physiological | | | | Score | J. 5 | | 50 |
|---|---|---|---|---|---|---|---|
| parameter | 3 | 2 | 1 | 0 | 1 | 2 | 3 |
| Respiration rate (per minute) | ≤8 | | 9–11 | 12–20 | | 21–24 | ≥25 |
| SpO <sub>2</sub> Scale 1 (%) | ≤91 | 92–93 | 94–95 | ≥96 | | | |
| SpO <sub>2</sub> Scale 2 (%) | ≤83 | 84–85 | 86–87 | 88–92<br>≥93 on air | 93–94 on<br>oxygen | 95–96 on<br>oxygen | ≥97 on<br>oxygen |
| Air or oxygen? | | Oxygen | | Air | | | |
| Systolic blood<br>pressure (mmHg) | ≤90 | 91–100 | 101–110 | 111–219 | | | ≥220 |
| Pulse (per minute) | ≤40 | | 41–50 | 51–90 | 91–110 | 111–130 | ≥131 |
| Consciousness | | | | Alert | | | CVPU |
| Temperature (°C) | ≤35.0 | | 35.1–36.0 | 36.1–38.0 | 38.1–39.0 | ≥39.1 | |

Note: the physiological parameter: 'Air or Oxygen' is evaluated by checking the use of the supplemental oxygen. For the SpO2 scale 2, to evaluate if the assessment is taken on room air or on oxygen, the answer to the question 'Was this measurement taken on room air' is used. Oxygen saturation measurements lower or equal to 92% are scored 0 to 3 in the SpO2 scale 2 independent if the measurement was taken on room air or not. Oxygen saturation measurements of 92% or more on room air will have a score 0 for the SpO2 scale 2. Oxygen saturation measurements of 93 or more taken on oxygen are scored 1 to 3 in the SpO2 scale 2 (last 3 columns)

The subjects for who the oxygen saturations levels need to be evaluated with the  $SpO_2$  scale 2, met following criteria at (or before) the time of randomization:

- Oxygen saturation of the last assessment before randomizing is lower or equal to 92%
- Chronic oxygen was used

The SpO<sub>2</sub> scale 2 will then be used for the NEWS2 calculation throughout the rest of the trial for the subject. The SpO<sub>2</sub> scale 1 will be used for the other subjects.

Note that for the NEWS2 by timepoint a subject receives supplemental oxygen if he received oxygen at the time of the measurement of oxygen saturation. For the NEWS(2) stratification this is checked within the randomization window as explained in Section 5.1.4

# **NEWS2 Category**

The NEWS 2 will be categorized into its clinical risk according to the following categories:

- No clinical risk: (score 0)
- Low clinical risk: (score 1-4)
- Medium clinical risk: (score 5 6, or 1 individual parameter with a score 3)
- High clinical risk: (score 7 and more)

In case a parameter is missing to calculate the NEWS 2 but based on the available information the NEWS 2 is 7 or more, the NEWS2 category will be 'High clinical risk'.

# 7.6.2. Analysis Methods

Descriptive statistics of the NEWS2 and the change from baseline will be shown by analysis timepoint. Additionally, a mean +/- SE graph of the scores over time will be provided.

A frequency table of the ACVPU score by timepoint and treatment group will be provided. Include in this table the safety follow-up visit, the Day 28 final study visit and the last study visit.

A tabulation of the clinical risk categories will be made per analysis timepoint. Include in this table the safety follow-up visit, the Day 28 final study visit and the last study visit.

A listing of the NEWS2 by analysis timepoint for each subject will be provided.

#### 8. RESISTANCE

# 8.1. Viral Phenotype

The pimodivir  $EC_{50}$  and oseltamivir  $IC_{50}$  with their fold change values will be analyzed at baseline and at all post-baseline visits with available data (FC = fold change in  $EC_{50}$  (IC<sub>50</sub>) value).

FC is calculated as the EC50 (or IC50) of the subject's influenza strain divided by the EC50 (or IC50) of a reference strain. If the patient EC50 (or IC50) is censored, the fold change value gets the same censor, e.g. patient EC50 = >20 nM, reference EC50 = 4nM, Fold Change value >5.

The following output will be provided:

- Emerging phenotypic resistance: descriptive statistics for FC in EC<sub>50</sub> and IC<sub>50</sub> value for pimodivir and oseltamivir respectively at baseline and at all post-baseline visits with available data. The number (%) of subjects by treatment arm with censored phenotype data (by lower and upper bound) at baseline and at all post-baseline visits with available data will also be shown.
- Descriptive statistics for fold change ratio of all post-baseline visits with available data versus baseline including geometric mean and 95% CI.
- A listing showing viral load data together with phenotype data (EC<sub>50</sub>, IC<sub>50</sub> and fold change values) per subject and influenza subtype for all available timepoints including screening/baseline.

# 8.2. Viral Genotype

Assessment of viral sequences will be done to determine amino-acid substitutions that may be associated with resistance to pimodivir and to other influenza antivirals if present as part of the SOC. To that end, genotypic data for PB2, PB1, PA, NA, HA and optionally other genome segments of the influenza virus will be gathered.

All positions in the gathered regions will be analyzed for all samples, overall and by influenza subtype.

The gathered regions most relevant for pimodivir are PB2, PB1 and PA, those for neuraminidase inhibitors (NAI) (including oseltamivir) are NA and HA

The following 12 amino-acid positions in PB2 are of interest: 306, 323, 324, 325, 337, 357, 363, 376, 378, 404, 406, 431, and 510.

The following mutations in NA, associated with resistance to oseltamivir, are of interest:

- For subtype H1N1: D199N, I223R, H275Y, and N295S
- For subtype H3N2: E119V, H274Y, R292K, and N294S

The list of positions of interest might be updated during the analysis.

A mutation is treatment-emerging at a specific (post-baseline) time-point if the amino-acid of the considered position is absent at screening/baseline and present at that timepoint.

The baseline is the collection of all polymorphisms present at any timepoint up to the first intake of study. A table with an overview of the time points underlying the "baseline" will be generated.

Data will be summarized using frequency tabulations (n and %). Displays and individual mutations should be presented for each genome segment separately (i.e. PB1, PB2, PA, NA and HA separately). The following output will be provided:

- Baseline polymorphisms: number (%) of subjects with available genotype data, with any baseline polymorphism, and the number of subjects per polymorphism, for all polymorphisms, per treatment arm.
- Baseline polymorphisms: number (%) of subjects with any baseline polymorphism and with specific baseline polymorphisms at the positions of interest.
- Frequency tabulations for the presence of all emerging mutations overall post-baseline.
- Frequency tabulations for the presence of all emerging mutations overall post-baseline at positions of interest.
- Listing for genotype data per subject for all available timepoints including screening/baseline including viral load data (include influenza subtype and influenza subtype category). A patient profile will be created including this data supplemented with the phenotypic data.

# 9. PHARMACOKINETICS/PHARMACODYNAMICS

Blood samples for PK assessments of pimodivir will be collected at the Day 1, 3, 5, 6 and/or Day 7 visit depending on when the subject is discharged from the hospital.

Descriptive statistics of pimodivir plasma concentration over time will be tabulated for the PK analysis set.

# 9.1. Pharmacokinetics

Based on the individual plasma concentration-time data from all subjects, exposure parameters of pimodivir will be derived using population PK modelling. The following exposure parameters will be derived for the samples collected after the first intake (Day 1), after the 5<sup>th</sup> intake (Day 3) and after the last intake (the last intake can be on Day 5, 6 or 7 and will be reported as Day 5 in the tables): AUC<sub>12h</sub>, C<sub>trough</sub>, and, if feasible, C<sub>max</sub>, and T<sub>max</sub>.

Descriptive statistics, including arithmetic mean, standard deviation, coefficient of variation, geometric mean, median, minimum, maximum, and interquartile range will be calculated at available timepoints for all available parameters for the PK analysis set.

# 9.2. Pharmacokinetic/Pharmacodynamic Relationships

Pharmacokinetic/Pharmacodynamic relationships will be analyzed for the PD analysis set. The exposure parameters AUC<sub>12h</sub> and C<sub>trough</sub> will be categorized into quartiles for Day 1, Day 3 and Day 5 (i.e.: after the last intake, this can be on Day 5, Day 6 or Day 7) (if available). Relationships of these parameters with the primary and selected secondary efficacy endpoints will be explored as follows.

The distribution of subjects over the hospital recovery scale on Day 6 will be tabulated per quartile for each exposure parameter for each PK timepoint.

The number and percentage of subjects with treatment-emergent adjudicated influenza complications will be tabulated for each quartile for each exposure parameter for each PK timepoint.

The Kaplan Meier estimates for the time to hospital discharge will be produced per quartile for each exposure parameter for each PK timepoint.

The Kaplan Meier estimates for the time from ICU admission to ICU discharge will be produced per each quartile for each exposure parameter for each PK timepoint.

The Kaplan Meier estimates for the time to return to daily activities will be produced per quartile for each exposure parameter for each PK timepoint.

The Kaplan Meier estimates for the time from start of mechanical ventilation to end of mechanical ventilation will be produced per each quartile for each exposure parameter for each PK timepoint.

The number and percentage of subjects readmitted to the hospital after the first discharge will be tabulated for each quartile for each exposure parameter for each PK timepoint.

Relationships of AUC<sub>12h</sub> with safety will be explored as follows. The number and percentage of subjects with the following treatment-emergent adverse events by AUC<sub>12h</sub> quartile for each PK timepoint will be tabulated:

- Any AE
- AEs of worst grade 3 or 4
- Deaths due to AE
- Serious AEs
- AEs for which study drug was permanently stopped
- AEs at least possibly related to study drug
- Confirmed diarrhea events

A frequency table of the worst treatment-emergent toxicity grades versus AUC<sub>12h</sub> quartile will be presented for the laboratory parameters AST, ALT, and total bilirubin.

Separate frequency table will be produced for the worst treatment-emergent toxicity grades at each PK timepoint.

# 10. HEALTH ECONOMICS

Following medical resource utilization data will be explored

# 10.1. Definitions

| Measurement | Formula |
|---|---|
| Number of medical care encounters | Medical care encounters other than those mandated per trial protocol, including surgeries and other selected procedures (inpatient and outpatient), as recorded on the eCRF. The number of medical care encounters is derived as the frequency of the medical encounters other than those mandated in the protocol (eCRF). |
| Type of practitioner for hospital outpatient department encounters | Type of practitioner as recorded in the eCRF in case of Outpatient Department is selected. |
| Frequency of visits of outpatient medical care encounters | Frequency of visits will be provided per outpatient medical encounter type (Hospital Outpatient Department Laboratory Department, Medical Practitioner Office, Home Care) |
| Number of outpatient medical care encounters | Similar to the description for number of medical care encounters, but only for outpatient medical care encounters, as recorded on the eCRF (Hospital Outpatient Department, Laboratory Department, Medical Practitioner Office, Home Care). |

# 10.2. Analysis Methods

Frequency tabulations of medical care encounters, per category (as defined above) and by medical encounter type, will be provided.

Frequency tabulations of the frequency of visits will be provided, per following medical encounter types:

- Hospital Outpatient Department,
- Laboratory Department,
- Medical Practitioner Office,
- Home Care

Frequency tabulations of the type of practitioner will be provided, for the Hospital Outpatient Department.

# **REFERENCES**

- 1. Guideline, I. H. T. The clinical evaluation of QT/QTc interval prolongation and proarrhythmic potential for non-antiarrhythmic drugs E14. Recommended for adoption at Step; 2006; 4.
- 2. Herdman M., Gudex C., Lloyd A., Janssen M. F., Kind P., Parkin D., Bonsel G., Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Quality of Life Research. 2011; 20:1727-36
- 3. Hodges J.L., Lehmann E.L., Estimates of location based on rank tests. The Annals of Mathematical Statistics. 1963; 34:598-611
- 4. Hurst H., Bolton J. Assessing the clinical significance of change scores recorded on subjective outcome measures. J. Manipulative Physiol Ther. 2004;27:26-35.
- 5. Jaeschke R., Singer J., Guyatt G.H.. Measurement of health status. Ascertaining the minimal clinically important difference. Control Clin Trials. 1989;10(4):407-415.
- 6. Lehmann E. L. Nonparametric confidence intervals for a shift parameter. The Annals of Mathematical Statistics 1963; 34:1507–1512.
- 7. Royal College of Physicians of London. National early warning score (NEWS): standardising the assessment of acute-illness severity in the NHS; 2012. www.rcplondon.ac.uk/resources/national-earlywarning-score-news
- 8. Royal College of Physicians of London. National early warning score (NEWS) 2: standardising the assessment of acute-illness severity in the NHS; 2017. https://www.rcplondon.ac.uk/projects/outputs/national-early-warning-score-news-2
- 9. United Nations publication, Standard Country or Area Codes for Statistical Use (M49 standard), https://unstats.un.org/unsd/methodology/m49/
- 10. White, I. R., Royston, P., & Wood, A. M. (2011). Multiple imputation using chained equations: issues and guidance for practice. Statistics in medicine, 30(4), 377-399.
- 11. Whitehead J. Sample size calculations for ordered categorical data, 1993. Statistics in medicine; 12:2257-2271.
- 12. World Health Organization. "WHO toxicity grading scale for determining the severity of adverse events."; 2003

# **ATTACHMENTS**

# ATTACHMENT 1. : ANTICIPATED EVENTS AND ANTICIPATED EVENT GROUPS

Table 8 shows an overview of the anticipated event groups with group number.

Table 9 indicates which adverse event preferred terms (MedDRA PT) are Anticipated Events (AnE) and Closely Related Medical Events (ME) based on MedDRA Version 18.1. These adverse events will be classified as an Anticipated Event according to the protocol term and are grouped into Anticipated Event Groups.

**Table 8: Anticipated Event groups** 

| Group Number | Grouped Term |
|--------------|-----------------------------|
| Group 1 | Infections and infestations |
| Group 2 | Diabetic complications |

Table 9: Anticipated Events (AnE) and Closely Related Medical Events (ME).

| Protocol Term | AnE | ME | MedDRA PT * | MedDRA | Grouped Term | Group |
|---|---|---|---|---|---|---|
| | | | | Code* | | Number |
| Pneumonia | $\boxtimes$ | | Pneumonia | 10035664 | Infections and infestations | 1 |
| Pneumonia | | $\boxtimes$ | Enterobacter pneumonia | 10054218 | Infections and infestations | 1 |
| Pneumonia | | $\boxtimes$ | Pneumonia haemophilus | 10035702 | Infections and infestations | 1 |
| Pneumonia | | $\boxtimes$ | Pneumonia staphylococcal | 10035734 | Infections and infestations | 1 |
| Pneumonia | | $\boxtimes$ | Pneumonia streptococcal | 10035735 | Infections and infestations | 1 |
| Bronchitis | $\boxtimes$ | | Bronchitis | 10006451 | Infections and infestations | 1 |
| Bronchitis | | $\boxtimes$ | Bronchitis bacterial | 10061736 | Infections and infestations | 1 |
| Bronchitis | | $\boxtimes$ | Bronchitis haemophilus | 10006460 | Infections and infestations | 1 |
| Sinus infection | $\boxtimes$ | | Sinusitis <sup>1</sup> | 10040753 | Infections and infestations | 1 |
| Sinus infection | | $\boxtimes$ | Acute sinusitis <sup>1</sup> | 10001076 | Infections and infestations | 1 |

| Protocol Term | AnE | ME | MedDRA PT * | MedDRA | Grouped Term | Group |
|---|---|---|---|---|---|---|
| | | | | Code* | 1 | Number |
| Sinus infection | | $\boxtimes$ | Chronic sinusitis <sup>1</sup> | 10009137 | Infections and infestations | 1 |
| Sinus infection | | $\boxtimes$ | Viral sinusitis | 10051513 | Infections and infestations | 1 |
| Ear infection | $\boxtimes$ | | Ear infection | 10014011 | Infections and infestations | 1 |
| Ear infection | | $\boxtimes$ | Middle ear effusion | 10062545 | Infections and infestations | 1 |
| Ear infection | | $\boxtimes$ | Otitis externa | 10033072 | Infections and infestations | 1 |
| Ear infection | | $\boxtimes$ | Otitis media | 10033078 | Infections and infestations | 1 |
| Ear infection | | $\boxtimes$ | Otitis media acute | 10033079 | Infections and infestations | 1 |
| Worsening of asthma, asthma attack <sup>2</sup> | | $\boxtimes$ | Asthma | 10003553 | NA | |
| Worsening of asthma, asthma attack <sup>2</sup> | | $\boxtimes$ | Asthmatic crisis | 10064823 | NA | |
| Worsening of asthma, asthma attack <sup>2</sup> | | $\boxtimes$ | Status asthmaticus | 10041961 | NA | |
| COPD exacerbation <sup>3</sup> | $\boxtimes$ | | Chronic obstructive pulmonary disease | 10009033 | NA | |
| COPD exacerbation <sup>3</sup> | | $\boxtimes$ | Emphysema | 10014561 | NA | |
| Complications of sickle cell disease, sickle cell crisis <sup>4</sup> | | $\boxtimes$ | Sickle cell anaemia | 10040641 | NA | |
| Complications of sickle cell disease, sickle cell crisis <sup>4</sup> | | $\boxtimes$ | Sickle cell anaemia with crisis | 10040642 | NA | |
| Complications of sickle cell disease, sickle cell crisis <sup>4</sup> | | $\boxtimes$ | Acute chest syndrome | 10051895 | NA | |
| Complications of sickle cell disease, sickle cell crisis <sup>4</sup> | | $\boxtimes$ | Ischaemic stroke | 10061256 | NA | |
| Complications of sickle cell disease, sickle cell crisis <sup>4</sup> | | $\boxtimes$ | Embolic stroke | 10014498 | NA | |
| Complications of sickle cell disease, sickle cell crisis <sup>4</sup> | | $\boxtimes$ | Deep vein thrombosis | 10051055 | NA | |
| Complications of sickle cell disease, sickle cell crisis <sup>4</sup> | | $\boxtimes$ | Pulmonary embolism | 10037377 | NA | |
| Complications of diabetes mellitus, diabetic ketoacidosis <sup>4</sup> | | | Diabetic complication | 10061104 | Diabetic complications | 2 |

| Protocol Term | AnE | ME | MedDRA PT * | MedDRA | Grouped Term | Group |
|---|---|---|---|---|---|---|
| | | | | Code* | | Number |
| Complications of diabetes mellitus, diabetic ketoacidosis <sup>4</sup> | | | Diabetic ketoacidosis | 10012671 | Diabetic complications | 2 |
| Complications of diabetes mellitus, diabetic ketoacidosis <sup>4</sup> | | | Diabetes mellitus <sup>5</sup> | 10012601 | Diabetic complications | 2 |
| Complications of diabetes mellitus, diabetic ketoacidosis <sup>4</sup> | | | Diabetic ketoacidotic hyperglycaemic coma | 10012672 | Diabetic complications | 2 |
| Complications of diabetes mellitus, diabetic ketoacidosis <sup>4</sup> | | | Hypoglycaemia | 10020993 | Diabetic complications | 2 |
| Complications of diabetes mellitus diabetic ketoacidosis <sup>4</sup> | | | Diabetic metabolic decompensation | 100126655 | Diabetic complications | 2 |
| Acute Respiartory Distress Syndrome (ARDS) | $\boxtimes$ | | Acute respiratory distress syndrome | 10001052 | NA | |
| Acute Respiartory Distress Syndrome (ARDS) | | $\boxtimes$ | Acute respiratory failure <sup>6</sup> | 10001053 | NA | |

<sup>&</sup>lt;sup>1</sup> Infectious etiology only

<sup>&</sup>lt;sup>2</sup> Please note that asthma aggravated codes to a PT of asthma. These PTs will be considered as anticipated events <u>only</u> if the subjects have documented those conditions (such as: asthma, COPD, Sickle cell disease, or diabetes) before enrolling the study.

<sup>&</sup>lt;sup>3</sup> Please note that chronic obstructive airways disease exacerbated codes to a PT of chronic obstructive pulmonary disease. These PTs will be considered as anticipated events only if the subjects have documented those conditions (such as: asthma, COPD, Sickle cell disease, or diabetes) before enrolling the study.

<sup>&</sup>lt;sup>4</sup> These PTs will be considered as anticipated events only if the subjects have documented those conditions (such as: asthma, COPD, Sickle cell disease, or diabetes) before enrolling the study.

<sup>&</sup>lt;sup>5</sup> Please note that diabetes mellitus aggravated and diabetes mellitus exacerbated codes to a PT of diabetes mellitus.

<sup>&</sup>lt;sup>6</sup> This event will be considered anticipated only if it occurs in the context of ARDS

# ATTACHMENT 2. : WHO TOXICITY GRADING SCALE FOR DETERMINING THE SEVERITY OF ADVERSE EVENTS (FEB 2003)

# **ABBREVIATIONS** (used in the table):

ULN = Upper Limit of Normal LLN = Lower Limit of Normal

 $R_x = Therapy$  IV = Intravenous

 $FEV_1$  = forced expiratory volume in 1 second

# **ESTIMATING SEVERITY GRADE**

For abnormalities NOT found elsewhere in the Toxicity Tables use the scale below to estimate grade of severity:

| GRADE 1 | Mild | Transient or mild discomfort (<48 hours); no medical intervention/therapy required. |
|---|---|---|
| GRADE 2 | Moderate | Mild to moderate limitation in activity; some assistance may be needed; no or minimal medical intervention/therapy required. |
| GRADE 3 | Severe | Marked limitation in activity; some assistance usually required; medical intervention/therapy required; hospitalizations possible. |
| GRADE 4 | Potentially life-<br>threatening <sup>a</sup> | Extreme limitation in activity; significant assistance required; significant medical intervention/therapy required; hospitalization or hospice care probable. |

a Revised by the sponsor

# **COMMENTS REGARDING THE USE OF THESE TABLES**

- For parameters not included in the following Toxicity Tables, sites should refer to the "Guide For Estimating Severity Grade" located above.
- Criteria are generally grouped by body system. Some protocols may have additional protocolspecific grading criteria, which will supersede the use of these tables for specified criteria.

| Item | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hematology | | | | |
| Hemoglobin | 9.5-10.5 gm/dL | 8.0-9.4 gm/dL | 6.5-7.9 gm/dL | <6.5 gm/dL |
| Absolute<br>Neutrophil<br>Count | 1,000-<br>1,500/mm³ | 750-999/mm <sup>3</sup> | 500-749/mm³ | <500/mm <sup>3</sup> |
| Platelets | 75,000-<br>99,000/mm <sup>3</sup> | 50,000-<br>74,999/mm <sup>3</sup> | 20,000-<br>49,999/mm <sup>3</sup> | <20,000/mm³ |
| Prothrombin<br>Time (PT) | ≥1.01 to ≤1.25 x<br>ULN | >1.25 to ≤1.50 x<br>ULN | >1.50 to ≤3.00 x<br>ULN | >3.00 x ULN |
| Activated Partial<br>Thromboplastin<br>Time (aPTT) | ≥1.01 to ≤1.66 x<br>ULN | >1.66 to ≤2.33 x<br>ULN | >2.33 to ≤3.00 x<br>ULN | >3.00 x ULN |
| Fibrinogen | ≥0.75 to ≤0.99 x<br>LLN | ≥0.50 to <0.75 x<br>LLN | ≥0.25 to <0.50 x<br>LLN | <0.25 x LLN |
| Fibrin Split<br>Product | 20-40 mcg/mL | 41-50 mcg/mL | 51-60 mcg/mL | >60 mcg/mL |
| Methemoglobin | 5.0-9.9% | 10.0-14.9% | 15.0-19.9% | >20.0% |
| <b>Liver Enzymes</b> | | | | |
| AST (SGOT) | ≥1.25 to ≤2.50 x<br>ULN | >2.50 to ≤5.00 x<br>ULN | >5.00 to ≤10.00 x ULN | >10.00 x ULN |
| ALT (SGPT) | ≥1.25 to ≤2.50 x<br>ULN | >2.50 to ≤5.00 x<br>ULN | >5.00 to ≤10.00 x ULN | >10.00 x ULN |
| Gamma-<br>glutamyltransfer<br>ase | ≥1.25 to ≤2.50 x<br>ULN | >2.50 to ≤5.00 x<br>ULN | >5.00 to ≤10.00<br>x ULN | >10.00 x ULN |
| Alkaline<br>Phosphatase | ≥1.25 to ≤2.50 x<br>ULN | >2.50 to ≤5.00 x<br>ULN | >5.00 to ≤10.00 x ULN | >10.00 x ULN |
| Amylase | ≥1.1 to ≤1.5 x<br>ULN | >1.5 to ≤2.0 x<br>ULN | >2.0 to ≤5.0 x<br>ULN | >5.0 x ULN |

| Item | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Chemistries | | | | |
| Hyponatremia | 130-135 mEq/L | 123-129 mEq/L | 116-122 mEq/L | <116 mEq/L or<br>mental status<br>changes or<br>seizures |
| Hypernatremia | 146-150 mEq/L | 151-157 mEq/L | 158-165 mEq/L | >165 mEq/L or<br>mental status<br>changes or<br>seizures |
| Hypokalemia | 3.0-3.4 mEq/L | 2.5-2.9 mEq/L | 2.0-2.4 mEq/L or intensive replacement Rx required or hospitalization required | <2.0 mEq/L or paresis or ileus or life-threatening arrhythmia |
| Hyperkalemia | 5.6-6.0 mEq/L | 6.1-6.5 mEq/L | 6.6-7.0 mEq/L | >7.0 mEq/L or life-threatening arrhythmia |
| Hypoglycemia | 55-64 mg/dL | 40-54 mg/dL | 30-39 mg/dL | <30 mg/dL or<br>mental status<br>changes or<br>coma |
| Hyperglycemia (note if fasting) | 116-160 mg/dL | 161-250 mg/dL | 251-500 mg/dL | >500 mg/dL or<br>ketoacidosis or<br>seizures |
| Hypocalcemia<br>(corrected for<br>albumin) | 8.4-7.8 mg/dL | 7.7-7.0 mg/dL | 6.9-6.1 mg/dL | <6.1 mg/dL or life-threatening arrhythmia or tetany |
| Hypercalcemia<br>(corrected for<br>albumin) | 10.6-11.5 mg/dL | 11.6-12.5 mg/dL | 12.6-13.5 mg/dL | >13.5 mg/dL<br>or life-<br>threatening<br>arrhythmia |

| Item | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hypomagnesem ia | 1.4-1.2 mEq/L | 1.1-0.9 mEq/L | 0.8-0.6 mEq/L | <0.6 mEq/L or life-threatening arrhythmia |
| Hypophosphate<br>mia | 2.0-2.4 mg/dL | 1.5-1.9 mg/dL or<br>replacement Rx<br>required | 1.0-1.4 mg/dL<br>intensive Rx or<br>hospitalization<br>required | <1.0 mg/dL or life-threatening arrhythmia |
| Hyperbilirubine mia | ≥1.1 to ≤1.5 x<br>ULN | >1.5 to ≤2.5 x<br>ULN | >2.5 to ≤5.0 x<br>ULN | >5.0 x ULN |
| BUN | ≥1.25 to ≤2.50 x<br>ULN | >2.50 to ≤5.00 x<br>ULN | >5.00 to ≤10.00 x ULN | >10.00 x ULN |
| CPK* | 3 to <6 x ULN | 6 to <10 x ULN | 10 to <20 x ULN | ≥20 x ULN |
| Creatinine | ≥1.1 to ≤1.5 x ULN | >1.5 to ≤3.0 x ULN | >3.0 to ≤6.0 x ULN | >6.0 x ULN or required dialysis |
| Lipase* | 1.1 to <1.5 x ULN | 1.5 to <3.0 x ULN | 3.0 to <5.0 x ULN | ≥5.0 x ULN |
| * Grading based on I | | DS) Table for Grading t | he Severity of Adult an | d Pediatric Adverse |

Events, version 2.0, November 2014.

| Urinalysis | | | | |
|---|---|---|---|---|
| Proteinuria | 1+ or <0.3% or <3g/L or 200 mg - 1 gm loss/day | or 3-10 g/L or | 4+ or >1.0% or<br>>10 g/L or<br>2-3.5 gm<br>loss/day | nephrotic<br>syndrome or<br>>3.5 gm<br>loss/day |
| Hematuria Cardiac Dysfunc | microscopic only | gross, no clots | gross + clots | obstructive or<br>required<br>transfusion |
| Cardiac Dysiunc | tion | | | |
| Cardiac Rhythm | - | asymptomatic,<br>transient signs,<br>no Rx required | recurrent/persist<br>ent; no Rx<br>required | requires Rx |
| Hypertension | transient inc. >20 mm; no Rx | recurrent,<br>chronic, > 20<br>mm, Rx required | requires acute Rx; no hospitalization | requires<br>hospitalization |

| Item | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hypotension | transient orthostatic hypotension, no Rx | symptoms<br>correctable with<br>oral fluids Rx | requires IV<br>fluids; no<br>hospitalization<br>required | requires<br>hospitalization |
| Pericarditis | minimal effusion | mild/moderate<br>asymptomatic<br>effusion, no Rx | symptomatic<br>effusion; pain;<br>ECG changes | tamponade;<br>pericardiocente<br>sis or surgery<br>required |
| Hemorrhage,<br>Blood Loss | microscopic/occu<br>lt | mild, no<br>transfusion | gross blood loss;<br>1-2 units<br>transfused | massive blood<br>loss; >3 units<br>transfused |
| Respiratory | | | | |
| Cough | transient; no Rx | treatment associated cough; local Rx | uncontrolled | - |
| Bronchospasm,<br>Acute | transient; no Rx<br><80-70% FEV <sub>1</sub><br>(or peak flow) | requires Rx<br>normalizes with<br>bronchodilator;<br>FEV <sub>1</sub> 50-70%<br>(or peak flow) | no normalization with bronchodilator; FEV <sub>1</sub> 25-50% (or peak flow retractions) | cyanosis: FEV <sub>1</sub> <25% (or peak flow) or intubated |
| Gastrointestinal | | | | |
| Stomatitis | mild discomfort;<br>no limits on<br>activity | some limits on eating/drinking | eating/talking<br>very limited | requires IV fluids |
| Nausea | mild discomfort;<br>maintains<br>reasonable<br>intake | moderate<br>discomfort;<br>intake decreased<br>significantly;<br>some activity<br>limited | severe<br>discomfort; no<br>significant<br>intake; activities<br>limited | minimal fluid<br>intake |

| Item | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Vomiting | transient emesis | occasional/moder<br>ate vomiting | orthostatic<br>hypotension or<br>IV fluids<br>required | hypotensive<br>shock or<br>hospitalization<br>required for IV<br>fluid therapy |
| Constipation | mild | moderate | severe | distensions<br>w/vomiting |
| Diarrhea | transient 3-4 loose stools/day | 5-7 loose stools/day | orthostatic hypotension or >7 loose stools/day or required IV fluids | hypotensive<br>shock or<br>hospitalization<br>for IV fluid<br>therapy<br>required |
| Neuro & Neuron | nuscular | | | |
| Neuro-<br>Cerebellar | slight<br>incoordination<br>dysdiadochokine<br>sis | intention tremor,<br>dysmetria, slurred<br>speech;<br>nystagmus | locomotor ataxia | incapacitated |
| Mood | mild anxiety or<br>depression | moderate anxiety<br>or depression and<br>Rx required | severe anxiety or<br>depression or<br>mania; needs<br>assistance | acute<br>psychosis;<br>incapacitated,<br>requires<br>hospitalization |
| Neuro Control (ADL = activities of daily living) | mild difficulty concentrating; no Rx; mild confusion/agitati on; ADL unaffected | moderate confusion/agitati on some limitation of ADL; minimal Rx | severe confusion/agitati on needs assistance for ADL; Rx required | toxic<br>psychosis;<br>hospitalization |
| Muscle Strength | subjective weakness no objective symptoms/ signs | mild objective<br>signs/symptoms<br>no decrease in<br>function | objective<br>weakness<br>function limited | paralysis |
| Other Parameter | rs | | | |

| Item | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Fever: oral, >12 hours | 37.7-38.5 °C or 100.0-101.5 °F | 38.6-39.5 °C or<br>101.6-102.9 °F | 39.6-40.5 °C or<br>103-105 °F | >40.5 °C or<br>>105 °F |
| Headache | mild, no Rx | transient, moderate; Rx required | severe; responds<br>to initial narcotic<br>therapy | intractable;<br>required<br>repeated<br>narcotic<br>therapy |
| Fatigue | no decrease in ADL | normal activity<br>decreased 25-<br>50% | normal activity<br>decreased >50%<br>can't work | unable to care for self |
| Allergic<br>Reaction | pruritus without rash | localized urticaria | generalized<br>urticaria;<br>angioedema | anaphylaxis |
| Local Reaction | tenderness or<br>erythema | induration <10<br>cm or phlebitis or<br>inflammation | induration >10 cm or ulceration | necrosis |
| Mucocutaneous | Erythema;<br>pruritus | diffuse, maculopapular rash, dry desquamation | vesiculation,<br>moist<br>desquamation, or<br>ulceration | exfoliative dermatitis, mucous membrane involvement, or erythema multiforme or suspected Stevens- Johnson or necrosis requiring surgery |

# ATTACHMENT 3. : WHO GRADING SCALE VITAL SIGNS

The following abnormalities are defined for vital signs:

| | | Vital Signs parameter | |
|---|---|---|---|
| Abnormality Code Pulse | | Code Pulse DBP* | |
| Abnormalities on actual v | alues | | |
| Abnormally low | < 45 bpm | ≤ 50 mmHg | ≤ 90 mmHg |
| Grade 1 or mild | | > 90 mmHg - < 100 mmHg | > 140 mmHg - < 160 mmHg |
| Grade 2 or moderate | - | $\geq 100 \text{ mmHg} - < 110 \text{ mmHg}$ | $\geq$ 160 mmHg - < 180 mmHg |
| Grade 3 or severe | - | ≥ 110 mmHg | ≥ 180 mmHg |
| Abnormally high | ≥ 120 bpm | - | - |

<sup>\*</sup> The classification of AEs related to hypotension and hypertension will be done according to the WHO grading scale

| | Vital Signs parameter | | |
|---|---|---|---|
| Abnormality Code | Temperature (°C/°F) | Respiratory rate (breaths per minute) | Oxygen Saturation (%) |
| Normal | | | ≥95% - 100% |
| Grade 1 or mild | 37.7 - 38.5 °C or<br>100.0 - 101.5 °F | 17-20 | ≥90% - <95% |
| Grade 2 or moderate | 38.6 - 39.5 °C or<br>101.6 - 102.9 °F | 21-25 | ≥85% - <90% |
| Grade 3 or severe | 39.6 - 40.5 °C or<br>103.0 - 105.0 °F | >25 | <85% |
| Grade 4 or potentially life-threatening | >40.5°C or<br>>105.0°F | | |

# ATTACHMENT 4. : ECG ABNORMALITIES

The following abnormalities are defined for ECG:

| | | ECG parameter | | |
|---|---|---|---|---|
| Abnormality Code | HR | PR | QRS | QT <sub>corrected</sub> |
| Abnormalities on actual values | | | | |
| Abnormally low | < 45 bpm | < 110 ms | - | - |
| Abnormally high | ≥ 120 bpm | > 220 ms | ≥ 120 ms | - |
| Borderline prolonged QT (males) | - | - | - | $450 \text{ ms} < \text{QTc} \le 480 \text{ ms}$ |
| Borderline prolonged QT (females) | - | - | - | $470 \text{ ms} < \text{QTc} \le 480 \text{ ms}$ |
| Prolonged QT | - | - | - | $480 \text{ ms} < \text{QTc} \le 500 \text{ ms}$ |
| Pathologically prolonged QT | - | - | - | QTc > 500 ms |
| Abnormalities on changes from base | line (ΔQTc) | | | |
| Normal QTc change | - | - | - | $\Delta QTc < 30 \text{ ms}$ |
| Borderline QTc change | - | - | - | $30 \text{ ms} \leq \Delta QTc \leq 60 \text{ ms}$ |
| Abnormally high QTc change | - | - | - | $\Delta QTc > 60 \text{ ms}$ |

# ATTACHMENT 5. : EQ-5D VALUATION INDEX

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 11111 | 1 | 11242 | 0,498 | 11423 | 0,606 | 11554 | 0,018 |
| 11112 | 0,879 | 11243 | 0,484 | 11424 | 0,437 | 11555 | -0,066 |
| 11113 | 0,848 | 11244 | 0,323 | 11425 | 0,26 | 12111 | 0,846 |
| 11114 | 0,635 | 11245 | 0,157 | 11431 | 0,653 | 12112 | 0,779 |
| 11115 | 0,414 | 11251 | 0,235 | 11432 | 0,596 | 12113 | 0,761 |
| 11121 | 0,837 | 11252 | 0,179 | 11433 | 0,582 | 12114 | 0,548 |
| 11122 | 0,768 | 11253 | 0,164 | 11434 | 0,412 | 12115 | 0,327 |
| 11123 | 0,75 | 11254 | 0,083 | 11435 | 0,236 | 12121 | 0,737 |
| 11124 | 0,537 | 11255 | -0,001 | 11441 | 0,475 | 12122 | 0,678 |
| 11125 | 0,316 | 11311 | 0,883 | 11442 | 0,419 | 12123 | 0,663 |
| 11131 | 0,796 | 11312 | 0,827 | 11443 | 0,404 | 12124 | 0,45 |
| 11132 | 0,74 | 11313 | 0,812 | 11444 | 0,27 | 12125 | 0,229 |
| 11133 | 0,725 | 11314 | 0,599 | 11445 | 0,131 | 12131 | 0,709 |
| 11134 | 0,512 | 11315 | 0,378 | 11451 | 0,209 | 12132 | 0,653 |
| 11135 | 0,291 | 11321 | 0,785 | 11452 | 0,153 | 12133 | 0,638 |
| 11141 | 0,584 | 11322 | 0,728 | 11453 | 0,138 | 12134 | 0,425 |
| 11142 | 0,527 | 11323 | 0,714 | 11454 | 0,057 | 12135 | 0,204 |
| 11143 | 0,513 | 11324 | 0,501 | 11455 | -0,027 | 12141 | 0,497 |
| 11144 | 0,352 | 11325 | 0,28 | 11511 | 0,556 | 12142 | 0,441 |
| 11145 | 0,186 | 11331 | 0,76 | 11512 | 0,5 | 12143 | 0,426 |
| 11151 | 0,264 | 11332 | 0,704 | 11513 | 0,485 | 12144 | 0,266 |
| 11152 | 0,208 | 11333 | 0,689 | 11514 | 0,404 | 12145 | 0,099 |
| 11153 | 0,193 | 11334 | 0,476 | 11515 | 0,32 | 12151 | 0,177 |
| 11154 | 0,112 | 11335 | 0,255 | 11521 | 0,458 | 12152 | 0,121 |
| 11155 | 0,028 | 11341 | 0,548 | 11522 | 0,401 | 12153 | 0,106 |
| 11211 | 0,906 | 11342 | 0,491 | 11523 | 0,387 | 12154 | 0,025 |
| 11212 | 0,837 | 11343 | 0,477 | 11524 | 0,306 | 12155 | -0,059 |
| 11213 | 0,819 | 11344 | 0,316 | 11525 | 0,222 | 12211 | 0,806 |
| 11214 | 0,606 | 11345 | 0,15 | 11531 | 0,433 | 12212 | 0,748 |
| 11215 | 0,385 | 11351 | 0,228 | 11532 | 0,377 | 12213 | 0,733 |
| 11221 | 0,795 | 11352 | 0,172 | 11533 | 0,362 | 12214 | 0,52 |
| 11222 | 0,736 | 11353 | 0,157 | 11534 | 0,281 | 12215 | 0,299 |
| 11223 | 0,721 | 11354 | 0,076 | 11535 | 0,197 | 12221 | 0,706 |
| 11224 | 0,508 | 11355 | -0,008 | 11541 | 0,328 | 12222 | 0,649 |
| 11225 | 0,287 | 11411 | 0,776 | 11542 | 0,272 | 12223 | 0,634 |
| 11231 | 0,767 | 11412 | 0,719 | 11543 | 0,257 | 12224 | 0,421 |
| 11232 | 0,711 | 11413 | 0,705 | 11544 | 0,176 | 12225 | 0,2 |
| 11233 | 0,696 | 11414 | 0,535 | 11545 | 0,092 | 12231 | 0,681 |
| 11234 | 0,483 | 11415 | 0,359 | 11551 | 0,17 | 12232 | 0,624 |
| 11235 | 0,262 | 11421 | 0,677 | 11552 | 0,114 | 12233 | 0,61 |
| 11241 | 0,555 | 11422 | 0,621 | 11553 | 0,099 | 12234 | 0,397 |

| | | | | | Statistical | Allaly SIS I lai | 1 030230721 LLS |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 12235 | 0,176 | 12424 | 0,35 | 13113 | 0,744 | 13252 | 0,075 |
| 12241 | 0,468 | 12425 | 0,174 | 13114 | 0,531 | 13253 | 0,06 |
| 12242 | 0,412 | 12431 | 0,566 | 13115 | 0,31 | 13254 | -0,021 |
| 12243 | 0,397 | 12432 | 0,51 | 13121 | 0,717 | 13255 | -0,105 |
| 12244 | 0,237 | 12433 | 0,495 | 13122 | 0,66 | 13311 | 0,779 |
| 12245 | 0,071 | 12434 | 0,325 | 13123 | 0,646 | 13312 | 0,723 |
| 12251 | 0,149 | 12435 | 0,149 | 13124 | 0,433 | 13313 | 0,708 |
| 12252 | 0,092 | 12441 | 0,389 | 13125 | 0,212 | 13314 | 0,495 |
| 12253 | 0,078 | 12442 | 0,332 | 13131 | 0,692 | 13315 | 0,274 |
| 12254 | -0,003 | 12443 | 0,318 | 13132 | 0,636 | 13321 | 0,681 |
| 12255 | -0,088 | 12444 | 0,184 | 13133 | 0,621 | 13322 | 0,624 |
| 12311 | 0,796 | 12445 | 0,044 | 13134 | 0,408 | 13323 | 0,61 |
| 12312 | 0,74 | 12451 | 0,122 | 13135 | 0,187 | 13324 | 0,397 |
| 12313 | 0,725 | 12452 | 0,066 | 13141 | 0,48 | 13325 | 0,176 |
| 12314 | 0,512 | 12453 | 0,051 | 13142 | 0,423 | 13331 | 0,656 |
| 12315 | 0,291 | 12454 | -0,03 | 13143 | 0,409 | 13332 | 0,6 |
| 12313 | 0,698 | 12455 | -0,114 | 13144 | 0,248 | 13333 | 0,585 |
| 12321 | 0,642 | 12511 | 0,469 | 13145 | 0,082 | 13334 | 0,372 |
| 12322 | 0,627 | 12512 | 0,409 | 13143 | 0,082 | 13335 | 0,151 |
| 12323 | | | | | 0,104 | | 0,131 |
| | 0,414 | 12513 | 0,398 | 13152 | | 13341 | |
| 12325 | 0,193 | 12514 | 0,317 | 13153 | 0,089 | 13342 | 0,387 |
| 12331 | 0,673 | 12515 | 0,233 | 13154 | 0,008 | 13343 | 0,373 |
| 12332 | 0,617 | 12521 | 0,371 | 13155 | -0,076 | 13344 | 0,212 |
| 12333 | 0,602 | 12522 | 0,315 | 13211 | 0,786 | 13345 | 0,046 |
| 12334 | 0,389 | 12523 | 0,3 | 13212 | 0,73 | 13351 | 0,124 |
| 12335 | 0,168 | 12524 | 0,219 | 13213 | 0,715 | 13352 | 0,068 |
| 12341 | 0,461 | 12525 | 0,135 | 13214 | 0,502 | 13353 | 0,053 |
| 12342 | 0,405 | 12531 | 0,346 | 13215 | 0,281 | 13354 | -0,028 |
| 12343 | 0,39 | 12532 | 0,29 | 13221 | 0,688 | 13355 | -0,112 |
| 12344 | 0,23 | 12533 | 0,275 | 13222 | 0,631 | 13411 | 0,672 |
| 12345 | 0,063 | 12534 | 0,194 | 13223 | 0,617 | 13412 | 0,615 |
| 12351 | 0,141 | 12535 | 0,11 | 13224 | 0,404 | 13413 | 0,601 |
| 12352 | 0,085 | 12541 | 0,241 | 13225 | 0,183 | 13414 | 0,431 |
| 12353 | 0,07 | 12542 | 0,185 | 13231 | 0,663 | 13415 | 0,255 |
| 12354 | -0,011 | 12543 | 0,17 | 13232 | 0,607 | 13421 | 0,573 |
| 12355 | -0,095 | 12544 | 0,089 | 13233 | 0,592 | 13422 | 0,517 |
| 12411 | 0,689 | 12545 | 0,005 | 13234 | 0,379 | 13423 | 0,502 |
| 12412 | 0,633 | 12551 | 0,083 | 13235 | 0,158 | 13424 | 0,333 |
| 12413 | 0,618 | 12552 | 0,027 | 13241 | 0,451 | 13425 | 0,156 |
| 12414 | 0,448 | 12553 | 0,012 | 13242 | 0,394 | 13431 | 0,549 |
| 12415 | 0,272 | 12554 | -0,069 | 13243 | 0,38 | 13432 | 0,492 |
| 12421 | 0,591 | 12555 | -0,153 | 13244 | 0,219 | 13433 | 0,478 |
| 12422 | 0,534 | 13111 | 0,815 | 13245 | 0,053 | 13434 | 0,308 |
| 12423 | 0,52 | 13112 | 0,759 | 13251 | 0,131 | 13435 | 0,132 |

| | | | | | Statistical | Anaiysis Piai | 1 030238/2FLZ3 |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 13441 | 0,371 | 14125 | 0,185 | 14314 | 0,435 | 14453 | 0,007 |
| 13442 | 0,315 | 14131 | 0,6 | 14315 | 0,247 | 14454 | -0,074 |
| 13443 | 0,3 | 14132 | 0,544 | 14321 | 0,588 | 14455 | -0,158 |
| 13444 | 0,166 | 14133 | 0,529 | 14322 | 0,532 | 14511 | 0,425 |
| 13445 | 0,027 | 14134 | 0,348 | 14323 | 0,517 | 14512 | 0,369 |
| 13451 | 0,105 | 14135 | 0,16 | 14324 | 0,337 | 14513 | 0,354 |
| 13452 | 0,049 | 14141 | 0,414 | 14325 | 0,149 | 14514 | 0,273 |
| 13453 | 0,034 | 14142 | 0,357 | 14331 | 0,564 | 14515 | 0,189 |
| 13454 | -0,047 | 14143 | 0,343 | 14332 | 0,508 | 14521 | 0,327 |
| 13455 | -0,131 | 14144 | 0,202 | 14333 | 0,493 | 14522 | 0,27 |
| 13511 | 0,452 | 14145 | 0,055 | 14334 | 0,312 | 14523 | 0,256 |
| 13512 | 0,396 | 14151 | 0,133 | 14335 | 0,124 | 14524 | 0,175 |
| 13513 | 0,381 | 14152 | 0,077 | 14341 | 0,378 | 14525 | 0,091 |
| 13514 | 0,3 | 14153 | 0,062 | 14342 | 0,321 | 14531 | 0,302 |
| 13515 | 0,216 | 14154 | -0,019 | 14343 | 0,307 | 14532 | 0,246 |
| 13521 | 0,354 | 14155 | -0,103 | 14344 | 0,166 | 14533 | 0,231 |
| 13522 | 0,297 | 14211 | 0,694 | 14345 | 0,019 | 14534 | 0,15 |
| 13523 | 0,287 | 14211 | 0,638 | 14351 | 0,019 | 14535 | 0,066 |
| 13524 | 0,202 | 14212 | 0,623 | 14351 | 0,041 | 14533 | 0,197 |
| 13525 | | | | 14352 | 0,041 | 14541 | 0,197 |
| | 0,118 | 14214 | 0,442 | | | | · · |
| 13531 | 0,329 | 14215 | 0,254 | 14354 | -0,055 | 14543 | 0,126 |
| 13532 | 0,273 | 14221 | 0,596 | 14355 | -0,139 | 14544 | 0,045 |
| 13533 | 0,258 | 14222 | 0,539 | 14411 | 0,601 | 14545 | -0,039 |
| 13534 | 0,177 | 14223 | 0,525 | 14412 | 0,545 | 14551 | 0,039 |
| 13535 | 0,093 | 14224 | 0,344 | 14413 | 0,53 | 14552 | -0,017 |
| 13541 | 0,224 | 14225 | 0,156 | 14414 | 0,382 | 14553 | -0,032 |
| 13542 | 0,168 | 14231 | 0,571 | 14415 | 0,228 | 14554 | -0,113 |
| 13543 | 0,153 | 14232 | 0,515 | 14421 | 0,502 | 14555 | -0,197 |
| 13544 | 0,072 | 14233 | 0,5 | 14422 | 0,446 | 15111 | 0,436 |
| 13545 | -0,012 | 14234 | 0,319 | 14423 | 0,431 | 15112 | 0,38 |
| 13551 | 0,066 | 14235 | 0,131 | 14424 | 0,283 | 15113 | 0,365 |
| 13552 | 0,01 | 14241 | 0,385 | 14425 | 0,13 | 15114 | 0,284 |
| 13553 | -0,005 | 14242 | 0,328 | 14431 | 0,478 | 15115 | 0,2 |
| 13554 | -0,086 | 14243 | 0,314 | 14432 | 0,422 | 15121 | 0,338 |
| 13555 | -0,17 | 14244 | 0,173 | 14433 | 0,407 | 15122 | 0,281 |
| 14111 | 0,723 | 14245 | 0,026 | 14434 | 0,259 | 15123 | 0,267 |
| 14112 | 0,667 | 14251 | 0,104 | 14435 | 0,105 | 15124 | 0,186 |
| 14113 | 0,652 | 14252 | 0,048 | 14441 | 0,318 | 15125 | 0,102 |
| 14114 | 0,471 | 14253 | 0,033 | 14442 | 0,262 | 15131 | 0,313 |
| 14115 | 0,283 | 14254 | -0,048 | 14443 | 0,247 | 15132 | 0,257 |
| 14121 | 0,624 | 14255 | -0,132 | 14444 | 0,126 | 15133 | 0,242 |
| 14122 | 0,568 | 14311 | 0,687 | 14445 | 0 | 15134 | 0,161 |
| 14123 | 0,553 | 14312 | 0,631 | 14451 | 0,078 | 15135 | 0,077 |
| 14124 | 0,373 | 14313 | 0,616 | 14452 | 0,022 | 15141 | 0,208 |

| | | | | | Statistical | Allaly SIS I lai | 1 030230721 LZ3 |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 15142 | 0,152 | 15331 | 0,277 | 21115 | 0,357 | 21254 | 0,026 |
| 15143 | 0,137 | 15332 | 0,221 | 21121 | 0,767 | 21255 | -0,058 |
| 15144 | 0,056 | 15333 | 0,206 | 21122 | 0,708 | 21311 | 0,826 |
| 15145 | -0,028 | 15334 | 0,125 | 21123 | 0,693 | 21312 | 0,77 |
| 15151 | 0,05 | 15335 | 0,041 | 21124 | 0,48 | 21313 | 0,755 |
| 15152 | -0,006 | 15341 | 0,172 | 21125 | 0,259 | 21314 | 0,542 |
| 15153 | -0,021 | 15342 | 0,116 | 21131 | 0,739 | 21315 | 0,321 |
| 15154 | -0,102 | 15343 | 0,101 | 21132 | 0,683 | 21321 | 0,728 |
| 15155 | -0,186 | 15344 | 0,02 | 21133 | 0,668 | 21322 | 0,671 |
| 15211 | 0,407 | 15345 | -0,064 | 21134 | 0,455 | 21323 | 0,657 |
| 15212 | 0,351 | 15351 | 0,014 | 21135 | 0,234 | 21324 | 0,444 |
| 15213 | 0,336 | 15352 | -0,042 | 21141 | 0,527 | 21325 | 0,223 |
| 15214 | 0,255 | 15353 | -0,057 | 21142 | 0,47 | 21323 | 0,703 |
| 15215 | 0,171 | 15354 | -0,138 | 21143 | 0,456 | 21332 | 0,647 |
| 15221 | 0,309 | 15355 | -0,222 | 21144 | 0,296 | 21333 | 0,632 |
| 15222 | 0,252 | 15411 | 0,381 | 21145 | 0,129 | 21333 | 0,419 |
| 15223 | 0,232 | 15411 | 0,325 | 21143 | 0,129 | 21335 | 0,198 |
| 15223 | 0,238 | 15412 | , and the second | 21151 | 0,207 | | 0,198 |
| | · · | | 0,31 | | , and the second | 21341 | |
| 15225 | 0,073 | 15414 | 0,229 | 21153 | 0,136 | 21342 | 0,434 |
| 15231 | 0,284 | 15415 | 0,145 | 21154 | 0,055 | 21343 | 0,42 |
| 15232 | 0,228 | 15421 | 0,282 | 21155 | -0,029 | 21344 | 0,26 |
| 15233 | 0,213 | 15422 | 0,226 | 21211 | 0,836 | 21345 | 0,093 |
| 15234 | 0,132 | 15423 | 0,211 | 21212 | 0,778 | 21351 | 0,171 |
| 15235 | 0,048 | 15424 | 0,13 | 21213 | 0,762 | 21352 | 0,115 |
| 15241 | 0,179 | 15425 | 0,046 | 21214 | 0,549 | 21353 | 0,1 |
| 15242 | 0,123 | 15431 | 0,258 | 21215 | 0,328 | 21354 | 0,019 |
| 15243 | 0,108 | 15432 | 0,202 | 21221 | 0,735 | 21355 | -0,065 |
| 15244 | 0,027 | 15433 | 0,187 | 21222 | 0,679 | 21411 | 0,719 |
| 15245 | -0,057 | 15434 | 0,106 | 21223 | 0,664 | 21412 | 0,663 |
| 15251 | 0,021 | 15435 | 0,022 | 21224 | 0,451 | 21413 | 0,648 |
| 15252 | -0,035 | 15441 | 0,153 | 21225 | 0,23 | 21414 | 0,478 |
| 15253 | -0,05 | 15442 | 0,097 | 21231 | 0,71 | 21415 | 0,302 |
| 15254 | -0,131 | 15443 | 0,082 | 21232 | 0,654 | 21421 | 0,62 |
| 15255 | -0,215 | 15544 | -0,038 | 21233 | 0,639 | 21422 | 0,564 |
| 15311 | 0,4 | 15545 | -0,122 | 21234 | 0,426 | 21423 | 0,549 |
| 15312 | 0,344 | 15551 | -0,044 | 21235 | 0,205 | 21424 | 0,38 |
| 15313 | 0,329 | 15552 | -0,1 | 21241 | 0,498 | 21425 | 0,204 |
| 15314 | 0,248 | 15553 | -0,115 | 21242 | 0,442 | 21431 | 0,596 |
| 15315 | 0,164 | 15554 | -0,196 | 21243 | 0,427 | 21432 | 0,54 |
| 15321 | 0,302 | 15555 | -0,28 | 21244 | 0,267 | 21433 | 0,525 |
| 15322 | 0,245 | 21111 | 0,877 | 21245 | 0,1 | 21434 | 0,355 |
| 15323 | 0,231 | 21112 | 0,809 | 21251 | 0,178 | 21435 | 0,179 |
| 15324 | 0,15 | 21113 | 0,791 | 21252 | 0,122 | 21441 | 0,419 |
| 15325 | 0,066 | 21114 | 0,578 | 21253 | 0,107 | 21442 | 0,362 |

| | | | | | Statistical | Anaiysis Piai | 1 030238/2FLZ |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 21443 | 0,348 | 22132 | 0,596 | 22321 | 0,641 | 22455 | -0,17 |
| 21444 | 0,213 | 22133 | 0,582 | 22322 | 0,585 | 22511 | 0,413 |
| 21445 | 0,074 | 22134 | 0,369 | 22323 | 0,57 | 22512 | 0,356 |
| 21451 | 0,152 | 22135 | 0,148 | 22324 | 0,357 | 22513 | 0,342 |
| 21452 | 0,096 | 22141 | 0,44 | 22325 | 0,136 | 22514 | 0,261 |
| 21453 | 0,081 | 22142 | 0,384 | 22331 | 0,617 | 22515 | 0,177 |
| 21454 | 0 | 22143 | 0,369 | 22332 | 0,56 | 22521 | 0,314 |
| 21455 | -0,084 | 22144 | 0,209 | 22333 | 0,546 | 22522 | 0,258 |
| 21511 | 0,499 | 22145 | 0,043 | 22334 | 0,333 | 22523 | 0,243 |
| 21512 | 0,443 | 22151 | 0,121 | 22335 | 0,112 | 22524 | 0,162 |
| 21513 | 0,428 | 22152 | 0,064 | 22341 | 0,404 | 22525 | 0,078 |
| 21514 | 0,347 | 22153 | 0,05 | 22342 | 0,348 | 22531 | 0,29 |
| 21515 | 0,263 | 22154 | -0,031 | 22343 | 0,333 | 22532 | 0,233 |
| 21521 | 0,401 | 22155 | -0,115 | 22344 | 0,173 | 22533 | 0,219 |
| 21522 | 0,344 | 22211 | 0,747 | 22345 | 0,007 | 22534 | 0,138 |
| 21523 | 0,33 | 22212 | 0,691 | 22351 | 0,085 | 22535 | 0,054 |
| 21524 | 0,249 | 22213 | 0,676 | 22352 | 0,028 | 22541 | 0,185 |
| 21525 | 0,165 | 22213 | 0,463 | 22353 | 0,028 | 22542 | 0,128 |
| 21523 | 0,103 | 22214 | 0,242 | 22354 | -0,067 | 22543 | 0,128 |
| 21531 | | 22221 | 0,648 | 22355 | -0,067 | 22544 | 0,033 |
| | 0,32 | | • | | | | • |
| 21533 | 0,305 | 22222 | 0,592 | 22411 | 0,632 | 22545 | -0,051 |
| 21534 | 0,224 | 22223 | 0,577 | 22412 | 0,576 | 22551 | 0,027 |
| 21535 | 0,14 | 22224 | 0,364 | 22413 | 0,561 | 22552 | -0,03 |
| 21541 | 0,271 | 22225 | 0,143 | 22414 | 0,392 | 22553 | -0,044 |
| 21542 | 0,215 | 22231 | 0,624 | 22415 | 0,216 | 22554 | -0,125 |
| 21543 | 0,2 | 22232 | 0,567 | 22421 | 0,534 | 22555 | -0,209 |
| 21544 | 0,119 | 22233 | 0,553 | 22422 | 0,477 | 23111 | 0,758 |
| 21545 | 0,035 | 22234 | 0,34 | 22423 | 0,463 | 23112 | 0,702 |
| 21551 | 0,113 | 22235 | 0,119 | 22424 | 0,293 | 23113 | 0,687 |
| 21552 | 0,057 | 22241 | 0,411 | 22425 | 0,117 | 23114 | 0,474 |
| 21553 | 0,042 | 22242 | 0,355 | 22431 | 0,509 | 23115 | 0,253 |
| 21554 | -0,039 | 22243 | 0,34 | 22432 | 0,453 | 23121 | 0,66 |
| 21555 | -0,123 | 22244 | 0,18 | 22433 | 0,438 | 23122 | 0,603 |
| 22111 | 0,778 | 22245 | 0,014 | 22434 | 0,269 | 23123 | 0,589 |
| 22112 | 0,72 | 22251 | 0,092 | 22435 | 0,093 | 23124 | 0,376 |
| 22113 | 0,705 | 22252 | 0,035 | 22441 | 0,332 | 23125 | 0,155 |
| 22114 | 0,492 | 22253 | 0,021 | 22442 | 0,276 | 23131 | 0,635 |
| 22115 | 0,271 | 22254 | -0,06 | 22443 | 0,261 | 23132 | 0,579 |
| 22121 | 0,678 | 22255 | -0,144 | 22444 | 0,127 | 23133 | 0,564 |
| 22122 | 0,621 | 22311 | 0,74 | 22445 | -0,013 | 23134 | 0,351 |
| 22123 | 0,606 | 22312 | 0,683 | 22451 | 0,066 | 23135 | 0,13 |
| 22124 | 0,393 | 22313 | 0,669 | 22452 | 0,009 | 23141 | 0,423 |
| 22125 | 0,172 | 22314 | 0,456 | 22453 | -0,005 | 23142 | 0,366 |
| 22131 | 0,653 | 22315 | 0,235 | 22454 | -0,086 | 23143 | 0,352 |

96

| | | | | | Statistical | Analysis Plar | 1 030238/2FLZ3 |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 23144 | 0,192 | 23333 | 0,528 | 23522 | 0,24 | 24155 | -0,16 |
| 23145 | 0,025 | 23334 | 0,315 | 23523 | 0,226 | 24211 | 0,637 |
| 23151 | 0,103 | 23335 | 0,094 | 23524 | 0,145 | 24212 | 0,581 |
| 23152 | 0,047 | 23341 | 0,387 | 23525 | 0,061 | 24213 | 0,566 |
| 23153 | 0,032 | 23342 | 0,33 | 23531 | 0,272 | 24214 | 0,385 |
| 23154 | -0,049 | 23343 | 0,316 | 23532 | 0,216 | 24215 | 0,198 |
| 23155 | -0,133 | 23344 | 0,156 | 23533 | 0,201 | 24221 | 0,539 |
| 23211 | 0,729 | 23345 | -0,011 | 23534 | 0,12 | 24222 | 0,482 |
| 23212 | 0,673 | 23351 | 0,067 | 23535 | 0,036 | 24223 | 0,468 |
| 23212 | 0,658 | 23352 | 0,007 | 23541 | 0,167 | 24224 | 0,287 |
| 23213 | 0,445 | 23353 | -0,004 | 23542 | 0,111 | 24225 | 0,099 |
| 23214 | 0,224 | 23354 | -0,004 | 23543 | 0,096 | 24223 | 0,514 |
| | | | , and the second | | * | | ŕ |
| 23221 | 0,631 | 23355 | -0,169 | 23544 | 0,015 | 24232 | 0,458 |
| 23222 | 0,575 | 23411 | 0,615 | 23545 | -0,069 | 24233 | 0,443 |
| 23223 | 0,56 | 23412 | 0,559 | 23551 | 0,009 | 24234 | 0,262 |
| 23224 | 0,347 | 23413 | 0,544 | 23552 | -0,047 | 24235 | 0,075 |
| 23225 | 0,126 | 23414 | 0,374 | 23553 | -0,062 | 24241 | 0,328 |
| 23231 | 0,606 | 23415 | 0,198 | 23554 | -0,143 | 24242 | 0,272 |
| 23232 | 0,55 | 23421 | 0,516 | 23555 | -0,227 | 24243 | 0,257 |
| 23233 | 0,535 | 23422 | 0,46 | 24111 | 0,666 | 24244 | 0,116 |
| 23234 | 0,322 | 23423 | 0,445 | 24112 | 0,61 | 24245 | -0,03 |
| 23235 | 0,101 | 23424 | 0,276 | 24113 | 0,595 | 24251 | 0,048 |
| 23241 | 0,394 | 23425 | 0,1 | 24114 | 0,414 | 24252 | -0,009 |
| 23242 | 0,338 | 23431 | 0,492 | 24115 | 0,227 | 24253 | -0,023 |
| 23243 | 0,323 | 23432 | 0,436 | 24121 | 0,568 | 24254 | -0,104 |
| 23244 | 0,163 | 23433 | 0,421 | 24122 | 0,511 | 24255 | -0,188 |
| 23245 | -0,004 | 23434 | 0,251 | 24123 | 0,497 | 24311 | 0,63 |
| 23251 | 0,074 | 23435 | 0,075 | 24124 | 0,316 | 24312 | 0,574 |
| 23252 | 0,018 | 23441 | 0,315 | 24125 | 0,128 | 24313 | 0,559 |
| 23253 | 0,003 | 23442 | 0,258 | 24131 | 0,543 | 24314 | 0,378 |
| 23254 | -0,078 | 23443 | 0,244 | 24132 | 0,487 | 24315 | 0,191 |
| 23255 | -0,162 | 23444 | 0,109 | 24133 | 0,472 | 24321 | 0,532 |
| 23311 | 0,722 | 23445 | -0,03 | 24134 | 0,291 | 24322 | 0,475 |
| 23312 | 0,666 | 23451 | 0,048 | 24135 | 0,104 | 24323 | 0,461 |
| 23313 | 0,651 | 23452 | -0,008 | 24141 | 0,357 | 24324 | 0,28 |
| 23314 | 0,438 | 23453 | -0,023 | 24142 | 0,3 | 24325 | 0,092 |
| 23315 | 0,217 | 23454 | -0,104 | 24143 | 0,286 | 24331 | 0,507 |
| 23321 | 0,624 | 23455 | -0,188 | 24144 | 0,145 | 24332 | 0,451 |
| 23322 | 0,567 | 23511 | 0,395 | 24145 | -0,002 | 24333 | 0,436 |
| 23323 | 0,553 | 23512 | 0,339 | 24151 | 0,077 | 24334 | 0,255 |
| 23324 | 0,34 | 23513 | 0,324 | 24152 | 0,02 | 24335 | 0,068 |
| 23325 | 0,119 | 23514 | 0,243 | 24153 | 0,006 | 24341 | 0,321 |
| 23331 | 0,599 | 23515 | 0,159 | 24154 | -0,076 | 24342 | 0,264 |
| 23332 | 0,543 | 23521 | 0,297 | 24155 | -0,16 | 24343 | 0,25 |
| | , | | , | | ŕ | | • |

97

| - | | | | | Statistical | Allary Sis 1 lai | 1 030230 / 21 LZ |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 24344 | 0,109 | 24533 | 0,175 | 25222 | 0,196 | 25411 | 0,324 |
| 24345 | -0,038 | 24534 | 0,094 | 25223 | 0,181 | 25412 | 0,268 |
| 24351 | 0,041 | 24535 | 0,01 | 25224 | 0,1 | 25413 | 0,253 |
| 24352 | -0,016 | 24541 | 0,14 | 25225 | 0,016 | 25414 | 0,172 |
| 24353 | -0,031 | 24542 | 0,084 | 25231 | 0,227 | 25415 | 0,088 |
| 24354 | -0,112 | 24543 | 0,069 | 25232 | 0,171 | 25421 | 0,226 |
| 24355 | -0,196 | 24544 | -0,012 | 25233 | 0,156 | 25422 | 0,169 |
| 24411 | 0,544 | 24545 | -0,096 | 25234 | 0,075 | 25423 | 0,155 |
| 24412 | 0,488 | 24551 | -0,018 | 25235 | -0,009 | 25424 | 0,074 |
| 24413 | 0,473 | 24552 | -0,074 | 25241 | 0,122 | 25425 | -0,01 |
| 24414 | 0,325 | 24553 | -0,089 | 25242 | 0,066 | 25431 | 0,201 |
| 24415 | 0,323 | 24554 | -0,089 | 25242 | 0,051 | 25432 | 0,145 |
| 24421 | 0,172 | 24555 | -0,254 | 25244 | -0,03 | 25433 | 0,143 |
| 24421 | , and the second | | | | · · | 25434 | 0,049 |
| 24422 | 0,389 | 25111<br>25112 | 0,379 | 25245<br>25251 | -0,114 | 25435 | -0,035 |
| 24423 | 0,375<br>0,227 | | 0,323 | | -0,036<br>-0,092 | 25441 | 0,096 |
| | , and the second | 25113 | 0,308 | 25252 | | | |
| 24425 | 0,073 | 25114 | 0,227 | 25253 | -0,107 | 25442 | 0,04 |
| 24431 | 0,421 | 25115 | 0,143 | 25254 | -0,188 | 25443 | 0,025 |
| 24432 | 0,365 | 25121 | 0,281 | 25255 | -0,272 | 25444 | -0,056 |
| 24433 | 0,35 | 25122 | 0,224 | 25311 | 0,343 | 25445 | -0,14 |
| 24434 | 0,202 | 25123 | 0,21 | 25312 | 0,287 | 25451 | -0,062 |
| 24435 | 0,049 | 25124 | 0,129 | 25313 | 0,272 | 25452 | -0,118 |
| 24441 | 0,262 | 25125 | 0,045 | 25314 | 0,191 | 25453 | -0,133 |
| 24442 | 0,205 | 25131 | 0,256 | 25315 | 0,107 | 25454 | -0,214 |
| 24443 | 0,191 | 25132 | 0,2 | 25321 | 0,245 | 25455 | -0,298 |
| 24444 | 0,069 | 25133 | 0,185 | 25322 | 0,188 | 25511 | 0,285 |
| 24445 | -0,057 | 25134 | 0,104 | 25323 | 0,174 | 25512 | 0,229 |
| 24451 | 0,022 | 25135 | 0,02 | 25324 | 0,093 | 25513 | 0,214 |
| 24452 | -0,035 | 25141 | 0,151 | 25325 | 0,009 | 25514 | 0,133 |
| 24453 | -0,05 | 25142 | 0,095 | 25331 | 0,22 | 25515 | 0,049 |
| 24454 | -0,131 | 25143 | 0,08 | 25332 | 0,164 | 25521 | 0,187 |
| 24455 | -0,215 | 25144 | -0,001 | 25333 | 0,149 | 25522 | 0,13 |
| 24511 | 0,369 | 25145 | -0,085 | 25334 | 0,068 | 25523 | 0,116 |
| 24512 | 0,312 | 25151 | -0,007 | 25335 | -0,016 | 25524 | 0,035 |
| 24513 | 0,298 | 25152 | -0,063 | 25341 | 0,115 | 25525 | -0,049 |
| 24514 | 0,217 | 25153 | -0,078 | 25342 | 0,059 | 25531 | 0,162 |
| 24515 | 0,133 | 25154 | -0,159 | 25343 | 0,044 | 25532 | 0,106 |
| 24521 | 0,27 | 25155 | -0,243 | 25344 | -0,037 | 25533 | 0,091 |
| 24522 | 0,214 | 25211 | 0,35 | 25345 | -0,121 | 25534 | 0,01 |
| 24523 | 0,199 | 25212 | 0,294 | 25351 | -0,043 | 25535 | -0,074 |
| 24524 | 0,118 | 25213 | 0,279 | 25352 | -0,099 | 25541 | 0,057 |
| 24525 | 0,034 | 25214 | 0,198 | 25353 | -0,114 | 25542 | 0,001 |
| 24531 | 0,246 | 25215 | 0,114 | 25354 | -0,195 | 25543 | -0,014 |
| 24532 | 0,189 | 25221 | 0,252 | 25355 | -0,279 | 25544 | -0,095 |

| - | | | | | Statistical | Allary Sis 1 lai | 1 030230 / 21 LZ |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 25545 | -0,179 | 31234 | 0,414 | 31423 | 0,537 | 32112 | 0,707 |
| 25551 | -0,101 | 31235 | 0,193 | 31424 | 0,368 | 32113 | 0,692 |
| 25552 | -0,157 | 31241 | 0,486 | 31425 | 0,191 | 32114 | 0,479 |
| 25553 | -0,172 | 31242 | 0,429 | 31431 | 0,584 | 32115 | 0,258 |
| 25554 | -0,253 | 31243 | 0,415 | 31432 | 0,527 | 32121 | 0,665 |
| 25555 | -0,337 | 31244 | 0,254 | 31433 | 0,513 | 32122 | 0,609 |
| 31111 | 0,85 | 31245 | 0,088 | 31434 | 0,343 | 32123 | 0,594 |
| 31112 | 0,794 | 31251 | 0,166 | 31435 | 0,167 | 32124 | 0,381 |
| 31113 | 0,779 | 31252 | 0,11 | 31441 | 0,406 | 32125 | 0,16 |
| 31114 | 0,566 | 31253 | 0,095 | 31442 | 0,35 | 32131 | 0,64 |
| 31115 | 0,345 | 31254 | 0,014 | 31443 | 0,335 | 32132 | 0,584 |
| 31121 | 0,752 | 31255 | -0,07 | 31444 | 0,201 | 32133 | 0,569 |
| 31121 | 0,695 | 31311 | 0,814 | 31445 | 0,062 | 32134 | 0,356 |
| 31122 | 0,681 | 31312 | 0,758 | 31451 | 0,14 | 32135 | 0,135 |
| 31123 | 0,468 | 31313 | 0,743 | 31452 | 0,084 | 32141 | 0,428 |
| 31124 | 0,247 | 31313 | 0,743 | 31453 | 0,069 | 32141 | 0,372 |
| 31123 | 0,727 | 31314 | 0,309 | 31454 | -0,012 | 32142 | 0,357 |
| | 0,727 | | , and the second | 31455 | -0,012 | 32143 | 0,197 |
| 31132 | , and the second | 31321 | 0,716 | | | | ŕ |
| 31133 | 0,656 | 31322 | 0,659 | 31511 | 0,487 | 32145 | 0,03 |
| 31134 | 0,443 | 31323 | 0,645 | 31512 | 0,431 | 32151 | 0,108 |
| 31135 | 0,222 | 31324 | 0,432 | 31513 | 0,416 | 32152 | 0,052 |
| 31141 | 0,515 | 31325 | 0,211 | 31514 | 0,335 | 32153 | 0,037 |
| 31142 | 0,458 | 31331 | 0,691 | 31515 | 0,251 | 32154 | -0,044 |
| 31143 | 0,444 | 31332 | 0,635 | 31521 | 0,389 | 32155 | -0,128 |
| 31144 | 0,283 | 31333 | 0,62 | 31522 | 0,332 | 32211 | 0,735 |
| 31145 | 0,117 | 31334 | 0,407 | 31523 | 0,318 | 32212 | 0,678 |
| 31151 | 0,195 | 31335 | 0,186 | 31524 | 0,237 | 32213 | 0,664 |
| 31152 | 0,139 | 31341 | 0,479 | 31525 | 0,153 | 32214 | 0,451 |
| 31153 | 0,124 | 31342 | 0,422 | 31531 | 0,364 | 32215 | 0,23 |
| 31154 | 0,043 | 31343 | 0,408 | 31532 | 0,308 | 32221 | 0,636 |
| 31155 | -0,041 | 31344 | 0,247 | 31533 | 0,293 | 32222 | 0,58 |
| 31211 | 0,821 | 31345 | 0,081 | 31534 | 0,212 | 32223 | 0,565 |
| 31212 | 0,765 | 31351 | 0,159 | 31535 | 0,128 | 32224 | 0,352 |
| 31213 | 0,75 | 31352 | 0,103 | 31541 | 0,259 | 32225 | 0,131 |
| 31214 | 0,537 | 31353 | 0,088 | 31542 | 0,203 | 32231 | 0,612 |
| 31215 | 0,316 | 31354 | 0,007 | 31543 | 0,188 | 32232 | 0,555 |
| 31221 | 0,723 | 31355 | -0,077 | 31544 | 0,107 | 32233 | 0,541 |
| 31222 | 0,666 | 31411 | 0,707 | 31545 | 0,023 | 32234 | 0,328 |
| 31223 | 0,652 | 31412 | 0,65 | 31551 | 0,101 | 32235 | 0,107 |
| 31224 | 0,439 | 31413 | 0,636 | 31552 | 0,045 | 32241 | 0,399 |
| 31225 | 0,218 | 31414 | 0,466 | 31553 | 0,03 | 32242 | 0,343 |
| 31231 | 0,698 | 31415 | 0,29 | 31554 | -0,051 | 32243 | 0,328 |
| 31232 | 0,642 | 31421 | 0,608 | 31555 | -0,135 | 32244 | 0,168 |
| 31233 | 0,627 | 31422 | 0,552 | 32111 | 0,763 | 32245 | 0,002 |

| | | | | | Statistical | Allaly SIS I lai | 1 030230721 1123 |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 32251 | 0,08 | 32435 | 0,08 | 33124 | 0,364 | 33313 | 0,639 |
| 32252 | 0,023 | 32441 | 0,32 | 33125 | 0,143 | 33314 | 0,426 |
| 32253 | 0,009 | 32442 | 0,263 | 33131 | 0,623 | 33315 | 0,205 |
| 32254 | -0,072 | 32443 | 0,249 | 33132 | 0,567 | 33321 | 0,612 |
| 32255 | -0,157 | 32444 | 0,115 | 33133 | 0,552 | 33322 | 0,555 |
| 32311 | 0,727 | 32445 | -0,025 | 33134 | 0,339 | 33323 | 0,541 |
| 32312 | 0,671 | 32451 | 0,053 | 33135 | 0,118 | 33324 | 0,328 |
| 32313 | 0,656 | 32452 | -0,003 | 33141 | 0,411 | 33325 | 0,107 |
| 32314 | 0,443 | 32453 | -0,018 | 33142 | 0,354 | 33331 | 0,587 |
| 32315 | 0,222 | 32454 | -0,099 | 33143 | 0,34 | 33331 | 0,531 |
| 32313 | 0,629 | 32455 | -0,183 | 33144 | 0,179 | 33333 | 0,516 |
| 32321 | 0,573 | 32511 | 0,4 | 33145 | 0,179 | 33333 | 0,303 |
| 32322 | 0,558 | 32512 | 0,344 | 33143 | 0,013 | 33335 | 0,082 |
| | | | | | | | 0,375 |
| 32324<br>32325 | 0,345 | 32513<br>32514 | 0,329 | 33152 | 0,035 | 33341 | 0,373 |
| 32323 | 0,124<br>0,604 | | 0,248 | 33153 | 0,02<br>-0,061 | 33342 | 0,318 |
| | | 32515 | 0,164 | 33154 | | 33343 | |
| 32332 | 0,548 | 32521 | 0,302 | 33155 | -0,145 | 33344 | 0,143 |
| 32333 | 0,533 | 32522 | 0,246 | 33211 | 0,717 | 33345 | -0,023 |
| 32334 | 0,32 | 32523 | 0,231 | 33212 | 0,661 | 33351 | 0,055 |
| 32335 | 0,099 | 32524 | 0,15 | 33213 | 0,646 | 33352 | -0,001 |
| 32341 | 0,392 | 32525 | 0,066 | 33214 | 0,433 | 33353 | -0,016 |
| 32342 | 0,336 | 32531 | 0,277 | 33215 | 0,212 | 33354 | -0,097 |
| 32343 | 0,321 | 32532 | 0,221 | 33221 | 0,619 | 33355 | -0,181 |
| 32344 | 0,161 | 32533 | 0,206 | 33222 | 0,562 | 33411 | 0,603 |
| 32345 | -0,006 | 32534 | 0,125 | 33223 | 0,548 | 33412 | 0,546 |
| 32351 | 0,072 | 32535 | 0,041 | 33224 | 0,335 | 33413 | 0,532 |
| 32352 | 0,016 | 32541 | 0,172 | 33225 | 0,114 | 33414 | 0,362 |
| 32353 | 0,001 | 32542 | 0,116 | 33231 | 0,594 | 33415 | 0,186 |
| 32354 | -0,08 | 32543 | 0,101 | 33232 | 0,538 | 33421 | 0,504 |
| 32355 | -0,164 | 32544 | 0,02 | 33233 | 0,523 | 33422 | 0,448 |
| 32411 | 0,62 | 32545 | -0,064 | 33234 | 0,31 | 33423 | 0,433 |
| 32412 | 0,564 | 32551 | 0,014 | 33235 | 0,089 | 33424 | 0,264 |
| 32413 | 0,549 | 32552 | -0,042 | 33241 | 0,382 | 33425 | 0,087 |
| 32414 | 0,379 | 32553 | -0,057 | 33242 | 0,325 | 33431 | 0,48 |
| 32415 | 0,203 | 32554 | -0,138 | 33243 | 0,311 | 33432 | 0,423 |
| 32421 | 0,522 | 32555 | -0,222 | 33244 | 0,15 | 33433 | 0,409 |
| 32422 | 0,465 | 33111 | 0,746 | 33245 | -0,016 | 33434 | 0,239 |
| 32423 | 0,451 | 33112 | 0,69 | 33251 | 0,062 | 33435 | 0,063 |
| 32424 | 0,281 | 33113 | 0,675 | 33252 | 0,006 | 33441 | 0,302 |
| 32425 | 0,105 | 33114 | 0,462 | 33253 | -0,009 | 33442 | 0,246 |
| 32431 | 0,497 | 33115 | 0,241 | 33254 | -0,09 | 33443 | 0,231 |
| 32432 | 0,441 | 33121 | 0,648 | 33255 | -0,174 | 33444 | 0,097 |
| 32433 | 0,426 | 33122 | 0,591 | 33311 | 0,71 | 33445 | -0,042 |
| 32434 | 0,256 | 33123 | 0,577 | 33312 | 0,654 | 33451 | 0,036 |

| | | | | | Statistical | Allary Sis T lai | 1 030230721 123 |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 33452 | -0,02 | 34141 | 0,345 | 34325 | 0,08 | 34514 | 0,204 |
| 33453 | -0,035 | 34142 | 0,288 | 34331 | 0,495 | 34515 | 0,12 |
| 33454 | -0,116 | 34143 | 0,274 | 34332 | 0,439 | 34521 | 0,258 |
| 33455 | -0,2 | 34144 | 0,133 | 34333 | 0,424 | 34522 | 0,201 |
| 33511 | 0,383 | 34145 | -0,014 | 34334 | 0,243 | 34523 | 0,187 |
| 33512 | 0,327 | 34151 | 0,064 | 34335 | 0,055 | 34524 | 0,106 |
| 33513 | 0,312 | 34152 | 0,008 | 34341 | 0,309 | 34525 | 0,022 |
| 33514 | 0,231 | 34153 | -0,007 | 34342 | 0,252 | 34531 | 0,233 |
| 33515 | 0,147 | 34154 | -0,088 | 34343 | 0,238 | 34532 | 0,177 |
| 33521 | 0,285 | 34155 | -0,172 | 34344 | 0,097 | 34533 | 0,162 |
| 33522 | 0,228 | 34211 | 0,625 | 34345 | -0,05 | 34534 | 0,081 |
| 33523 | 0,214 | 34212 | 0,569 | 34351 | 0,028 | 34535 | -0,003 |
| 33524 | 0,133 | 34213 | 0,554 | 34352 | -0,028 | 34541 | 0,128 |
| 33525 | 0,049 | 34214 | 0,373 | 34353 | -0,043 | 34542 | 0,072 |
| 33531 | 0,26 | 34215 | 0,185 | 34354 | -0,124 | 34543 | 0,057 |
| 33532 | 0,204 | 34221 | 0,527 | 34355 | -0,208 | 34544 | -0,024 |
| 33533 | 0,189 | 34222 | 0,47 | 34411 | 0,532 | 34545 | -0,108 |
| 33534 | 0,108 | 34223 | 0,456 | 34412 | 0,476 | 34551 | -0,03 |
| 33535 | 0,024 | 34224 | 0,275 | 34413 | 0,461 | 34552 | -0,086 |
| 33541 | 0,155 | 34225 | 0,087 | 34414 | 0,313 | 34553 | -0,101 |
| 33542 | 0,099 | 34231 | 0,502 | 34415 | 0,159 | 34554 | -0,182 |
| 33543 | 0,084 | 34232 | 0,446 | 34421 | 0,433 | 34555 | -0,266 |
| 33544 | 0,003 | 34233 | 0,431 | 34422 | 0,377 | 35111 | 0,367 |
| 33545 | -0,081 | 34234 | 0,25 | 34423 | 0,362 | 35112 | 0,311 |
| 33551 | -0,003 | 34235 | 0,062 | 34424 | 0,214 | 35113 | 0,296 |
| 33552 | -0,059 | 34241 | 0,316 | 34425 | 0,061 | 35114 | 0,215 |
| 33553 | -0,074 | 34242 | 0,259 | 34431 | 0,409 | 35115 | 0,131 |
| 33554 | -0,155 | 34243 | 0,245 | 34432 | 0,353 | 35121 | 0,269 |
| 33555 | -0,239 | 34244 | 0,104 | 34433 | 0,338 | 35122 | 0,212 |
| 34111 | 0,654 | 34245 | -0,043 | 34434 | 0,19 | 35123 | 0,198 |
| 34112 | 0,598 | 34251 | 0,035 | 34435 | 0,036 | 35124 | 0,117 |
| 34113 | 0,583 | 34252 | -0,021 | 34441 | 0,249 | 35125 | 0,033 |
| 34114 | 0,402 | 34253 | -0,036 | 34442 | 0,193 | 35131 | 0,244 |
| 34115 | 0,214 | 34254 | -0,117 | 34443 | 0,178 | 35132 | 0,188 |
| 34121 | 0,555 | 34255 | -0,201 | 34444 | 0,057 | 35133 | 0,173 |
| 34122 | 0,499 | 34311 | 0,618 | 34445 | -0,069 | 35134 | 0,092 |
| 34123 | 0,484 | 34312 | 0,562 | 34451 | 0,009 | 35135 | 0,008 |
| 34124 | 0,304 | 34313 | 0,547 | 34452 | -0,047 | 35141 | 0,139 |
| 34125 | 0,116 | 34314 | 0,366 | 34453 | -0,062 | 35142 | 0,083 |
| 34131 | 0,531 | 34315 | 0,178 | 34454 | -0,143 | 35143 | 0,068 |
| 34132 | 0,475 | 34321 | 0,519 | 34455 | -0,227 | 35144 | -0,013 |
| 34133 | 0,46 | 34322 | 0,463 | 34511 | 0,356 | 35145 | -0,097 |
| 34134 | 0,279 | 34323 | 0,448 | 34512 | 0,330 | 35143 | -0,019 |
| 34135 | 0,091 | 34324 | 0,268 | 34513 | 0,285 | 35151 | -0,075 |
| 54155 | 0,071 | 5-152-1 | 0,200 | 57515 | 0,203 | 33132 | 0,075 |

101

| | | | | | Statistical | Allary Sis T lai | 1 030230721 123 |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 35153 | -0,09 | 35342 | 0,047 | 35531 | 0,15 | 41215 | 0,299 |
| 35154 | -0,171 | 35343 | 0,032 | 35532 | 0,094 | 41221 | 0,686 |
| 35155 | -0,255 | 35344 | -0,049 | 35533 | 0,079 | 41222 | 0,629 |
| 35211 | 0,338 | 35345 | -0,133 | 35534 | -0,002 | 41223 | 0,615 |
| 35212 | 0,282 | 35351 | -0,055 | 35535 | -0,086 | 41224 | 0,411 |
| 35213 | 0,267 | 35352 | -0,111 | 35541 | 0,045 | 41225 | 0,2 |
| 35214 | 0,186 | 35353 | -0,126 | 35542 | -0,011 | 41231 | 0,661 |
| 35215 | 0,102 | 35354 | -0,207 | 35543 | -0,026 | 41232 | 0,605 |
| 35221 | 0,24 | 35355 | -0,291 | 35544 | -0,107 | 41233 | 0,59 |
| 35222 | 0,183 | 35411 | 0,312 | 35545 | -0,191 | 41234 | 0,387 |
| 35223 | 0,169 | 35412 | 0,256 | 35551 | -0,113 | 41235 | 0,176 |
| 35224 | 0,088 | 35413 | 0,241 | 35552 | -0,169 | 41241 | 0,456 |
| 35225 | 0,004 | 35414 | 0,16 | 35553 | -0,184 | 41242 | 0,4 |
| 35231 | 0,215 | 35415 | 0,076 | 35554 | -0,265 | 41243 | 0,385 |
| 35232 | 0,159 | 35421 | 0,213 | 35555 | -0,349 | 41244 | 0,231 |
| 35233 | 0,144 | 35422 | 0,157 | 41111 | 0,813 | 41245 | 0,07 |
| 35234 | 0,063 | 35423 | 0,137 | 41112 | 0,757 | 41251 | 0,149 |
| 35235 | -0,021 | 35424 | 0,061 | 41113 | 0,742 | 41252 | 0,092 |
| 35241 | 0,11 | 35425 | -0,023 | 41114 | 0,539 | 41253 | 0,072 |
| 35241 | 0,054 | 35431 | 0,189 | 41115 | 0,339 | 41254 | -0,004 |
| 35242 | 0,034 | | 0,133 | | | | -0,004 |
| | | 35432<br>35433 | | 41121 | 0,714 | 41255 | • |
| 35244 | -0,042 | 35433 | 0,118 | 41122 | 0,658 | 41311 | 0,777 |
| 35245 | -0,126 | 35434 | 0,037 | 41123 | 0,643 | 41312 | 0,721 |
| 35251 | -0,048 | 35435 | -0,047 | 41124 | 0,44 | 41313 | 0,706 |
| 35252 | -0,104 | 35441 | 0,084 | 41125 | 0,229 | 41314 | 0,503 |
| 35253 | -0,119 | 35442 | 0,028 | 41131 | 0,69 | 41315 | 0,291 |
| 35254 | -0,2 | 35443 | 0,013 | 41132 | 0,634 | 41321 | 0,678 |
| 35255 | -0,284 | 35444 | -0,068 | 41133 | 0,619 | 41322 | 0,622 |
| 35311 | 0,331 | 35445 | -0,152 | 41134 | 0,416 | 41323 | 0,607 |
| 35312 | 0,275 | 35451 | -0,074 | 41135 | 0,204 | 41324 | 0,404 |
| 35313 | 0,26 | 35452 | -0,13 | 41141 | 0,485 | 41325 | 0,193 |
| 35314 | 0,179 | 35453 | -0,145 | 41142 | 0,429 | 41331 | 0,654 |
| 35315 | 0,095 | 35454 | -0,226 | 41143 | 0,414 | 41332 | 0,598 |
| 35321 | 0,233 | 35455 | -0,31 | 41144 | 0,26 | 41333 | 0,583 |
| 35322 | 0,176 | 35511 | 0,273 | 41145 | 0,099 | 41334 | 0,38 |
| 35323 | 0,162 | 35512 | 0,217 | 41151 | 0,177 | 41335 | 0,168 |
| 35324 | 0,081 | 35513 | 0,202 | 41152 | 0,121 | 41341 | 0,449 |
| 35325 | -0,004 | 35514 | 0,121 | 41153 | 0,106 | 41342 | 0,393 |
| 35331 | 0,208 | 35515 | 0,037 | 41154 | 0,025 | 41343 | 0,378 |
| 35332 | 0,152 | 35521 | 0,175 | 41155 | -0,059 | 41344 | 0,224 |
| 35333 | 0,137 | 35522 | 0,118 | 41211 | 0,784 | 41345 | 0,063 |
| 35334 | 0,056 | 35523 | 0,104 | 41212 | 0,728 | 41351 | 0,141 |
| 35335 | -0,028 | 35524 | 0,023 | 41213 | 0,713 | 41352 | 0,085 |
| 35341 | 0,103 | 35525 | -0,062 | 41214 | 0,51 | 41353 | 0,07 |

| | | | | | Statistical | Analysis Plai | 1 030238/2FLZ3 |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 41354 | -0,011 | 41543 | 0,17 | 42232 | 0,518 | 42421 | 0,491 |
| 41355 | -0,095 | 41544 | 0,089 | 42233 | 0,504 | 42422 | 0,434 |
| 41411 | 0,676 | 41545 | 0,005 | 42234 | 0,3 | 42423 | 0,42 |
| 41412 | 0,62 | 41551 | 0,083 | 42235 | 0,089 | 42424 | 0,257 |
| 41413 | 0,605 | 41552 | 0,027 | 42241 | 0,37 | 42425 | 0,087 |
| 41414 | 0,442 | 41553 | 0,012 | 42242 | 0,313 | 42431 | 0,466 |
| 41415 | 0,272 | 41554 | -0,069 | 42243 | 0,299 | 42432 | 0,41 |
| 41421 | 0,577 | 41555 | -0,153 | 42244 | 0,144 | 42433 | 0,395 |
| 41422 | 0,521 | 42111 | 0,726 | 42245 | -0,016 | 42434 | 0,232 |
| 41423 | 0,506 | 42111 | 0,720 | 42251 | 0,062 | 42435 | 0,063 |
| 41424 | 0,343 | 42113 | 0,655 | 42252 | 0,002 | 42441 | 0,294 |
| 41425 | 0,174 | 42113 | 0,452 | 42253 | -0,009 | 42442 | 0,238 |
| | | | | 42254 | -0,009 | | 0,238 |
| 41431 | 0,553 | 42115<br>42121 | 0,241 | | · · | 42443 | ŕ |
| 41432 | 0,497 | | 0,628 | 42255 | -0,174 | 42444 | 0,093 |
| 41433 | 0,482 | 42122 | 0,572 | 42311 | 0,69 | 42445 | -0,042 |
| 41434 | 0,319 | 42123 | 0,557 | 42312 | 0,634 | 42451 | 0,036 |
| 41435 | 0,149 | 42124 | 0,353 | 42313 | 0,619 | 42452 | -0,021 |
| 41441 | 0,381 | 42125 | 0,142 | 42314 | 0,416 | 42453 | -0,035 |
| 41442 | 0,325 | 42131 | 0,603 | 42315 | 0,205 | 42454 | -0,116 |
| 41443 | 0,31 | 42132 | 0,547 | 42321 | 0,592 | 42455 | -0,2 |
| 41444 | 0,18 | 42133 | 0,532 | 42322 | 0,536 | 42511 | 0,383 |
| 41445 | 0,044 | 42134 | 0,329 | 42323 | 0,521 | 42512 | 0,326 |
| 41451 | 0,122 | 42135 | 0,118 | 42324 | 0,317 | 42513 | 0,312 |
| 41452 | 0,066 | 42141 | 0,399 | 42325 | 0,106 | 42514 | 0,231 |
| 41453 | 0,051 | 42142 | 0,342 | 42331 | 0,567 | 42515 | 0,147 |
| 41454 | -0,03 | 42143 | 0,328 | 42332 | 0,511 | 42521 | 0,284 |
| 41455 | -0,114 | 42144 | 0,173 | 42333 | 0,496 | 42522 | 0,228 |
| 41511 | 0,469 | 42145 | 0,013 | 42334 | 0,293 | 42523 | 0,213 |
| 41512 | 0,413 | 42151 | 0,091 | 42335 | 0,082 | 42524 | 0,132 |
| 41513 | 0,398 | 42152 | 0,034 | 42341 | 0,363 | 42525 | 0,048 |
| 41514 | 0,317 | 42153 | 0,02 | 42342 | 0,306 | 42531 | 0,26 |
| 41515 | 0,233 | 42154 | -0,061 | 42343 | 0,292 | 42532 | 0,203 |
| 41521 | 0,371 | 42155 | -0,145 | 42344 | 0,137 | 42533 | 0,189 |
| 41522 | 0,315 | 42211 | 0,698 | 42345 | -0,023 | 42534 | 0,108 |
| 41523 | 0,3 | 42212 | 0,641 | 42351 | 0,055 | 42535 | 0,024 |
| 41524 | 0,219 | 42213 | 0,627 | 42352 | -0,002 | 42541 | 0,155 |
| 41525 | 0,135 | 42214 | 0,423 | 42353 | -0,016 | 42542 | 0,098 |
| 41531 | 0,346 | 42215 | 0,212 | 42354 | -0,097 | 42543 | 0,084 |
| 41532 | 0,29 | 42221 | 0,599 | 42355 | -0,181 | 42544 | 0,003 |
| 41533 | 0,275 | 42222 | 0,543 | 42411 | 0,589 | 42545 | -0,081 |
| 41534 | 0,194 | 42223 | 0,528 | 42412 | 0,533 | 42551 | -0,003 |
| 41535 | 0,11 | 42224 | 0,325 | 42413 | 0,518 | 42552 | -0,06 |
| 41541 | 0,241 | 42225 | 0,113 | 42414 | 0,355 | 42553 | -0,074 |
| 41542 | 0,185 | 42231 | 0,575 | 42415 | 0,186 | 42554 | -0,155 |
| | • | | • | | • | | |

| | | | | | Statistical | Allalysis I lai | 1 030230721 LL3 |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 42555 | -0,239 | 43244 | 0,127 | 43433 | 0,378 | 44122 | 0,467 |
| 43111 | 0,709 | 43245 | -0,034 | 43434 | 0,215 | 44123 | 0,452 |
| 43112 | 0,653 | 43251 | 0,045 | 43435 | 0,045 | 44124 | 0,278 |
| 43113 | 0,638 | 43252 | -0,012 | 43441 | 0,277 | 44125 | 0,098 |
| 43114 | 0,435 | 43253 | -0,027 | 43442 | 0,221 | 44131 | 0,499 |
| 43115 | 0,223 | 43254 | -0,108 | 43443 | 0,206 | 44132 | 0,442 |
| 43121 | 0,61 | 43255 | -0,192 | 43444 | 0,076 | 44133 | 0,428 |
| 43122 | 0,554 | 43311 | 0,673 | 43445 | -0,06 | 44134 | 0,254 |
| 43123 | 0,539 | 43312 | 0,617 | 43451 | 0,018 | 44135 | 0,074 |
| 43124 | 0,336 | 43313 | 0,602 | 43452 | -0,038 | 44141 | 0,318 |
| 43125 | 0,125 | 43314 | 0,399 | 43453 | -0,053 | 44142 | 0,262 |
| 43131 | 0,586 | 43315 | 0,187 | 43454 | -0,134 | 44143 | 0,247 |
| 43132 | 0,53 | 43321 | 0,574 | 43455 | -0,134 | 44144 | 0,11 |
| 43133 | 0,515 | 43322 | 0,518 | 43511 | 0,365 | 44145 | -0,032 |
| 43134 | 0,312 | 43323 | 0,503 | 43512 | 0,309 | 44151 | 0,047 |
| 43135 | 0,512 | 43324 | 0,303 | 43513 | 0,309 | 44152 | -0,01 |
| 43133 | 0,381 | 43325 | 0,089 | 43514 | 0,234 | 44153 | -0,01 |
| 43141 | 0,325 | 43323 | * | 43515 | | 44154 | -0,105 |
| | | | 0,55 | | 0,129 | | ŕ |
| 43143 | 0,31 | 43332 | 0,494 | 43521 | 0,267 | 44155 | -0,189 |
| 43144 | 0,156 | 43333 | 0,479 | 43522 | 0,211 | 44211 | 0,593 |
| 43145 | -0,005 | 43334 | 0,276 | 43523 | 0,196 | 44212 | 0,536 |
| 43151 | 0,073 | 43335 | 0,064 | 43524 | 0,115 | 44213 | 0,522 |
| 43152 | 0,017 | 43341 | 0,345 | 43525 | 0,031 | 44214 | 0,348 |
| 43153 | 0,002 | 43342 | 0,289 | 43531 | 0,242 | 44215 | 0,168 |
| 43154 | -0,079 | 43343 | 0,274 | 43532 | 0,186 | 44221 | 0,494 |
| 43155 | -0,163 | 43344 | 0,12 | 43533 | 0,171 | 44222 | 0,438 |
| 43211 | 0,68 | 43345 | -0,041 | 43534 | 0,09 | 44223 | 0,423 |
| 43212 | 0,624 | 43351 | 0,037 | 43535 | 0,006 | 44224 | 0,249 |
| 43213 | 0,609 | 43352 | -0,019 | 43541 | 0,137 | 44225 | 0,069 |
| 43214 | 0,406 | 43353 | -0,034 | 43542 | 0,081 | 44231 | 0,47 |
| 43215 | 0,195 | 43354 | -0,115 | 43543 | 0,066 | 44232 | 0,413 |
| 43221 | 0,582 | 43355 | -0,199 | 43544 | -0,015 | 44233 | 0,399 |
| 43222 | 0,525 | 43411 | 0,572 | 43545 | -0,099 | 44234 | 0,225 |
| 43223 | 0,511 | 43412 | 0,516 | 43551 | -0,021 | 44235 | 0,045 |
| 43224 | 0,307 | 43413 | 0,501 | 43552 | -0,077 | 44241 | 0,289 |
| 43225 | 0,096 | 43414 | 0,338 | 43553 | -0,092 | 44242 | 0,233 |
| 43231 | 0,557 | 43415 | 0,168 | 43554 | -0,173 | 44243 | 0,218 |
| 43232 | 0,501 | 43421 | 0,473 | 43555 | -0,257 | 44244 | 0,082 |
| 43233 | 0,486 | 43422 | 0,417 | 44111 | 0,622 | 44245 | -0,06 |
| 43234 | 0,283 | 43423 | 0,402 | 44112 | 0,565 | 44251 | 0,018 |
| 43235 | 0,072 | 43424 | 0,239 | 44113 | 0,551 | 44252 | -0,039 |
| 43241 | 0,352 | 43425 | 0,07 | 44114 | 0,377 | 44253 | -0,053 |
| 43242 | 0,296 | 43431 | 0,449 | 44115 | 0,197 | 44254 | -0,134 |
| 43243 | 0,281 | 43432 | 0,393 | 44121 | 0,523 | 44255 | -0,218 |

104

| - | | | | | | <i>j</i> | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 44311 | 0,586 | 44445 | -0,087 | 45134 | 0,074 | 45323 | 0,144 |
| 44312 | 0,529 | 44451 | -0,009 | 45135 | -0,01 | 45324 | 0,063 |
| 44313 | 0,515 | 44452 | -0,065 | 45141 | 0,121 | 45325 | -0,021 |
| 44314 | 0,341 | 44453 | -0,08 | 45142 | 0,065 | 45331 | 0,19 |
| 44315 | 0,161 | 44454 | -0,16 | 45143 | 0,05 | 45332 | 0,134 |
| 44321 | 0,487 | 44455 | -0,245 | 45144 | -0,031 | 45333 | 0,119 |
| 44322 | 0,431 | 44511 | 0,339 | 45145 | -0,115 | 45334 | 0,038 |
| 44323 | 0,416 | 44512 | 0,282 | 45151 | -0,037 | 45335 | -0,046 |
| | | | | | | | • |
| 44324 | 0,242 | 44513 | 0,268 | 45152 | -0,093 | 45341 | 0,085 |
| 44325 | 0,062 | 44514 | 0,187 | 45153 | -0,108 | 45342 | 0,029 |
| 44331 | 0,463 | 44515 | 0,103 | 45154 | -0,189 | 45343 | 0,014 |
| 44332 | 0,406 | 44521 | 0,24 | 45155 | -0,273 | 45344 | -0,067 |
| 44333 | 0,392 | 44522 | 0,184 | 45211 | 0,321 | 45345 | -0,151 |
| 44334 | 0,218 | 44523 | 0,169 | 45212 | 0,264 | 45351 | -0,073 |
| 44335 | 0,038 | 44524 | 0,088 | 45213 | 0,25 | 45352 | -0,129 |
| 44341 | 0,282 | 44525 | 0,004 | 45214 | 0,169 | 45353 | -0,144 |
| 44342 | 0,226 | 44531 | 0,216 | 45215 | 0,085 | 45354 | -0,225 |
| 44343 | 0,211 | 44532 | 0,159 | 45221 | 0,222 | 45355 | -0,309 |
| 44344 | 0,074 | 44533 | 0,145 | 45222 | 0,166 | 45411 | 0,294 |
| 44345 | -0,068 | 44534 | 0,064 | 45223 | 0,151 | 45412 | 0,238 |
| 44351 | 0,011 | 44535 | -0,02 | 45224 | 0,07 | 45413 | 0,223 |
| 44352 | -0,046 | 44541 | 0,111 | 45225 | -0,014 | 45414 | 0,142 |
| 44353 | -0,06 | 44542 | 0,054 | 45231 | 0,198 | 45415 | 0,058 |
| 44354 | -0,141 | 44543 | 0,04 | 45232 | 0,141 | 45421 | 0,196 |
| 44355 | -0,225 | 44544 | -0,041 | 45233 | 0,127 | 45422 | 0,139 |
| 44411 | 0,504 | 44545 | -0,126 | 45234 | 0,046 | 45423 | 0,125 |
| 44412 | 0,448 | 44551 | -0,047 | 45235 | -0,039 | 45424 | 0,044 |
| 44413 | 0,433 | 44552 | -0,104 | 45241 | 0,092 | 45425 | -0,04 |
| 44414 | 0,29 | 44553 | -0,118 | 45242 | 0,036 | 45431 | 0,171 |
| 44415 | 0,142 | 44554 | -0,199 | 45243 | 0,021 | 45432 | 0,115 |
| 44421 | 0,406 | 44555 | -0,283 | 45244 | -0,06 | 45433 | 0,1 |
| 44422 | 0,35 | 45111 | 0,349 | 45245 | -0,144 | 45434 | 0,019 |
| 44423 | 0,335 | | 0,293 | 45251 | -0,066 | 45435 | -0,065 |
| | | 45112 | | | | | |
| 44424 | 0,192 | 45113 | 0,278 | 45252 | -0,122 | 45441 | 0,066 |
| 44425 | 0,043 | 45114 | 0,197 | 45253 | -0,137 | 45442 | 0,01 |
| 44431 | 0,381 | 45115 | 0,113 | 45254 | -0,218 | 45443 | -0,005 |
| 44432 | 0,325 | 45121 | 0,251 | 45255 | -0,302 | 45444 | -0,086 |
| 44433 | 0,31 | 45122 | 0,195 | 45311 | 0,313 | 45445 | -0,17 |
| 44434 | 0,167 | 45123 | 0,18 | 45312 | 0,257 | 45451 | -0,092 |
| 44435 | 0,019 | 45124 | 0,099 | 45313 | 0,242 | 45452 | -0,148 |
| 44441 | 0,226 | 45125 | 0,015 | 45314 | 0,161 | 45453 | -0,163 |
| 44442 | 0,169 | 45131 | 0,226 | 45315 | 0,077 | 45454 | -0,244 |
| 44443 | 0,155 | 45132 | 0,17 | 45321 | 0,215 | 45455 | -0,328 |
| 44444 | 0,036 | 45133 | 0,155 | 45322 | 0,159 | 45511 | 0,255 |

105

| | | | | | Statistical | Allaly SIS I lai | 1 030236721 LL |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 45512 | 0,199 | 51151 | -0,05 | 51335 | -0,059 | 51524 | -0,009 |
| 45513 | 0,184 | 51152 | -0,106 | 51341 | 0,072 | 51525 | -0,093 |
| 45514 | 0,103 | 51153 | -0,121 | 51342 | 0,016 | 51531 | 0,119 |
| 45515 | 0,019 | 51154 | -0,202 | 51343 | 0,001 | 51532 | 0,063 |
| 45521 | 0,157 | 51155 | -0,286 | 51344 | -0,08 | 51533 | 0,048 |
| 45522 | 0,101 | 51211 | 0,307 | 51345 | -0,164 | 51534 | -0,033 |
| 45523 | 0,086 | 51212 | 0,251 | 51351 | -0,086 | 51535 | -0,117 |
| 45524 | 0,005 | 51213 | 0,236 | 51352 | -0,142 | 51541 | 0,014 |
| 45525 | -0,079 | 51214 | 0,155 | 51353 | -0,157 | 51542 | -0,042 |
| 45531 | 0,132 | 51215 | 0,071 | 51354 | -0,238 | 51543 | -0,057 |
| 45532 | 0,076 | 51221 | 0,209 | 51355 | -0,322 | 51544 | -0,138 |
| 45533 | 0,061 | 51222 | 0,152 | 51411 | 0,281 | 51545 | -0,222 |
| 45534 | -0,02 | 51223 | 0,138 | 51412 | 0,225 | 51551 | -0,144 |
| 45535 | -0,104 | 51224 | 0,057 | 51413 | 0,21 | 51552 | -0,2 |
| 45541 | 0,027 | 51225 | -0,027 | 51414 | 0,129 | 51553 | -0,215 |
| 45542 | -0,029 | 51231 | 0,184 | 51415 | 0,045 | 51554 | -0,296 |
| 45543 | -0,044 | 51232 | 0,128 | 51421 | 0,182 | 51555 | -0,238 |
| 45544 | -0,125 | 51233 | 0,113 | 51421 | 0,182 | 52111 | 0,249 |
| 45545 | -0,123 | 51234 | 0,032 | 51423 | 0,111 | 52111 | 0,193 |
| 45551 | | | * | | * | | 0,178 |
| | -0,131 | 51235 | -0,052 | 51424 | 0,03 | 52113 | |
| 45552 | -0,187 | 51241 | 0,079 | 51425 | -0,054 | 52114 | 0,097 |
| 45553 | -0,202 | 51242 | 0,023 | 51431 | 0,158 | 52115 | 0,013 |
| 45554 | -0,283 | 51243 | 0,008 | 51432 | 0,102 | 52121 | 0,151 |
| 45555 | -0,367 | 51244 | -0,073 | 51433 | 0,087 | 52122 | 0,095 |
| 51111 | 0,336 | 51245 | -0,157 | 51434 | 0,006 | 52123 | 0,08 |
| 51112 | 0,28 | 51251 | -0,079 | 51435 | -0,078 | 52124 | -0,001 |
| 51113 | 0,265 | 51252 | -0,135 | 51441 | 0,053 | 52125 | -0,085 |
| 51114 | 0,184 | 51253 | -0,15 | 51442 | -0,003 | 52131 | 0,126 |
| 51115 | 0,1 | 51254 | -0,231 | 51443 | -0,018 | 52132 | 0,07 |
| 51121 | 0,238 | 51255 | -0,315 | 51444 | -0,099 | 52133 | 0,055 |
| 51122 | 0,181 | 51311 | 0,3 | 51445 | -0,183 | 52134 | -0,026 |
| 51123 | 0,167 | 51312 | 0,244 | 51451 | -0,105 | 52135 | -0,11 |
| 51124 | 0,086 | 51313 | 0,229 | 51452 | -0,161 | 52141 | 0,021 |
| 51125 | 0,002 | 51314 | 0,148 | 51453 | -0,176 | 52142 | -0,035 |
| 51131 | 0,213 | 51315 | 0,064 | 51454 | -0,257 | 52143 | -0,05 |
| 51132 | 0,157 | 51321 | 0,202 | 51455 | -0,341 | 52144 | -0,131 |
| 51133 | 0,142 | 51322 | 0,145 | 51511 | 0,242 | 52145 | -0,215 |
| 51134 | 0,061 | 51323 | 0,131 | 51512 | 0,186 | 52151 | -0,137 |
| 51135 | -0,023 | 51324 | 0,05 | 51513 | 0,171 | 52152 | -0,193 |
| 51141 | 0,108 | 51325 | -0,035 | 51514 | 0,09 | 52153 | -0,208 |
| 51142 | 0,052 | 51331 | 0,177 | 51515 | 0,006 | 52154 | -0,289 |
| 51143 | 0,037 | 51332 | 0,121 | 51521 | 0,144 | 52155 | -0,373 |
| 51144 | -0,044 | 51333 | 0,106 | 51522 | 0,087 | 52211 | 0,221 |
| 51145 | -0,128 | 51334 | 0,025 | 51523 | 0,073 | 52212 | 0,164 |

106

| | | | | | Statistical | Anaiysis Piai | 1 030238/2FLZ |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 52213 | 0,15 | 52352 | -0,229 | 52541 | -0,073 | 53225 | -0,131 |
| 52214 | 0,069 | 52353 | -0,244 | 52542 | -0,129 | 53231 | 0,08 |
| 52215 | -0,016 | 52354 | -0,325 | 52543 | -0,144 | 53232 | 0,024 |
| 52221 | 0,122 | 52355 | -0,409 | 52544 | -0,225 | 53233 | 0,009 |
| 52222 | 0,066 | 52411 | 0,194 | 52545 | -0,309 | 53234 | -0,072 |
| 52223 | 0,051 | 52412 | 0,138 | 52551 | -0,231 | 53235 | -0,156 |
| 52224 | -0,03 | 52413 | 0,123 | 52552 | -0,287 | 53241 | -0,025 |
| 52225 | -0,114 | 52414 | 0,042 | 52553 | -0,302 | 53242 | -0,081 |
| 52231 | 0,098 | 52415 | -0,042 | 52554 | -0,383 | 53243 | -0,096 |
| 52232 | 0,041 | 52421 | 0,096 | 52555 | -0,467 | 53244 | -0,177 |
| 52233 | 0,027 | 52422 | 0,04 | 53111 | 0,232 | 53245 | -0,261 |
| 52234 | -0,054 | 52423 | 0,025 | 53112 | 0,176 | 53251 | -0,183 |
| 52235 | -0,139 | 52424 | -0,056 | 53113 | 0,161 | 53252 | -0,239 |
| 52241 | -0,008 | 52425 | -0,14 | 53114 | 0,08 | 53253 | -0,254 |
| 52242 | -0,064 | 52431 | 0,071 | 53115 | -0,004 | 53254 | -0,335 |
| 52243 | -0,079 | 52432 | 0,015 | 53121 | 0,134 | 53255 | -0,419 |
| 52244 | -0,16 | 52433 | 0,019 | 53122 | 0,077 | 53311 | 0,196 |
| 52245 | -0,244 | 52434 | -0,081 | 53123 | 0,063 | 53311 | 0,14 |
| 52251 | -0,166 | 52435 | -0,165 | 53124 | -0,019 | 53313 | 0,125 |
| 52252 | , and the second | 52441 | -0,163 | 53124 | -0,103 | | 0,123 |
| | -0,222 | | • | | | 53314 | |
| 52253 | -0,237 | 52442 | -0,09 | 53131 | 0,109 | 53315 | -0,04 |
| 52254 | -0,317 | 52443 | -0,105 | 53132 | 0,053 | 53321 | 0,098 |
| 52255 | -0,402 | 52444 | -0,186 | 53133 | 0,038 | 53322 | 0,041 |
| 52311 | 0,213 | 52445 | -0,27 | 53134 | -0,043 | 53323 | 0,027 |
| 52312 | 0,157 | 52451 | -0,192 | 53135 | -0,127 | 53324 | -0,055 |
| 52313 | 0,142 | 52452 | -0,248 | 53141 | 0,004 | 53325 | -0,139 |
| 52314 | 0,061 | 52453 | -0,263 | 53142 | -0,052 | 53331 | 0,073 |
| 52315 | -0,023 | 52454 | -0,344 | 53143 | -0,067 | 53332 | 0,017 |
| 52321 | 0,115 | 52455 | -0,428 | 53144 | -0,148 | 53333 | 0,002 |
| 52322 | 0,059 | 52511 | 0,155 | 53145 | -0,232 | 53334 | -0,079 |
| 52323 | 0,044 | 52512 | 0,099 | 53151 | -0,154 | 53335 | -0,163 |
| 52324 | -0,037 | 52513 | 0,084 | 53152 | -0,21 | 53341 | -0,032 |
| 52325 | -0,121 | 52514 | 0,003 | 53153 | -0,225 | 53342 | -0,088 |
| 52331 | 0,09 | 52515 | -0,081 | 53154 | -0,306 | 53343 | -0,103 |
| 52332 | 0,034 | 52521 | 0,057 | 53155 | -0,39 | 53344 | -0,184 |
| 52333 | 0,019 | 52522 | 0,001 | 53211 | 0,203 | 53345 | -0,268 |
| 52334 | -0,062 | 52523 | -0,014 | 53212 | 0,147 | 53351 | -0,19 |
| 52335 | -0,146 | 52524 | -0,095 | 53213 | 0,132 | 53352 | -0,246 |
| 52341 | -0,015 | 52525 | -0,179 | 53214 | 0,051 | 53353 | -0,261 |
| 52342 | -0,071 | 52531 | 0,032 | 53215 | -0,033 | 53354 | -0,342 |
| 52343 | -0,086 | 52532 | -0,024 | 53221 | 0,105 | 53355 | -0,426 |
| 52344 | -0,167 | 52533 | -0,039 | 53222 | 0,048 | 53411 | 0,177 |
| 52345 | -0,251 | 52534 | -0,12 | 53223 | 0,034 | 53412 | 0,121 |
| 52351 | -0,173 | 52535 | -0,204 | 53224 | -0,047 | 53413 | 0,106 |

107

| | | | | | Statistical | Analysis i lai | 1 030230 / 21 1220 |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 53414 | 0,025 | 53553 | -0,319 | 54242 | -0,108 | 54431 | 0,027 |
| 53415 | -0,059 | 53554 | -0,4 | 54243 | -0,123 | 54432 | -0,029 |
| 53421 | 0,078 | 53555 | -0,484 | 54244 | -0,204 | 54433 | -0,044 |
| 53422 | 0,022 | 54111 | 0,205 | 54245 | -0,288 | 54434 | -0,125 |
| 53423 | 0,007 | 54112 | 0,149 | 54251 | -0,21 | 54435 | -0,209 |
| 53424 | -0,074 | 54113 | 0,134 | 54252 | -0,266 | 54441 | -0,078 |
| 53425 | -0,158 | 54114 | 0,053 | 54253 | -0,281 | 54442 | -0,134 |
| 53431 | 0,054 | 54115 | -0,031 | 54254 | -0,362 | 54443 | -0,149 |
| 53432 | -0,002 | 54121 | 0,107 | 54255 | -0,446 | 54444 | -0,23 |
| 53433 | -0,017 | 54122 | 0,05 | 54311 | 0,169 | 54445 | -0,314 |
| 53434 | -0,098 | 54123 | 0,036 | 54312 | 0,113 | 54451 | -0,236 |
| 53435 | -0,182 | 54124 | -0,045 | 54313 | 0,098 | 54452 | -0,292 |
| 53441 | -0,051 | 54125 | -0,129 | 54314 | 0,017 | 54453 | -0,307 |
| 53442 | -0,107 | 54131 | 0,082 | 54315 | -0,067 | 54454 | -0,388 |
| 53443 | -0,122 | 54132 | 0,026 | 54321 | 0,071 | 54455 | -0,472 |
| 53444 | -0,203 | 54133 | 0,011 | 54322 | 0,014 | 54511 | 0,111 |
| 53445 | -0,287 | 54134 | -0,07 | 54323 | 0 | 54512 | 0,055 |
| 53451 | -0,209 | 54135 | -0,154 | 54324 | -0,081 | 54513 | 0,04 |
| 53452 | -0,265 | 54141 | -0,023 | 54325 | -0,165 | 54514 | -0,041 |
| 53453 | -0,28 | 54142 | -0,079 | 54331 | 0,046 | 54515 | -0,125 |
| 53454 | -0,361 | 54143 | -0,094 | 54332 | -0,01 | 54521 | 0,013 |
| 53455 | -0,445 | 54144 | -0,175 | 54333 | -0,025 | 54522 | -0,044 |
| 53511 | 0,138 | 54145 | -0,259 | 54334 | -0,106 | 54523 | -0,058 |
| 53512 | 0,082 | 54151 | -0,181 | 54335 | -0,19 | 54524 | -0,139 |
| 53513 | 0,067 | 54152 | -0,237 | 54341 | -0,059 | 54525 | -0,223 |
| 53514 | -0,014 | 54153 | -0,252 | 54342 | -0,115 | 54531 | -0,012 |
| 53515 | -0,098 | 54154 | -0,333 | 54343 | -0,13 | 54532 | -0,068 |
| 53521 | 0,04 | 54155 | -0,417 | 54344 | -0,211 | 54533 | -0,083 |
| 53522 | -0,017 | 54211 | 0,176 | 54345 | -0,295 | 54534 | -0,164 |
| 53523 | -0,032 | 54212 | 0,12 | 54351 | -0,217 | 54535 | -0,248 |
| 53524 | -0,113 | 54213 | 0,105 | 54352 | -0,273 | 54541 | -0,117 |
| 53525 | -0,197 | 54214 | 0,024 | 54353 | -0,288 | 54542 | -0,173 |
| 53531 | 0,015 | 54215 | -0,06 | 54354 | -0,369 | 54543 | -0,188 |
| 53532 | -0,041 | 54221 | 0,078 | 54355 | -0,453 | 54544 | -0,269 |
| 53533 | -0,056 | 54222 | 0,022 | 54411 | 0,15 | 54545 | -0,353 |
| 53534 | -0,137 | 54223 | 0,007 | 54412 | 0,094 | 54551 | -0,275 |
| 53535 | -0,221 | 54224 | -0,074 | 54413 | 0,079 | 54552 | -0,331 |
| 53541 | -0,09 | 54225 | -0,158 | 54414 | -0,002 | 54553 | -0,346 |
| 53542 | -0,146 | 54231 | 0,053 | 54415 | -0,086 | 54554 | -0,427 |
| 53543 | -0,161 | 54232 | -0,003 | 54421 | 0,052 | 54555 | -0,511 |
| 53544 | -0,242 | 54233 | -0,018 | 54422 | -0,005 | 55111 | 0,122 |
| 53545 | -0,326 | 54234 | -0,099 | 54423 | -0,019 | 55112 | 0,066 |
| 53551 | -0,248 | 54235 | -0,183 | 54424 | -0,1 | 55113 | 0,051 |
| 53552 | -0,304 | 54241 | -0,052 | 54425 | -0,184 | 55114 | -0,03 |

108

| | | | | | Statistical | Allalysis Flai | 1 030238/2FLZ3UU |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 55115 | -0,114 | 55254 | -0,445 | 55443 | -0,232 | | |
| 55121 | 0,024 | 55255 | -0,529 | 55444 | -0,313 | | |
| 55122 | -0,033 | 55311 | 0,086 | 55445 | -0,397 | | |
| 55123 | -0,048 | 55312 | 0,03 | 55451 | -0,319 | | |
| 55124 | -0,129 | 55313 | 0,015 | 55452 | -0,375 | | |
| 55125 | -0,213 | 55314 | -0,066 | 55453 | -0,39 | | |
| 55131 | -0,001 | 55315 | -0,15 | 55454 | -0,471 | | |
| 55132 | -0,057 | 55321 | -0,013 | 55455 | -0,555 | | |
| 55133 | -0,072 | 55322 | -0,069 | 55511 | 0,028 | | |
| 55134 | -0,153 | 55323 | -0,084 | 55512 | -0,028 | | |
| 55135 | -0,237 | 55324 | -0,165 | 55513 | -0,043 | | |
| 55141 | -0,106 | 55325 | -0,249 | 55514 | -0,124 | | |
| 55142 | -0,162 | 55331 | -0,037 | 55515 | -0,208 | | |
| 55143 | -0,177 | 55332 | -0,093 | 55521 | -0,208 | | |
| 55144 | -0,177 | 55333 | -0,108 | 55522 | -0,127 | | |
| 55145 | -0,342 | 55334 | -0,189 | 55523 | -0,127 | | |
| 55151 | -0,264 | 55335 | -0,189 | 55524 | -0,142 | | |
| 55152 | -0,204 | 55341 | -0,273 | 55525 | -0,223 | | |
| 55153 | -0,335 | 55342 | -0,142 | 55531 | -0,095 | | |
| 55154 | -0,416 | 55343 | -0,213 | 55532 | -0,151 | | |
| 55155 | -0,5 | 55344 | -0,294 | 55533 | -0,166 | | |
| 55211 | 0,093 | 55345 | -0,378 | 55534 | -0,247 | | |
| 55212 | 0,037 | 55351 | -0,3 | 55535 | -0,331 | | |
| 55213 | 0,022 | 55352 | -0,356 | 55541 | -0,2 | | |
| 55214 | -0,059 | 55353 | -0,371 | 55542 | -0,256 | | |
| 55215 | -0,143 | 55354 | -0,452 | 55543 | -0,271 | | |
| 55221 | -0,005 | 55355 | -0,536 | 55544 | -0,352 | | |
| 55222 | -0,062 | 55411 | 0,067 | 55545 | -0,436 | | |
| 55223 | -0,076 | 55412 | 0,011 | 55551 | -0,358 | | |
| 55224 | -0,157 | 55413 | -0,004 | 55552 | -0,414 | | |
| 55225 | -0,241 | 55414 | -0,085 | 55553 | -0,429 | | |
| 55231 | -0,03 | 55415 | -0,169 | 55554 | -0,51 | | |
| 55232 | -0,086 | 55421 | -0,032 | 55555 | -0,594 | | |
| 55233 | -0,101 | 55422 | -0,088 | | | | |
| 55234 | -0,182 | 55423 | -0,103 | | | | |
| 55235 | -0,266 | 55424 | -0,184 | | | | |
| 55241 | -0,135 | 55425 | -0,268 | | | | |
| 55242 | -0,191 | 55431 | -0,056 | | | | |
| 55243 | -0,206 | 55432 | -0,112 | | | | |
| 55244 | -0,287 | 55433 | -0,127 | | | | |
| 55245 | -0,371 | 55434 | -0,208 | | | | |
| 55251 | -0,293 | 55435 | -0,292 | | | | |
| 55252 | -0,349 | 55441 | -0,161 | | | | |
| 55253 | -0,364 | 55442 | -0,217 | | | | |

#### ATTACHMENT 6. : HRS DERIVATION

The HRS categories should be evaluated from 6 to 1. First check if the subject falls in category 6 (has the subject died?) if not then we evaluate category 5, if not 5 then evaluate category 4 and so on.

The HRS is evaluated at baseline and per day, relative to the first study drug intake.

The baseline HRS is covering the full baseline/screening/day 1 visit which can occur on 2 days. Timing of first study drug intake is not taken into account.

#### Note:

• VSOXYSAT is assessed 3 times per day (or per baseline visit). In case one of the assessments says 'N' then the final result for that day (or baseline visit) is 'N', else if one of the assessments is 'NA' then the final result is 'NA' else if one of the assessments is missing then final result is missing.

```
So a combination of 'Y', "", "N" → result ='N'
'Y', "", "NA" → result ='NA'
'Y; 'Y', '' → result =''
'Y; 'Y', 'Y' → result ='Y'
```

On the baseline visit, on days at or after HO end date or on the day of discontinuation it might be that less than 3 assessments are done. Therefore, take only the records into account from the dataset on those days as planned. The same rules above apply to derive the final result per day when more than 1 assessment is collected.

- In case the subject withdrew from the study, the HRS will be set to missing from the next day onwards.
- In case of chronic oxygen use and multiple CMARTN values on a day we consider the worst value: In case one of the values is 'N' then final result for that day (or baseline visit) is 'N', else if one of the assessments is missing then final result is missing.
- The list of types of supplemental oxygen and invasive mechanical ventilation can be extended depending on the medical review (see DPS part 2 or Excel sheet of the medical review)
- The list of hospitalization terms (i.e.: ICU or WARD) can be extended depending on the medical review (see DPS part 2 or Excel sheet of the medical review).
- If the Subjects has no HO data, the subject is considered to be in the hospital during the trial. All other aspect of the HRS will be evaluated according to the derivation below.
- In case the readiness for discharge (RDISHOSP) is assessed more than once per day (baseline visit) we consider the worst value: in case one of the values is 'N' then the final result of that day (or baseline visit) is 'N'

Some clarification is required for following categories:

#### 6. Death

When DM.DTHDTC<=(date of assessment)

# 5. Requiring invasive mechanical ventilation;

When CMSTDTC<=(date of assessment) <=CMENDTC where CMADMTP="INVASIVE MECHANICAL VENTILATION"

And CMADMDSC in ('Through Endotracheal tube' 'Through Tracheostomy tube' or 'Through ECMO')

# 4. Admitted to the ICU;

From the HO data set:

hostdy <=(day of assessment)<=hoendy hoterm = 'ICU'

From the SS data set:

SSTESTCD= 'REQICU' and SSSTRESC='Y'

Or SSTESTCD= 'REASICU' and SSSTRESC='Y'

Or both REQICU and REAICU is missing and NOT (RDISHOSP = 'Y' on the day of assessment and RDISHOSP = 'Y' on the day (baseline visit) before)

OR

From the HO data set:

hostdy <=(day of assessment)<=hoendy

hoterm = 'WARD'

From the SS data set:

SSTESTCD='REASICU' and SSSTRESC='Y'

OR

SSTESTCD='REQICU' and SSSTRESC='Y'

# 3. Non-ICU hospitalization, requiring supplemental oxygen

# **Non-ICU hospitalization:**

hostdy <=(day of assessment)<=hoendy

hoterm = 'Hospital inpatient Department (WARD)'

NOT (RDISHOSP='Y' on the day of assessment and RDISHOSP='Y' on day(baseline visit) before)

OR

hostdy <=(day of assessment)<=hoendy

hoterm = 'ICU'

NOT (RDISHOSP='Y' on the day of assessment and RDISHOSP='Y' on day(baseline visit) before)

OR

(day of assessment)=hoendy+1 RDISHOSP='N' on day(baseline visit) before

OR

In case re-hospitalization occurred (there is a day between the HOENDY of the previous record and HOSTDY of the next record)

(day of assessment) = HOSTDY (of the re-hospitalization)

NOT (RDISHOSP='Y' on the day of assessment and RDISHOSP='Y' on day(baseline visit) before)

#### **AND**

# Requiring supplemental oxygen:

'Receiving supplemental oxygen through a face mask or nasal cannula and not being able to sustain a blood oxygen saturation of  $\geq 94\%$  when breathing room air for 15 minutes at any time on the day of assessment.'

FAOBJ=CHRONIC OXYGEN USE and FAORRES='N'

CMADMTP in ("Non-Invasive Mechanical Ventilation", "Nasal Cannula", "Venturi Mask", "Simple Face Mask", "Nonrebreathing Face Mask with Reservoir and One-Way Valve".)

CMTRT=SUPPLEMENTAL OXYGEN and CMSTDTC <= date of assessment <= CMENDTC

VSOXYSAT in ('N' 'NA') at any time during the day of assessment (OR is missing)

OR

'If supplemental oxygen was provided chronically pre-influenza infection (based on medical history), that amount of supplemental oxygen is exceeded to prevent hypoxia, tachypnea or dyspnea at some point on the day of assessment.'

FAOBJ=CHRONIC OXYGEN USE and FAORRES='Y'

CMARTN = 'N'

CMADMTP in ("Non-Invasive Mechanical Ventilation", "Nasal Cannula", "Venturi Mask", "Simple Face Mask", "Nonrebreathing Face Mask with Reservoir and One-Way Valve".) and CMTRT=SUPPLEMENTAL OXYGEN and CMSTDTC <= date of assessment <= CMENDTC

OR

'Not receiving supplemental oxygen and Having a blood oxygen saturation of <94% when breathing room air for 15 minutes at any measurement on the day of assessment'

No record in cm with oxygen supplementation

VSOXYSAT='N' at any time on the day of assessment OR [VSTESTCD='OXYSAT' and VSORRES<94% and VSOXSMRA='Y']

OR

'Not receiving supplemental oxygen and in case of known pre-influenza SpO2 <94% (eg, due to COPD), the current blood oxygen saturation on room air is lower than pre-influenza infection levels by at least 3%.'

No record in cm with oxygen supplementation

VSEVINTX= PRE-INFLUENZA INFECTION and VSTESTCD='OXYSAT and 'VSORRES<94% and VSRMAIR='Y'

VSORRES and VSTESTCD=OXYSAT (of day of assessment) < [ VSORRES and VSEVINTX= PRE-INFLUENZA INFECTION and VSTESTCD='OXYSAT and VSRMAIR='Y' - 3 ]

# 2. Non-ICU hospitalization, not requiring supplemental oxygen

hostdy <=(day of assessment)<=hoendy

hoterm = 'Hospital inpatient Department (WARD)'

NOT (RDISHOSP='Y' on the day of assessment and RDISHOSP='Y' on day(baseline visit) before)

hostdy <=(day of assessment)<=hoendy

hoterm = 'ICU'

NOT (RDISHOSP='Y' on the day of assessment and RDISHOSP='Y' on day(baseline visit) before)

OR

(day of assessment)=hoendy+1 RDISHOSP='N' on day(baseline visit) before

OR

In case re-hospitalization occurred (there is a day between the HOENDY of the previous record and HOSTDY of the next record)

(day of assessment) = HOSTDY (of the re-hospitalization)

NOT (RDISHOSP='Y' on the day of assessment and RDISHOSP='Y' on day(baseline visit) before)

# 1. Not hospitalized

# Some examples

# Discharge against medical advice

If a subject is discharged 'against medical advice' on the day prior to the day of assessment, the subject will be considered as hospitalized (evaluating the others aspects of the HRS to define the correct category, e.g.: requiring supplemental oxygen, on the day of assessment)

We have a discharged against medical advice if on the day the subject is discharged (according to the HO dataset) the investigator indicated he is not ready and his SS status is discharged,

| | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | Day 8 |
|---|---|---|---|---|---|---|
| Status (HO) | Hospitalized | Hospitalized | Hospitalized | Discharged | Home | Home |
| Case 1 | | | | | | |
| ready (SS) | Not ready | Not ready | Not ready | Not ready | | |
| Status(SS) | hospitalized | hospitalized | hospitalized | Hospitalized | discharged | |
| Against medical advice? | | | | | NO | |
| HRS | >1 | >1 | >1 | >1 | >1 | HOME |
| Case 2 | | | | | | |
| ready (SS) | Not ready | Not ready | Not ready | Not ready | Ready | |
| Status(SS) | hospitalized | hospitalized | hospitalized | Hospitalized | discharged | |
| Against medical advice? | | | | | NO | |
| HRS | >1 | >1 | >1 | >1 | >1 | HOME |
| Case 3 | | | | | | |
| ready (SS) | Not ready | Not ready | Not ready | Not ready | Not ready | |
| Status(SS) | hospitalized | hospitalized | hospitalized | Hospitalized | discharged | |
| Against medical advice? | | | | | NO | |
| HRS | >1 | >1 | >1 | >1 | >1 | HOME |
| Case 4 | | | | | | |
| ready (SS) | Not ready | Not ready | Not ready | Not ready | | |
| Status(SS) | hospitalized | hospitalized | hospitalized | Discharged | | |

| Against medical advice? | | | | YES | | |
|---|---|---|---|---|---|---|
| HRS | >1 | >1 | >1 | >1 | >1 | Missing |
| Case 5 | | | | | | |
| ready (SS) | Not ready | Not ready | Not ready | Ready | | |
| Status(SS) | hospitalized | hospitalized | hospitalized | discharged | | |
| Against | | | | NO | | |
| medical advice? | | | | NO | | |
| HRS | >1 | >1 | >1 | >1 | HOME | HOME |
| Case 6 | | | | | | |
| ready (SS) | Not ready | Not ready | Not ready | Ready | | |
| Status(SS) | hospitalized | hospitalized | hospitalized | hospitalized | discharged | |
| Against | | | | | | |
| _ | | | | NO | | |
| medical | | | | NO | | |
| advice? | <b>&gt;1</b> | >1 | >1 | | HOME | HOME |
| | >1 | >1 | >1 | NO >1 | HOME | HOME |
| advice? | >1 | >1 | >1 | | НОМЕ | HOME |
| advice?<br>HRS | >1<br>Not ready | >1<br>Not ready | >1 Ready | | HOME | HOME<br> |
| advice?<br>HRS<br>Case 7 | | | | >1 | | |
| advice?<br>HRS Case 7 ready (SS) Status(SS) Against | Not ready | Not ready | Ready | >1 Ready hospitalized | | |
| advice?<br>HRS Case 7 ready (SS) Status(SS) Against medical | Not ready | Not ready | Ready | >1<br>Ready | | |
| advice?<br>HRS Case 7 ready (SS) Status(SS) Against | Not ready | Not ready | Ready | >1 Ready hospitalized | | |
| advice? HRS Case 7 ready (SS) Status(SS) Against medical advice? HRS | Not ready<br>hospitalized | Not ready<br>hospitalized | Ready<br>hospitalized | >1 Ready hospitalized NO | <br>discharged | |
| advice? HRS Case 7 ready (SS) Status(SS) Against medical advice? HRS Case 8 | Not ready<br>hospitalized | Not ready<br>hospitalized | Ready hospitalized | >1 Ready hospitalized NO HOME | <br>discharged | <br>HOME |
| advice? HRS Case 7 ready (SS) Status(SS) Against medical advice? HRS Case 8 ready (SS) | Not ready hospitalized >1 Not ready | Not ready hospitalized >1 Not ready | Ready hospitalized >1 Not ready | >1 Ready hospitalized NO HOME | <br>discharged | |
| advice? HRS Case 7 ready (SS) Status(SS) Against medical advice? HRS Case 8 | Not ready<br>hospitalized | Not ready<br>hospitalized | Ready hospitalized | >1 Ready hospitalized NO HOME | <br>discharged | <br>HOME |
| advice? HRS Case 7 ready (SS) Status(SS) Against medical advice? HRS Case 8 ready (SS) Status(SS) Against medical | Not ready hospitalized >1 Not ready | Not ready hospitalized >1 Not ready | Ready hospitalized >1 Not ready | >1 Ready hospitalized NO HOME | <br>discharged | <br>HOME |
| advice? HRS Case 7 ready (SS) Status(SS) Against medical advice? HRS Case 8 ready (SS) Status(SS) Against | Not ready hospitalized >1 Not ready | Not ready hospitalized >1 Not ready | Ready hospitalized >1 Not ready discharged | >1 Ready hospitalized NO HOME | <br>discharged | <br>HOME |

Only in case 4 above we have a discharge against medical advice which would lead to missing values from day 8 onwards. The HRS on day 7 is defined by the other aspects of the HRS (requiring oxygen, ICU,...) on day 7 and not copied from day 6.

# Requiring supplemental oxygen

| | Case 1 | Case 2 | Case 3 | Case 4 | Case 5 | Case 6 |
|---|---|---|---|---|---|---|
| supplemental oxygen (CM) | YES | YES | NO | NO | NO | NO |
| Chronic oxygen use | No | yes | Not used | Not used | Not used | Not used |
| returned to prior level? | Not used | N | Not used | Not used | Not used | Not used |
| pre influenza infection levels | Not used | Not used | Not used | Not used | Not used | 93 |
| Oxysat record < pre-influenza level at any moment during the day sustain >94% Oxy sat (VSOXYSAT) Oxysat record <94% at any moment during the day | Not used N' missing or 'NA' Not used | Not used N' missing or 'NA' Not used | Not used<br>N' at any<br>time during<br>the day | Not used Missing or NA yes | Not used YEs yes | yes<br>Not used<br>Not used |
| REQUIRING SUPPLEMENTAL OXYGEN? | YES | YES | YES | YES | YES | YES |

# To pay attention to

| | Case 7 | Case 8 | Case 9 | Case 10 | Case 11 | Case 12 |
|---|---|---|---|---|---|---|
| supplemental oxygen (CM) | YES | No | No | YEs | YEs | YEs |
| Chronic oxygen use | No | Not used | Yes | Yes | Yes | Yes |
| returned to prior level? | Not used | Not used | N | Missing | N | у |
| pre influenza infection levels | Not used | 93 | Not used | Not used | Not used | Not used |
| Oxysat record < pre-influenza level at any moment during the day | not used | yes | Not used | Not used | Not used | Not used |
| sustain >94% Oxy sat (VSOXYSAT) | missing | yes | Missing | Missing | Yes | Yes |
| Oxysat record <94% at any moment during the day | yes | Not used | Missing | Not used | Not used | yes |
| REQUIRING SUPPLEMENTAL OXYGEN? | NO | YES | NO | YES | YES | NO |